## MASTER STATISTICAL ANALYSIS PLAN

MASTER PROTOCOL: COV-01 (COMMUNITY)

INDUSTRY ALLIANCE PLATFORM TRIAL TO ASSESS THE EFFICACY AND SAFETY OF MULTIPLE CANDIDATE AGENTS FOR THE TREATMENT OF COVID-19 IN HOSPITALIZED PATIENTS

**AUTHOR: PPD** 

VERSION NUMBER AND DATE: AMENDMENT 1 v1.0, 23Apr2021

### MASTER STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

Master Statistical Analysis Plan (SAP) Amendment v1.0 (dated 23Apr2021) for master protocol COV-01

| | Name | Signature | Date (DDMmmYYYY) |
|-----------|------|-----------|------------------|
| Author: | PPD | PPD | |
| Position: | PPD | | |
| Company: | CCI | | |

Upon review of this document, the undersigned approves this version of the master SAP, authorizing that the content is acceptable for the reporting of this study.

| | Name | Signature | Date (DDMmmYYYY) |
|---------------|-------------|-----------|------------------|
| Approved by: | PPD | PPD | |
| Position: | PPD | | |
| Company: | CCI | | |
| On behalf of: | PPD | | |
| Position: | PPD | | |
| Company: | CCI | | |
| | | PPD | |
| Approved by: | PPD | | |
| Position: | PPD | | |
| Company: | Amgen, Inc. | | |



## **MODIFICATION HISTORY**

| Unique Identifier<br>for this Version | Date of the<br>Document<br>Version | Author | Significant Changes from Previous Version |
|---|---|---|---|
| Final, v1.0 | 18Nov2020 | PPD | Not Applicable – First Version |
| Amendment 1 v1.0 | 23Apr2021 | PPD | Updated Master Protocol version on which the Master SAP is based from version 3, dated 22-Oct-2020, to version 4, dated 16-Apr-2021. Updated definition of the data cut-off date for the Interim, Primary and Final Analyses of a sub-protocol in order to prevent potential inadvertent unblinding of patients randomized to the placebo plus SoC treatment group of another subprotocol included in the shared placebo plus SoC control arm of the sub-protocol of interest; Clarified that the 'concurrent' definition for selection of the concurrent placebo plus SoC patients for the control arm of a sub-protocol will be assessed on a site-by-site basis rather than across all sites; Updated definition of the safety analysis set so that patients randomized to the placebo arm of sub-protocol X selected for the shared placebo plus SoC control arm of sub-protocol Y who started taking subprotocol Y candidate agent for another indication after baseline will be presented under the shared placebo plus SoC control arm for sub-protocol Y safety analysis; Clarified that data collected during a discharge visit will also be mapped using time window for the by-visit summaries; |

CCI

PPD

Version Number: Version Date:

Amendment 1, v1.0 23Apr2021

Amgen Inc Master Protocol COV-01 

Master Statistical Analysis Plan

Added summaries further broken down by sub-protocol for the shared placebo plus SoC control arm to Sections 9 to 12;

Added a tipping point sensitivity analysis for the primary efficacy endpoint;

For each key secondary efficacy endpoint, removed the last observation carried forward (LOCF) sensitivity analysis as well as sensitivity analysis based on observed data (when applicable), and added a multiple imputation sensitivity analysis;

Clarified that the 95% two-sided confidence interval (CI) obtained from a logistic regression model will be the 95% two-sided Wald CI;

Added subgroup analyses by time since hospital admission at Study Day 1 ( $\leq$  5 days or > 5 days) for the primary and key secondary efficacy endpoints.

For each subprotocol, added separate summaries for patients randomized to the placebo plus SoC treatment group of the concerned sub-protocol for the prior and concomitant medications summaries as well as all safety summaries;

Added risk difference and associated 95% two-sided Wald CI for the treatment comparison of the overall incidence of serious treatment-emergent adverse events (TEAEs) and overall incidence of adverse events of special interest (when applicable for a sub-protocol);

Added summary of most common (5%) non-serious adverse events (AEs)

PPD

Version Number: Version Date: Amendment 1, v1.0 23Apr2021



## TABLE OF CONTENTS

| 1. | INTRODUCTION | 11 |
|---|---|---|
| 2. | STUDY OBJECTIVES | 11 |
| 2.1. | Primary Objective | 11 |
| 2.2. | Key Secondary Objectives | 11 |
| 2.3. | Other Secondary Objectives | 11 |
| 2.4. | Exploratory Objectives | 12 |
| 3. | STUDY DESIGN | 13 |
| 3.1. | General Description | 13 |
| 3.2. | Schedule of Activities | 16 |
| 3.3. | Changes to Planned Analyses from Master Protocol | 16 |
| 4. | PLANNED ANALYSES | 16 |
| 4.1. | IDMC Safety Analyses | 16 |
| 4.2. | Interim Analyses | 17 |
| 4.3. | Primary Analysis | 19 |
| 4.4. | Final Analysis | 20 |
| 4.5. | Selection of the Control Arm for an Analysis | 21 |
| 5. | ANALYSIS SETS | 22 |
| 5.1. | Full Analysis Set | 22 |
| 5.2. | Safety Analysis Set | 22 |
| 5.3. | Process for Analysis Set Assignment | 23 |
| CCI | Manai N | Amazamalina arritaturud C |
| PPD | Version Number:<br>Version Date: | Amendment 1, v1.0<br>23Apr2021 |

| 6. | GENERAL CONSIDERATIONS | 23 |
|---|---|---|
| 6.1. | Study Day | 23 |
| 6.2. | Baseline | 24 |
| 6.3. | Unscheduled Visits, Retests, Discharge, and Early Termination Data | 24 |
| 6.4. | Windowing Conventions | 25 |
| 6.5. | Common Calculations | 25 |
| 7. | STATISTICAL CONSIDERATIONS | 25 |
| 7.1. | Sample Size Calculation | 25 |
| 7.2. | Missing data | 27 |
| 7.3. | Statistical Tests | 27 |
| 7.4. | Multiple Comparisons/ Multiplicity | 27 |
| 7.5. | Multicenter Studies | 28 |
| 7.6. | Adjustments for Covariates and Factors to be Included in Analyses | 28 |
| 7.7. | Examination of Subgroups | 29 |
| 7.8. | Software Version | 31 |
| 8. | OUTPUT PRESENTATIONS | 31 |
| 9. | DISPOSITION AND WITHDRAWALS | 32 |
| <b>9.1.</b><br>9.1. | Disposition | 32<br>33 |
| 9.2. | Protocol Deviations | 33 |
| 10. | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 33 |
| 10.1. | Derivations | 34 |
| CCI<br>PPD | Version Number: Amendmen Version Date: 23 | nt 1, v1.0<br>3Apr2021 |

| 11. | DISEAS | SE HISTORY | 34 |
|---|---|---|---|
| 11.1. | | Derivations | 36 |
| 12. | MEDIC | CAL HISTORY | 37 |
| 13. | PRIOR | AND CONCOMITANT MEDICATIONS | 38 |
| 14. | EXPOS | URE TO STUDY DRUG | 39 |
| 15. | COMP | LIANCE WITH STUDY DRUG | 40 |
| 16. | <b>EFFIC</b> | ACY ENDPOINTS | 40 |
| 16.1. | | Primary Efficacy | 4( |
| 16. | 1.1. | Time to Confirmed Clinical Recovery through Day 29, without Re-Hospitalization Throug Day 29 | gh |
| 16 | 1.2. | Missing Data Imputation Method for Primary Efficacy Endpoint | |
| | 1.3. | Main Analysis of Primary Efficacy Endpoint | |
| | 1.4. | Sensitivity Analyses for Primary Efficacy Endpoint | |
| 16. | 1.5. | Supplementary Analyses for Primary Efficacy Endpoint | |
| 16.2. | | Secondary Efficacy | 47 |
| 16. | 2.1. | Secondary Efficacy Endpoints | |
| | 16.2.1.1. | Incidence of Patients with Oxygen-Free Recovery at Day 29 | |
| 1 | 16.2.1.2. | Incidence of Patients with ≥ 2-point Improvement from Baseline or Fit for Discharge on the Ordinal Scale at Day 29 | |
| 1 | 16.2.1.3. | Incidence of All-Cause Mortality through Day 29 | |
| | 16.2.1.4. | Distribution of Patients across the Categories of the 8-point Ordinal Scale for Clinical Sev | erity |
| 1 | 16.2.1.5. | at Days 8, 15, and 29 | |
| | 16.2.1.6. | Number of ICU Days from Day 1 through Day 29 | |
| | 16.2.1.7. | Number of Invasive Mechanical Ventilator Days from Day 1 through Day 29 | |
| | 16.2.1.8. | Incidence of Patients with Clinical Recovery by Days 8, 15, and 29 | |
| 1 | 16.2.1.9. | Incidence of Patients with Sustained Clinical Recovery as Confirmed by Day 60 Follow-ur | |
| 16. | 2.2. | Missing Data Imputation Method for Secondary Efficacy Endpoints | - |
| | 16.2.2.1. | Binary Endpoints | |
| | 16.2.2.2. | Ordinal Endpoints | |
| | 2.3. | Main Analysis of Secondary Efficacy Endpoints | |
| | 16.2.3.1. | Binary Endpoints | |
| | 16.2.3.2. | Ordinal Endpoints | |
| 16. | 2.4. | Sensitivity Analyses for Secondary Efficacy Endpoints | 54 |

CCI

PPD

Version Number: Version Date: Amendment 1, v1.0 23Apr2021



| Master Statistic | cal Analysis Plan | |
|---|---|---|
| 16.2.5. | Supplementary Analyses for Secondary Efficacy Endpoints | 50 |
| 16.3. | Exploratory Efficacy | 5' |
| | Exploratory Efficacy | |
| 16.4. | Additional Efficacy | |
| 16.4.1. | Additional Efficacy Endpoint | |
| 16.4.1.1. | Incidence of All-Cause Mortality through Day 60 | |
| 16.4.2.<br>16.4.3. | Missing Data Imputation Method for Additional Efficacy Endpoint Analysis of Additional Efficacy Endpoint | |
| 16.4.3.<br>16.4.4. | Sensitivity Analyses for Additional Efficacy Endpoint | |
| 16.4.5. | Supplementary Analyses for Additional Efficacy Endpoint | |
| 10.1.5. | supprementary interfect for industrial Enviously Emaperature | |
| 16.5. | Interim Analysis | 69 |
| 16.5.1. | Interim Analysis for Futility | |
| | · | |
| | NY ENDROINEG | <b>7</b> 1 |
| 17. SAFET | Y ENDPOINTS | 71 |
| 17.1. | Adverse Events | |
| 17.1.1. | All TEAEs | · |
| 17.1.1.1. | CTC Grading for AEs | |
| CCI | | |
| | Version Number | er: Amendment 1, v1.0 |
| PPD | Version Date: | 23Anr2021 |

### Master Statistical Analysis Plan

| 17.1.1.2. | Relationship to Study Drug, Non-Study Drug, and Study Procedure | |
|---|---|---|
| 17.1.2. | Fatal Adverse Events | |
| 17.1.3. | Serious Adverse Events | |
| 17.1.4. | Most Common Non-Serious Adverse Events | |
| 17.1.5. | TEAEs Leading to Dose Modifications | |
| 17.1.6. | TEAEs Leading to Discontinuation of Study Treatment | |
| 17.1.7. | AESIs | |
| 17.2. | Laboratory Evaluations | 74 |
| 17.2.1. | Laboratory Normalization | |
| 17.2.2. | CTCAE Toxicity Grades | |
| 17.2.3. | Laboratory Reference Ranges | 76 |
| 17.2 | V'4.1C' | 7. |
| 17.3. | Vital Signs | |
| 17.3.1. | Vital Signs Markedly Abnormal Criteria | T |
| 17.4. | ECG Evaluations | 78 |
| 17.5. | Physical Examination | 78 |
| | NOT SUMMARIZED OR PRESENTED | |
| APPENDIX 1 | PARTIAL DATE CONVENTIONS | 80 |
| Algorithm for T | reatment Emergence of Adverse Events | 80 |
| Algorithm for P | rior / Concomitant Medications | 81 |
| APPENDIX 2 | PROGRAMMING CONVENTIONS FOR OUTPUTS | 82 |
| Dates & Times. | | 82 |
| Spelling Format | | 82 |
| Paper Size, Orio | entation, and Margins | 82 |
| Fonts | | 82 |
| Presentation of | Treatment arms | 82 |
| Presentation of | Nominal Visits | 83 |
| CCI | | |
| PPD | Version Number:<br>Version Date: | Amendment 1, v1.0<br>23Apr2021 |

| Master Statistica | l Anal | vsis | Plar |
|-------------------|--------|------|------|
|-------------------|--------|------|------|


| Descriptive Statis | tics |
|---|---|
| Percentages | 83 |
| p-values | 83 |
| Listings | 84 |
| CCI | |
| APPENDIX 4 | VASOPRESSOR DRUG CODES AS PER THE WHO DRUG GLOBAL DICTIONARY, SEPTEMBER 2020, VERSION B3 |
| APPENDIX 5 | LABORATORY ASSESSMENTS 109 |
| APPENDIX 6 | CTCAE TOXICITY GRADE, VERSION 5.0111 |


#### 1. Introduction

This master statistical analysis plan (SAP) describes the rules and conventions to be used in the presentation and analysis of efficacy and safety data for protocol COV-01 (COMMUNITY). It describes the data to be summarized and analyzed, including specifics of the statistical analyses to be performed.

This master SAP is based on amendment 4 of the master protocol, dated 16-Apr-2021.

Presentation and analysis of efficacy and safety data specific to the sub-protocols as well as to the pharmacokinetic (PK) and pharmacodynamic (PD) endpoints will be described in separate sub-protocol SAPs.

#### 2. STUDY OBJECTIVES

#### 2.1. PRIMARY OBJECTIVE

The primary objective is to evaluate time to confirmed clinical recovery.

#### 2.2. KEY SECONDARY OBJECTIVES

The key secondary objectives are:

- To evaluate oxygen-free recovery;
- To evaluate improvement or being fit-for-discharge;
- To evaluate all-cause mortality.

#### 2.3. OTHER SECONDARY OBJECTIVES

The other secondary objectives are:

- To evaluate the distribution across categories on the 8-point ordinal scale, and the worst outcome;
- To evaluate intensive care unit (ICU) days;
- To evaluate invasive mechanical ventilator days;



- To evaluate clinical recovery;
- To evaluate sustained clinical recovery;
- To evaluate the safety of candidate agents as add-on therapy to standard of care (SoC) in patients with COVID-19.

## 2.4. EXPLORATORY OBJECTIVES



PPD

Version Number: Amendment 1, v1.0
Version Date: 23Apr2021

Amgen Inc

Master Statistical Analysis Plan

#### 3. STUDY DESIGN

#### 3.1. GENERAL DESCRIPTION

Coronavirus disease 2019 (COVID-19) Multiple Agents and Modulators Unified Industry Members Trial (COMMUNITY) is an adaptive, randomized, placebo-controlled platform study designed to rapidly evaluate candidate agents in the treatment of COVID-19. The study will include hospitalized adult patients (≥18 years of age) who have infection with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), the virus that causes COVID-19, as confirmed by laboratory tests and/or point of care tests. For inclusion, patients will need to be hospitalized with a clinical status of Grade 2 (hospitalized, on invasive mechanical ventilation or ECMO) to Grade 5 (hospitalized, not requiring supplemental oxygen, requiring ongoing medical care [COVID-19 related or otherwise]), as defined by an 8-point ordinal scale for clinical severity (refer to Section 16.1.1).

This study aims to identify efficacious candidate agents for treatment of COVID-19. The candidate agents may include, but will not be limited to, antivirals, vascular agents or immunomodulatory agents. Each sub-protocol will specify a single candidate agent or a combination of candidate agents to be administered.

The Master Protocol outlines the overall design of the study, including the population, inclusion and exclusion criteria, randomization scheme, primary, secondary, and exploratory endpoints, study design, statistical methodology, and planned analyses that are common for all candidate agents to be tested. The Master Protocol is structured such that multiple candidate agents from different pharmaceutical companies can be evaluated simultaneously. The plan is to add candidate agents as they are identified and/or to remove therapies based on results of interim analyses (IAs; e.g., due to futility or if they are considered unsafe). The shared placebo control group for a candidate agent will include only patients randomized during the same period in which the candidate agent is opened for enrollment (refer to Section 4.5). Patients will be randomized equally to either the candidate agent plus SoC or placebo plus SoC in a double-blind fashion. Patients who are randomized to placebo plus SoC will be subsequently randomized equally to a matching placebo corresponding to an available candidate agent whose sub-protocol the patient qualified for (i.e., a 2-stage randomization). Each patient in the placebo plus SoC group will receive one type of placebo. Therefore, patients may be aware of which sub-protocol they were randomized to but not whether they will receive active agent or placebo investigational product. The comparator group of a candidate agent will include patients randomized to any matching placebo for a candidate agent available at the time of randomization for that agent (refer to Section 4.5).

Patients will be screened on Day -1 (the day before the first dose of study treatment [candidate agent plus SoC or

Version Number: Amendment 1, v1.0 PPD Version Date: 23Apr2021

Amgen Inc Master Protocol COV-01 

Master Statistical Analysis Plan

placebo plus SoC] is scheduled) or Day 1 and will remain in the hospital from Day 1 until discharge. All patients will receive SoC treatment, either with blinded candidate agent or matching blinded placebo. The SoC will be based on appropriate local written guidelines in place at the site at the time of treatment in the study; the SoC may change during the course of the study as new information about treating COVID-19 becomes available. Dosing with the study treatment (as an add-on to SoC) will commence on Day 1. Patients will be assessed daily while hospitalized. If they are discharged from the hospital prior to Day 15, they will have study visits at Days 15 and 29 as an outpatient by telemedicine. The last day of primary assessments will be Day 29. An end-of-study visit will be conducted on Day 60 (± 4 days) via telemedicine (unless the patient is still hospitalized in which case it would be conducted in person).

Sub-protocols will outline the scientific rationale, additional eligibility criteria (if necessary), treatment dose and regimen, statistical analysis populations, and other specifics unique to each candidate agent. The sub-protocols may define adverse events of special interest (AESIs) and can include PK and/or PD assessments that are appropriate for the specific candidate agent. In order to enroll, a patient must meet all entry criteria for both the Master Protocol and at least one active sub-protocol.

The study will evaluate the candidate agents as an add-on to the SoC to assess safety and efficacy. IAs may be performed for each candidate agent to evaluate futility for candidate agents.

Patients will be stratified at randomization by baseline clinical severity of 2 on the 8-point ordinal scale (yes/no) and remdesivir use at baseline (yes/no).

Enrollment of patients will be continuous throughout the study for each candidate agent until the total number of planned patients for that agent is enrolled or until futility criteria is met at an IA, or if the agent is considered unsafe.

In addition, centers may elect to participate in separate Investigator-initiated studies collecting additional data on patients, as their resources permit.


Figure 1 Study Schema (with hypothetical example)



FA=final analysis; IA=interim analysis; PA = primary analysis; SoC=standard of care. '×' indicates that futility boundary has been met.

Note: IA1 and IA2 will be planned at information fractions of approximately 25% and 55% of expected number of recoveries i.e., after approximately 123 and 270 patients have met the primary endpoint of confirmed clinical recovery on a particular candidate agent plus SoC and placebo plus SoC, respectively.

Note: PA will occur after approximately 350 patients have been randomized to an active agent plus SoC and have had the opportunity to complete the Day 29 visit.

Note: FA will occur after all patients randomized to that agent plus SoC and the concurrent placebo plus SoC controls have had the opportunity to complete the Day 60 visit.

Note: In the above example, Agents #1, #2, and #5 met the futility boundary at IA1, while Agent #3 met the futility boundary at IA2, and so those agents could be discontinued in the study due to futility.

Note: Patients who are randomized to placebo plus SoC will be subsequently randomized equally to a matching placebo corresponding to an available agent whose sub-protocol the patient qualified for (i.e., a 2-stage randomization).



## 3.2. SCHEDULE OF ACTIVITIES

An example of a schedule of activities can be found in Section 1.3 of the Master Protocol. Each sub-protocol may have its own schedule of activities.

#### 3.3. CHANGES TO PLANNED ANALYSES FROM MASTER PROTOCOL

The 'average ordinal scale for clinical severity score over Day 1 to Day 29' other secondary efficacy endpoint is
updated to 'average ordinal scale for clinical severity score over Day 2 to Day 29' since Day 1 is the baseline
value.

#### 4. PLANNED ANALYSES

The following analyses will be performed for each sub-protocol:

- Independent data monitoring committee (IDMC) safety analyses;
- IAs for futility reviewed by the IDMC;
- Primary analysis;
- Final analysis.

#### 4.1. IDMC SAFETY ANALYSES

An IDMC will monitor ongoing data to ensure patient well-being and safety as well as study integrity. The IDMC will be asked to make recommendations to the joint steering committee (JSC) regarding early termination or modification of the evaluation of a candidate agent.

The JSC will evaluate the IDMC recommendation(s) to make decisions on the candidate agent(s) within the study, and it will provide guidance, advice, and recommendations to the program on relevant clinical issues related to the strategy, implementation, and conduct of the study.

Unless otherwise indicated, definitions and derivations for the IDMC safety analyses will be based on those required for the primary analysis contained in this SAP (refers to Section 4.3). The data cut-off for the first IDMC safety meeting will be 4 weeks after the first patient is randomized into any sub-protocol. Thereafter, the data-cut will be

Version Number: Amendment 1, v1.0 Version Date: 23Apr2021

Master Statistical Analysis Plan

Amgen Inc Master Protocol COV-01 

approximately every 4 weeks. Each sub-protocol other than the one to which the very first patient was randomized to will start to be included in the monthly IDMC safety meetings 4 weeks after the first patient is randomized into the sub-protocol. Safety outputs will be based on the safety analysis set (refer to Section 5.2).

The Biostatistics study team will remain blinded to the IDMC safety analysis results. Once the programs have been produced and validated by the Colombia Biostatistics study team in a blinded fashion, these programs will be sent to Colombia Unblinded statistician, independent from the study team, who will apply the randomization schedule and provide the IDMC members with a set of unblinded outputs. The list of the unblinded personnel (i.e., Unblinded Biostatistics team members as well as recipients of the unblinded results sent by Colombia Unblinded Biostatistician) will be documented in the Unblinding Plan, which will be finalized before the data cutoff for the first IDMC safety analysis.

Refer to the IDMC Charter for more details about the IDMC composition, responsibilities, meeting frequency, list of outputs to be provided, etc.

#### 4.2. INTERIM ANALYSES

Each candidate agent will be evaluated for futility at up to two IAs. For sub-studies under the master protocol, an IA will take place after:

- The appropriate number of primary efficacy endpoint events has occurred (refer to Section 16.5);
- Sponsor authorization of this SAP;
- Sponsor authorization of the analysis sets (refer to Section 5.3);
- Interim or final database lock of each sub-protocol contributing to the shared control group of the candidate agent, as appropriate;
- Interim database lock of the concerned candidate agent (refer to Data Management [DM] Interim Database Lock Plan).

The data cut-off date will be the date when approximately the required number of events is reached for an IA (refer to Section 16.5.1) and the last patient having the event is from the sub-protocol of interest for the IA, because if the last patient with an event is from a sub-protocol other than the one of interest, the patient's treatment arm will automatically be unblinded since those patients can only be included in the shared placebo plus SoC control arm of the sub-protocol of interest. Efficacy outputs will be based on the full analysis set (FAS; refer to Section 5.1) and

PPD


CCI

Amgen Inc Master Protocol COV-01 

include data from patients who have had the opportunity to complete the Day 29 study visit or discontinued from study before or on the IA data cut-off date, whichever occur first, while safety outputs will be based on the safety analysis set (refer to Section 5.2) and include all data included in the database at the time of the interim database lock.

Unless otherwise specified, definitions and derivations for the IAs will be based on those required for the primary analysis contained in this SAP (refers to Section 4.3).

As for the IDMC safety analyses, results of each IA will be reviewed by the IDMC. The IDMC will be asked to make recommendations to the JSC regarding early termination of the evaluation of a candidate agent due to futility based on pre-defined stopping rules (refer to Section 16.5.1).

The JSC will evaluate the IDMC recommendation(s) to make decisions on the candidate agent(s) within the study, and it will provide guidance, advice, and recommendations to the program on relevant clinical issues related to the strategy, implementation, and conduct of the study.

Due to the shared placebo plus SoC treatment arm, both the Biostatistics study team and Colombinded statistician, independent from the study team, will be involved in the monitoring of the overall number of patients having met the primary endpoint of confirmed clinical recovery through Day 29, without re-hospitalization through Day 29 (refer to Section 16.1.1), across a particular candidate agent plus SoC and its contemporaneous shared placebo plus SoC treatment arms to confirm the timing of each IA. Once the programs have been produced and validated by the Biostatistics study team in a blinded fashion, these programs will be sent to Colombinded statistician who will apply the randomization schedule and inform Blinded statistician of the overall number of patients having the event (n) and overall number of patients included in the analysis (N). No results by treatment arm will be generated by the programs and no information by treatment arm will be shared with Blinded statistician (refer to the Unblinding Plan for the list of the unblinded personnel i.e. Colombinded statistician, etc.).

The GO Biostatistics study team will remain blinded to the IA results. Once the programs have been produced and validated by the GO Biostatistics study team in a blinded fashion, these programs will be sent to GO Unblinded statistician, independent from the study team, who will apply the randomization schedule and provide the IDMC members with a set of unblinded outputs. The list of the unblinded personnel (i.e. GO Unblinded Biostatistics team members as well as recipients of the unblinded results sent by GO Unblinded Biostatistician) will be documented in the Unblinding Plan, which will be finalized before the data cut-off for the first IDMC safety analysis.



Refer to the IDMC Charter for more details about the IDMC composition, responsibilities, meeting frequency, list of outputs to be provided, etc.

#### 4.3. PRIMARY ANALYSIS

The primary analysis for a candidate agent will take place after:

- Approximately 350 patients have been randomized to the candidate agent plus SoC active arm of the sub-protocol of interest and approximately 350 patients have been randomized to the shared placebo plus SoC control arm of the sub-protocol of interest (refer to Section 4.5), and last patient randomized into one of these two arms is from the sub-protocol of interest, because if the last randomized patient is from a sub-protocol other than the one of interest, the patient's treatment arm will automatically be unblinded since those patients can only be included in the shared placebo plus SoC control arm of the sub-protocol of interest;
- The last patient randomized to that candidate agent plus SoC treatment arm or its concurrent shared placebo
  plus SoC control arm have had the opportunity to complete the Day 29 study visit or discontinued from study
  before or on the Day 29 study visit;
- Sponsor authorization of this SAP;
- Sponsor authorization of the analysis sets (refer to Section 5.3);
- Interim or final database lock of each sub-protocol contributing to the shared control group of the candidate agent, as applicable;
- Interim database lock of the concerned candidate agent database (refer to DM Interim Database Lock Plan).

The data cut-off date will be the date the last patient completed the Day 29 study visit or discontinued from the study before or on the Day 29 study visit, whichever occurs first.

With the following exception, all planned analyses identified in this SAP will be performed by Biostatistics at the time of the primary analysis of a sub-protocol. The exception is the summary and analysis of the secondary efficacy endpoint incidence of sustained clinical recovery as confirmed by Day 60 (refer to Section 16.2.1.9) which will be performed at the time of the final analysis of a sub-protocol (refer to Section 4.4).

For each sub-protocol, additional outputs to be produced at the time of the primary analysis may be specified in sub-protocol SAPs.

| CCI | | |
|-----|----------------------------------|--------------------------------|
| PPD | Version Number:<br>Version Date: | Amendment 1, v1.0<br>23Apr2021 |
| CCI | | |

Master Statistical Analysis Plan

Amgen Inc Master Protocol COV-01 

The Gold Biostatistics study team will remain blinded to the results of the primary analysis. Once the programs have been produced and validated by the Gold Biostatistics study team in a blinded fashion, these programs will be sent to Gold Unblinded statistician, independent from the study team, who will apply the randomization schedule and provide to a pre-identified and limited number of people within the Sponsor of the concerned subprotocol with a set of unblinded outputs. The list of the unblinded personnel (i.e., Gold Unblinded Biostatistics team members as well as recipients of the unblinded results sent by Gold Unblinded Biostatistician) will be documented in the Unblinding Plan, which will be finalized before the data cut-off for the first IDMC safety analysis.

#### 4.4. FINAL ANALYSIS

The final analysis for a candidate agent will take place after:

- Approximately 350 patients have been randomized to the active arm of the sub-protocol of interest and approximately 350 patients have been randomized to the shared placebo plus SoC control arm of the sub-protocol of interest (refer to Section 4.5), and last patient randomized into one of these two treatment arms is from the sub-protocol of interest, because if the last randomized patient is from a sub-protocol other than the one of interest, the patient's treatment arm will automatically be unblinded since those patients can only be included in the shared placebo plus SoC control arm of the sub-protocol of interest;
- The last patient randomized to that candidate agent plus SoC treatment arm and its concurrent shared placebo
  plus SoC control arm (refer to Section 4.5) have had the opportunity to complete the Day 60 visit or
  discontinued from the study,
- Sponsor authorization of this SAP,
- Interim or final database lock of each sub-protocol contributing to the shared control group of the candidate agent, as applicable;
- Final database lock of the concerned candidate agent.

Unless otherwise specified, definitions and derivations for the final analysis will be based on those required for the primary analysis contained in this SAP (refer to Section 4.3). The outputs to be produced at the time of the final analysis of a sub-protocol are:

• Summary of patient disposition (refer to Section 9.1);

PPD


CCI

- Summary of protocol deviations (refer to Section 9.2)
- Summary of concomitant medications (refer to Section 13);
- Summary and analysis of the incidence of sustained clinical recovery as confirmed by Day 60 (other secondary efficacy endpoint; refer to Section 16.2.3.1);
- Summary of all-cause mortality through Day 60 (additional efficacy endpoint; refer to Section 16.4.3);
- All summaries planned for the AEs (refer to Section 17.1).

For each sub-protocol, additional outputs to be produced at the time of the final analysis may be specified in subprotocol SAPs.

The Biostatistics study team will remain blinded to the results of the final analysis of each subprotocol with the exception of the final analysis of the last sub-protocol reaching this milestone. Once the programs have been produced and validated by the Bollin Biostatistics study team in a blinded fashion, these programs will be sent to Unblinded statistician, independent from the study team, who will apply the randomization schedule and provide to a pre-identified and limited number of people within the Sponsor of the concerned sub-protocol with a set of unblinded outputs. The list of the unblinded personnel (i.e., The list of the unblinded Biostatistics team members as well as recipients of the unblinded results sent by Unblinded Biostatistician) will be documented in the Unblinding Plan, which will be finalized before the data cut-off for the first IDMC safety analysis.

#### 4.5. SELECTION OF THE CONTROL ARM FOR AN ANALYSIS

The subset of the placebo plus SoC group, regardless of which sub-protocol the placebo patient belongs, enrolled concurrently to an active agent with matching inclusion/exclusion criteria will serve as the control arm for the analysis of a candidate agent. An exception to this definition is that if a sub-protocol X is not open at a site for screening, the concurrent placebo from other active sub-protocol(s) at that site will not be eligible for inclusion in the control arm for sub-protocol X. This is because patient's eligibility for sub-protocol X cannot be determined without sub-protocol consent and obtaining consent for a sub-protocol is not possible until that sub-protocol is opened at a site for screening. It is to be noted that a patient randomized to the placebo arm of sub-protocol X taking the candidate agent of sub-protocol Y for another approved indication (based on data collected on the Concomitant Medications page of the eCRF) at the time of randomization will not be eligible for the control arm of the sub-protocol Y.

For each sub-protocol and each site, 'concurrently' is defined as the period starting on the date the site was opened

Version Number: Amendment 1, v1.0 PPD Version Date: 23Apr2021 for screening for the sub-protocol and ending on the date of the last patient randomized into that sub-protocol for an interim, primary, and final analyses. For IDMC safety analyses, the date of the data cut-off will be used in lieu of the date of the last patient randomized into the sub-protocol.

#### 5. ANALYSIS SETS

For purposes of analysis, the analysis sets in this section are defined for all sub-protocols. Specific additional analysis sets may be defined in sub-protocols or their corresponding sub-protocol SAPs.

#### 5.1. FULL ANALYSIS SET

For each sub-protocol, the full analysis set (FAS) will contain all patients who were randomized to the sub-protocol candidate agent plus SoC arm as well as all patients who were randomized to any placebo plus SoC arm included in the control arm of the candidate agent (refer to Section 4.5).

For displays and analyses based on FAS, patients will be classified according to randomized treatment.

#### 5.2. SAFETY ANALYSIS SET

For each sub-protocol, the safety analysis set will contain all patients included in the FAS (refer to Section 5.1) who took at least one dose study drug. If there is any doubt whether a patient was treated or not, he/she will be assumed treated with the study drug for the purposes of analysis.

For analyses and displays based on the safety analysis set, patients will be classified according to the actual treatment received (based on data captured on the interactive web response system [IWRS]). That is, a patient randomized to a placebo plus SoC arm who received at least one dose of the candidate agent during the course of the study will be classified under the candidate agent plus SoC arm and a patient randomized to the candidate agent plus SoC arm who never received the candidate agent will be classified under the control arm.

If a patient randomized to the placebo arm of sub-protocol X is selected for the control arm of sub-protocol Y (refer to Section 4.5) and begins taking the candidate agent of sub-protocol Y for another approved indication after randomization as a concomitant medication (based on data captured on the *Concomitant Medications* page of the eCRF), this patient will still be presented under the control arm of sub-protocol Y for summaries based on the safety analysis set and a listing of all AEs will be provided for such patients, if they exist.

PPD


#### 5.3. PROCESS FOR ANALYSIS SET ASSIGNMENT

The analysis sets that will be used to summarize, analyze, and list the data collected during the course of this study are all defined based on objective criteria only. That is, none of the analysis set definitions included in this SAP contains subjective criteria (e.g., major protocol deviation potentially having an impact on the efficacy data). Hence, the authorization of this SAP will also stand for the agreement and authorization of the inclusion/exclusion of each patient in each of these analysis sets.

If analysis sets defined in a sub-protocol SAP involve subjective criteria, the process for analysis set assignment prior to interim, primary or final database locks will be detailed in the sub-protocol SAPs.

#### 6. GENERAL CONSIDERATIONS

#### 6.1. STUDY DAY

Study day will be calculated from the day of the first dose of the study drug for patients who received at least one dose of study drug and from the day of randomization for randomized patients who were never dosed, and will be used to show start/stop day of assessments and events.

Study day will be computed as follows:

- Study Day = (Date of interest –Date of first dose of study drug/randomization, as appropriate) + 1 if the date of interest is on or after the date of first dose of study drug/randomization, as appropriate;
- Study Day = (Date of interest Date of first dose of study drug/randomization, as appropriate) if the date of interest is prior to the date of first dose of study drug/randomization, as appropriate.

Based on these formula, Study Day 1 will be the day of the first dose of the study drug for patients who received at least one dose of study drug and the day of randomization for randomized patients who were never dosed.

In the situation where the date of interest is partial or missing, Study Day and any corresponding durations will be considered as missing in the analyses and the date of interest will be presented as partial or missing in the listings.


#### **6.2.** BASELINE

Unless otherwise specified, baseline is defined as the last non-missing measurement (including unscheduled measurements) taken prior to the first dose of study drug for patients who received at least one dose of study drug and as the last non-missing measurement (including unscheduled measurements) taken prior to randomization for randomized patients who were never dosed. In the case where the last non-missing measurement and first dose of study drug/randomization dates coincide, time will be considered. If time is not collected, missing or unknown, measurements taken on the same day of the first dose, or same day as randomization for subjects not dosed, will be considered as the baseline measurement unless the assessment was scheduled to be collected post-first dose/post-randomization in the master/sub-protocol (refer to Section 3.2).

For adverse events (AEs) commencing on the date of the first dose of study drug/randomization, time of onset of the AE will be considered when determining if the event was pre-baseline (not treatment-emergent) or post-baseline (treatment-emergent). Medications that are ongoing or commencing on the date of the first dose of study drug/randomization will be considered as concomitant medications (refer to Section 13). Partial or completely missing AE and medication dates will be handled as described in Appendix 1.

# 6.3. UNSCHEDULED VISITS, RETESTS, DISCHARGE, AND EARLY TERMINATION DATA

For by-visit summaries, data recorded at the nominal visit will be presented. That is, unscheduled visits will not be included in by-visit summaries but might contribute to the baseline timepoint (refer to Section 6.2) and/or worst/maximum/minimum post-baseline value, where required (e.g., shift table).

In case of a retest when retest is defined as having a blood sample tested twice, the latest available measurement for that blood sample will be used for the by-visit summaries. In case of a retest when retest is defined as having two blood samples collected on the same day, results from the last blood sample will be used for the by-visit summaries.

Refer to Section 6.4 for the conventions to map discharge and early termination data to protocol-defined visit windows. Discharge and early termination data might also contribute to the worst/maximum/minimum post-baseline value, where required (e.g. shift table).

Listings will include all scheduled, unscheduled, retest, discharge, and early discontinuation data.

PPD


#### **6.4.** WINDOWING CONVENTIONS

Discharge and early termination data will be mapped based on the scheduled Study Day of each scheduled visit with adjusted protocol-defined visit window, as specified in the appropriate sub-protocol schedule of activities (refer to Section 3.2).

If discharge or early termination data are mapped to a scheduled visit for which data from the scheduled visit are also available (i.e., non-missing), the data collected at the scheduled visit will be used in the by-visit summaries. If discharge or early termination data are mapped to a scheduled visit for which data from the scheduled visit are not available (i.e., missing), data from the discharge or early termination visit will be used in the by-visit summaries, as applicable.

#### 6.5. COMMON CALCULATIONS

Change from baseline will be calculated as:

• Change from baseline = Observed value at post-baseline visit – Baseline value

Percent change from baseline will be calculated as:

• Percent change from baseline = (Change from baseline / Baseline value) \* 100

#### 7. STATISTICAL CONSIDERATIONS

For continuous data, descriptive statistics (i.e., n [number of patients with available data], mean, standard deviation [SD], minimum, 25<sup>th</sup> percentile (Q1), median, 75<sup>th</sup> percentile (Q3), and maximum values) will be presented by treatment arm and visit, when applicable.

For categorical data, the number and percentage of patients in each category will be presented by treatment arm and visit, when applicable.

#### 7.1. SAMPLE SIZE CALCULATION

A total of up to 350 patients are planned to be randomized to each candidate agent plus SoC. Simultaneously, patients will be randomized to placebo plus SoC throughout the course of the study. The subset of shared placebo

PPD


Master Statistical Analysis Plan

plus SoC treatment arm, regardless of which sub-protocol the placebo belongs, enrolled concurrently to an active agent with matching inclusion/exclusion criteria will serve as comparator (refer to Section 4.5). The primary efficacy endpoint to compare selected treatment plus SoC to placebo plus SoC included in the control arm will be the time to confirmed clinical recovery through Day 29 i.e., fit for discharged (defined by achieving a score of 6, 7 or 8 on the 8-point ordinal scale for clinical severity status), without re-hospitalization through Day 29 (refer to Section 16.1.1).

Assuming a median time to confirmed clinical recovery of 11 days for patients randomized to a candidate agent plus SoC arm compared with 15 days for those randomized to its concurrent placebo plus SoC arm, 350 patients are needed per arm in order to observe 490 confirmed clinical recovery events between the 2 treatment arms being compared at the primary analysis of a sub-protocol. This sample size will provide approximately 88% power to detect a hazard ratio (HR) of 1.364 for the occurrence of the confirmed clinical recovery events, when comparing each candidate agent plus SoC with their concurrent placebo plus SoC arm, at a one-sided significance level of 0.025.

This sample size will provide the following information about the key secondary efficacy endpoints:

- Assuming the oxygen-free recovery rate at Day 29 is 65% for the concurrent placebo plus SoC arm of a
  candidate agent, a sample size of 350 patients per arm will provide approximately 80% power to detect a 9.7%
  absolute increase in the proportion of patients who have oxygen-free recovery at Day 29 in the candidate agent
  plus SoC arm;
- Assuming 70% of patients randomized to the concurrent placebo plus SoC arm of a candidate agent achieve at least 2-point improvement from baseline on the 8-point ordinal scale or are fit for discharge at Day 29, 350 patients per arm will provide approximately 80% power to detect a 9.2% absolute increase in this proportion with a candidate agent plus SoC arm at Day 29;
- Assuming the all-cause mortality rate through Day 29 is 15% for the concurrent placebo plus SoC arm of a candidate agent, a sample size of 350 patients per arm will provide 80% power to detect an absolute reduction of 6.75% (8.25% rate for the candidate agent plus SoC arm) in the mortality rate by Day 29. Assuming a mortality rate of 15% for the concurrent placebo plus SoC arm of a candidate agent and 19% for the candidate agent plus SoC arm (i.e., an adverse treatment effect of 4%) with a sample size of 350 per arm, the chance to observe a decrease in the mortality rate of at least 1% with a candidate agent plus SoC arm compared to its concurrent placebo plus SoC arm is approximately 4%.

The sample size calculation was performed using EAST 6.5.

| CCI | | |
|-----|----------------------------------|--------------------------------|
| PPD | Version Number:<br>Version Date: | Amendment 1, v1.0<br>23Apr2021 |
| CCI | | |

For a sub-protocol where the primary analysis population is a subset of the randomized population, the sample size may be adjusted as applicable to power the designated primary analysis population as appropriate.

Each candidate agent may be evaluated for futility at up to two IAs (refer to Section 16.5).

#### 7.2. MISSING DATA

Missing efficacy data will be handled as described in Sections 16.1.2, 16.2.2, and 16.3.2 of this SAP.

Missing safety data will not be imputed. Partially or completely missing AE and medication dates will be handled as described in Appendix 1.

#### 7.3. STATISTICAL TESTS

Unless otherwise specified, all statistical tests will be conducted at the two-sided 0.05 significance level at the primary analysis. Confidence Intervals (CIs) will be two-sided with 95% coverage, unless otherwise specified.

#### 7.4. MULTIPLE COMPARISONS/ MULTIPLICITY

No adjustment to control the family-wise type I error over the two IAs and the primary analysis of a candidate agent is needed as both IAs will be for futility only (refer to Section 16.5).

At the time of the primary analysis of each candidate agent, the primary efficacy endpoint will be tested at the 0.05 alpha level. Then, a hierarchical testing procedure will be used to test the three key secondary hypotheses (refer to Section 16.2.3.1). With this approach when a particular null hypothesis is rejected, the alpha allocated to that hypothesis can be reallocated to other hypothesis tests. The hierarchical testing procedure will be implemented in the following order:

- 1. Primary endpoint: Time to confirmed clinical recovery through Day 29, without re-hospitalization through Day 29 (refer to Sections 16.1.1 and 16.1.3);
- 2. Key Secondary endpoint: Incidence of oxygen-free recovery at Day 29 (refer to Sections 16.2.1.1 and 16.2.3.1);
- 3. Key secondary endpoint: Incidence of  $\geq$  2-point improvement from baseline or fit for discharge on the ordinal scale at Day 29 (refer to Sections 16.2.1.2 and 16.2.3.1);



Master Statistical Arialysis Flai

4. Key secondary endpoint: Incidence of all-cause mortality through Day 29 (refer to Sections 16.2.1.3 and 16.2.3.1).

In the hierarchical testing procedure, the formal testing can be performed for a step only when the statistical significance is declared for all the endpoints tested in the previous steps. If the testing sequence is stopped at a particular step, only nominal p-value will be provided for the remaining endpoints in the testing sequence.

Only nominal p-values will be provided for the non-key secondary endpoints and no statistical inference will be performed for the CCI and and safety endpoints.

#### 7.5. MULTICENTER STUDIES

This study will be conducted by multiple investigators at multiple centers. For each sub-protocol, data from all patients included in the candidate agent plus SoC arm will be pooled together in the analyses of the sub-protocol, regardless of the patient's centers. Similarly, data from all patients included in the control arm of the candidate agent will be pooled together in the analyses of the sub-protocol, regardless of the patient's centers.

Statistical analyses will be adjusted for the countries. Subgroup analyses by country might be performed for the primary and key secondary efficacy endpoints (refer to Sections 7.7, 16.1.5, and 16.2.5).

If data are too sparse for at least one country (i.e., less than 10% of FAS patients, regardless of the treatment arm), countries will be pooled into regions based on geographical area (e.g., North America, Latin America, Western Europe, Eastern Europe, and Rest of the World). In that case, statistical analyses will be adjusted for regions instead of countries.

For each sub-protocol, determination of the countries or regions to be included in the statistical models will be finalized in a blinded fashion before a sub-protocol database lock for an IA or Primary Analysis (refer to Sections 4.2 and 4.3) based on emerging data.

# 7.6. ADJUSTMENTS FOR COVARIATES AND FACTORS TO BE INCLUDED IN ANALYSES

The analyses will be adjusted for the following covariates and factors. For details of their inclusion in the models, refer to Sections 16.1.3, 16.2.3, and 16.3.3.

• Baseline value of the concerned endpoint, when applicable;



- Baseline clinical severity score of 2 randomization strata (yes or no), as captured on the IWRS;
- Remdesivir at baseline randomization strata (yes or no), as captured on the IWRS;
- Country (or region; refer to Section 7.5).

Sensitivity analyses replacing the randomization strata as captured in IWRS by the randomization strata as derived based on the data captured on the electronic case report form (eCRF) might be performed if at least 10% of the patients are mis-stratified at the time of randomization for a stratification variable (refer to Section 16.1.4) i.e.,

- Baseline clinical severity score of 2 (yes or no) as captured on the Ordinal Scale for Clinical Severity page of the eCRF;
- Remdesivir use at baseline (yes or no) based on data collected on the *Concomitant Medications* page of the eCRF (i.e., medications that were taken by a patient on the day the patient was randomized to a sub-protocol).

#### 7.7. EXAMINATION OF SUBGROUPS

Subgroup analyses will be conducted as supplementary analyses for the primary and key secondary efficacy endpoints as stated in Sections 16.1.5 and 16.2.5, respectively.

The subgroups are:

- Age (years) at informed consent ( $\ge 18 \le 49, \ge 50 \le 64; \ge 65 \le 84 \text{ or } \ge 85$ );
- Sex (male or female);
- Race (White, Black or African American or Other);
- Ethnicity (Hispanic or Latino or not Hispanic or Latino);
- Country (or region; refer to Section 7.5);
- Obesity co-morbidity at screening (BMI <  $30 \text{ kg/m}^2 \text{ or BMI} \ge 30 \text{ kg/m}^2$ );
- Diabetes co-morbidity at screening (yes or no);
- Cardiovascular disease co-morbidity at screening (yes or no);
- Hypertension co-morbidity at screening (yes or no);

- Chronic lung disease co-morbidity at screening (yes or no);
- Chronic liver disease co-morbidity at screening (yes or no);
- Kidney disease co-morbidity at screening (yes or no);
- Immunosuppressive/Immunocompromise disorder co-morbidity at screening (yes or no);
- Time since hospital admission ( $\leq 5$  days or > 5 days; refer to Section 11.1);
- Baseline clinical severity score of 2 randomization strata (yes or no) as captured on the IWRS;
- Disease severity at baseline (2, 3, 4, or 5) based on the ordinal scale for clinical severity as captured on the *Ordinal Scale for Clinical Severity* page on the eCRF;
- Disease severity score of 2, 3 or 4 (yes or no) at baseline based on the ordinal scale for clinical severity as captured on the *Ordinal Scale for Clinical Severity* page on the eCRF
- Remdesivir use at baseline randomization strata (yes or no) as captured on the IWRS;
- Concomitant use of remdesivir at any time during the period of the endpoint of interest (yes or no) based on collected on the *Concomitant Medications* page of the eCRF (for concomitant use definition, refer to Section 13). The concomitant use of remdesivir at any time during the period of the endpoint of interest in the 'yes' subgroup will be further broken down by duration of concomitant use of remdesivir, where the duration of concomitant use categories (e.g., < x days or ≥ x days) will be determined in a blinded fashion based on emerging data before the interim database lock of a candidate agent primary analysis;
- Dexamethasone use at baseline (yes or no) based on data collected on the *Concomitant Medications* page of the eCRF (i.e., medications that were being taken by a patient on the day the patient was randomized to a subprotocol);
- Concomitant use of dexamethasone at any time during the period of the endpoint of interest (yes or no) based on data collected on the *Concomitant Medications* page of the eCRF (for concomitant use definition, refer to Section 13). The concomitantly use dexamethasone at any time during the period of the endpoint of interest 'yes' subgroup will be further broken down by duration of concomitant use of dexamethasone, where the duration of concomitant use categories (e.g., < x days or ≥ x days) will be determined in a blinded fashion based on emerging data before the interim database lock of a candidate agent primary analysis.

For age subgroups, if data are too sparse for the ' $\geq$  18 -  $\leq$  49' or ' $\geq$  50 -  $\leq$  64' subgroups (i.e., less than 10% of FAS


patients, regardless of the treatment arm), these two subgroups will be pooled together into a ' $\geq$  18 -  $\leq$  64' subgroup. Similarly, if data are too sparse for the ' $\geq$  65 -  $\leq$  84 or ' $\geq$  85' subgroups, these two subgroups will be pooled together in a ' $\geq$  65' subgroup. If even after pooled two subgroups, the resulting ' $\geq$  18 -  $\leq$  64' or ' $\geq$  65' subgroup is still less than 10% of FAS patients, regardless of the treatment arm, only descriptive statistics will be provided for the concerned subgroup.

For race subgroups, if data are too sparse for the 'Black or African American' or 'Other' subgroups (i.e., less than 10% of FAS patients, regardless of the treatment arm), the 'Black or African American' and 'Other' subgroups will be pooled together into a 'Non-White' subgroup. If even after having pooled these two subgroups the number of patients in the resulting 'Non-White' subgroup is still less than 10% of FAS patients, regardless of the treatment arm, only descriptive statistics will be provided for the 'Non-White' subgroup.

For the disease severity at baseline subgroups, if data are too sparse for the subgroups of patients with a disease severity at baseline of 3 or 4 (i.e., less than 10% of FAS patients, regardless of the treatment arm), these two subgroups will be pooled together. If data are too sparse for the subgroup of patients with a disease severity at baseline of 2, pooled 3/4 (if applicable) or 5, only descriptive statistics will be provided for the concerned subgroups. That is, the subgroup of patients with a disease severity at baseline of 2 or 5 will not be pooled with any other subgroup.

For any other subgroups, if data are too sparse (i.e., less than 10% of FAS patients for a subgroup, regardless of the treatment arm), only descriptive statistics will be provided for the concerned subgroups.

Additional subgroups might be defined based on emerging data to explore the impact of medical therapy in COVID-19 with proven efficacy (e.g., vaccine use, other evolving SoC, etc.). The decision to add such subgroups and their definition will be taken in a blinded fashion before the interim database lock of a candidate agent primary analysis based on data captured on the *Concomitant Medications* page of the eCRF.

#### 7.8. SOFTWARE VERSION

All analyses will be conducted using SAS version 9.4.

#### 8. OUTPUT PRESENTATIONS

Appendix 2 shows conventions for presentation of data in outputs.

PPD


CCI

Amgen Inc Master Protocol COV-01

Master Statistical Analysis Plan


The table, figure, and listing (TFL) shells provided with this SAP describe the presentations for each sub-protocol in accordance with this master SAP and therefore, the format and content of the summary tables, figures, and listings to be provided by **CCI** Biostatistics. If a sub-protocol has additional endpoints or analyses, additional TFL shells will be provided with the sub-protocol SAP.

#### 9. DISPOSITION AND WITHDRAWALS

All patients who provide informed consent will be accounted for in this study.

#### 9.1. DISPOSITION

Number and percentages of patients treated, ongoing on study drug, who completed/discontinued early from treatment (including reason for withdrawal), ongoing in study, and who completed/discontinued early from the study (including reason for withdrawal) will be provided overall and by treatment arm based on the FAS. The control arm of a candidate agent (refer to Section 4.5) will be further broken down by sub-protocol. It is to be noted that the number and percentage of patients ongoing on study drug and ongoing in study will be excluded from the summary at the time of the final analysis.

In addition, a Kaplan-Meier curve (product-limit estimate) of time to discontinuation from study, in days, for each treatment arm will be provided along with a summary of the associated statistics including, the 25<sup>th</sup>, 50<sup>th</sup> (median), and 75<sup>th</sup> percentiles, and their corresponding two-sided 95% CIs. The control arm of a candidate agent (refer to Section 4.5) will be further broken down by sub-protocol. Patients who are ongoing in the study at the time of an analysis will be censored at the date of the last contact before or on the date of the data cut-off for the analysis and patients who completed the study will be censored at study completion. The standard errors (SEs) will be computed using the Greenwood's formula, the CI for the median will be calculated according to Brookmeyer and Crowley (1982), and the CIs for the survival function estimates at above mentioned time points will be derived from the Kaplan-Meier estimates using the log-log transformation

Number of patients included and excluded from each analysis set (including reason for exclusion) will be summarized overall and by treatment arm based on the FAS. The control arm of a candidate agent (refer to Section 4.5) will be further broken down by sub-protocol.

Listings for randomization schemes/codes and disposition data will be provided separately.

PPD


CCI

#### 9.1.1. **DERIVATIONS**

 Time to discontinuation from study (days) = (Date of study discontinuation – Date of Study Day 1 [refer to Section 6.1]) + 1

Date of study discontinuation will be captured on the *Disposition* page of the eCRF.

Patients who are ongoing in the study at the time of an analysis will be censored at the date of the last contact before or on the date of the data cut-off for the analysis and patients who completed the study will be censored at study completion.

#### 9.2. PROTOCOL DEVIATIONS

All protocol deviations (critical, major, and minor) will be recorded in the clinical trial management system (CTMS) protocol deviations log for the duration of the study (refer to the Protocol Deviations Management Plan for the definition of critical, major, and minor protocol deviations). Site-level identified protocol deviations will be replicated for all patients ongoing in the study at the site at the time of the protocol deviation and presented in the summary outputs as patient-level protocol deviation.

Number and percentage of patients with critical and major protocol deviations will be provided overall and by treatment arm based on the FAS for each category of protocol deviations specified in the Protocol Deviations Management Plan. The control arm of a candidate agent (refer to Section 4.5) will be further broken down by subprotocol.

A listing of all protocol deviations (critical, major, and minor) will be provided.

#### 10. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

The following demographic and other baseline characteristics will be reported for this study:

- Age (years) in integers, calculated relative to date of consent:
  - As a continuous variable;
  - As a categorical variable ( $\ge 18 \le 49, \ge 50 \le 64, \ge 65 \le 84, \text{ or } \ge 85$ );
- Sex (male or female);



- Childbearing potential for female patients only (yes or no) and reasons if not of childbearing potential;
- Race:
  - American Indian or Alaska Native, Asian, Black or African American, Native Hawaiian or Other Pacific Islanders, White, multiple, not reported, or unknown;
  - o White, Black or African American, others, not reported, or unknown;
- Ethnicity (Hispanic or Latino, not Hispanic or Latino, not reported, or unknown);
- Country;
- Region (if applicable, refer to Section 7.5);
- Height (cm);
- Weight (kg);
- Body Mass Index (BMI) (kg/m<sup>2</sup>);

Demographic and other baseline characteristics will be summarized overall and by treatment arm based on the FAS. The control arm of a candidate agent (refer to Section 4.5) will be further broken down by sub-protocol. No statistical testing will be carried out for any demographic or other baseline characteristic.

Demographic and other baseline characteristics data will be listed.

#### 10.1. DERIVATIONS

BMI, in kg/m<sup>2</sup>, will be calculated as follows:

• BMI  $(kg/m^2)$  = Weight  $(kg)/[Height (m)^2]$ 

#### 11. DISEASE HISTORY

The following disease history endpoints will be summarized overall and by treatment arm based on the FAS. The control arm of a candidate agent (refer to Section 4.5) will be further broken down by sub-protocol.

• Time since onset of first COVID-19 symptom(s) (days) – calculated relative to Study Day 1 (refer to Section



6.1)

- Time since COVID-19 diagnosis (days) calculated relative to Study Day 1;
- Time since hospital admission (days) calculated relative to Study Day 1;
- Patients on supplemental oxygen at Study Day 1 (yes or no);
- Type of supplemental oxygen only for patients receiving supplemental oxygen at Study Day 1;
- Time since start of supplemental oxygen (days) calculated relative to Study Day 1 only for patients on supplemental oxygen at Study Day 1;
- Patients receiving ICU/high dependency unit (HDU)-level care at Study Day 1 (yes or no);
- Time since start of ICU/HDU-level care (days) calculated relative to Study Day 1 only for patients receiving ICU/HDU-level care at Study Day 1;
- Patients on invasive mechanical ventilation at Study Day 1 (yes or no);
- Type of invasive mechanical ventilation at Study Day 1 only for patients on invasive mechanical ventilation at Study Day 1;
- Time since start of invasive mechanical ventilation (days) calculated relative to Study Day 1 only for patients on invasive mechanical ventilation at Study Day 1;
- Patients diagnosed with acute respiratory distress syndrome (ARDS; yes or no);
- Time since ARDS diagnosis (days) calculated related to Study Day 1 only for patients diagnosed with ARDS;
- Patients with or without each of the following COVID-19 symptoms at screening. For each symptom, patients with the symptom will be further broken down by severity (mild, moderate, severe, or unknown):
  - o Cough;
  - o Fever;
  - o Myalgia;
  - o Diarrhea;
  - o Dyspnea;


- o Fatigue/malaise;
- Loss of appetite;
- Loss of smell;
- Loss of taste.
- Baseline clinical severity score (2, 3, 4, or 5, as well as 2 or 3/4/5) as captured on the *Ordinal Scale for Clinical Severity* page of the eCRF;
- NEWS2 total score at baseline;
- Oxygen saturation (SpO<sub>2</sub>; %) at baseline;
- Fraction of Inspired Oxygen (FiO<sub>2</sub>; %) at baseline.

All disease history characteristics will be listed.

#### 11.1. DERIVATIONS

Time since events, in days, will be calculated as follows:

- Time since onset of first COVID-19 symptom(s) (days) = (Date of Study Day 1 [refer to Section 6.1] Date of onset of first COVID-19 symptom[s]); date of onset of COVID-19 symptoms as captured on the *Medical History* page of the eCRF;
- Time since COVID-19 diagnosis (days) = (Date of Study Day 1 Date of COVID-19 diagnosis); date of COVID-19 diagnosis as captured on the *Medical History* page of the eCRF;
- Time since hospital admission (days) = (Date of Study Day 1 Date of hospital admission); where date of hospital admission will be the earliest date of hospital admission captured on the *Hospitalization* page of the eCRF;
- Time since start of supplemental oxygen (days) = (Date of Study Day 1 Date of start of supplemental oxygen) if patient is already on supplemental oxygen at Study Day 1; where the date of start of supplemental oxygen will be earliest date of start of supplemental oxygen as captured on the *Supplemental Oxygen and Mechanical Ventilation* page of the eCRF. That is, time since start of supplemental oxygen will not be computed for patients not on supplemental oxygen at Study Day 1;


- Time since start of ICU/HDU-level care (days) = (Date of Study Day 1 Date of start of ICU/HDU-level care) if patient is already receiving ICU/HDU-level care at Study Day 1; where the date of start of ICU/HDU-level care will be the earliest date of start of ICU/HDU-level care captured on the *Hospitalization* page of the eCRF; That is, time since start of ICU/HDU-level care will not be computed for patients not receiving ICU/HDU-level care at Study Day 1;
- Time since start of invasive mechanical ventilation (days) = (Date of Study Day 1 Date of start of invasive mechanical ventilation) if patient is already on invasive mechanical ventilation at Study Day 1; where the date of start of invasive mechanical ventilation will be the earliest date of start of invasive mechanical ventilation captured on the Supplemental Oxygen and Mechanical Ventilation page of the eCRF. That is, time since start of invasive mechanical ventilation will not be computed for patients not on invasive mechanical ventilation at Study Day 1.
- Time since ARDS diagnosis (days) = (Date of Study Day 1 Date of ARDS diagnosis) if patient was diagnosed with ARDS at screening; where the date of start of ARDS diagnosis as captured on the *Medical History* of the eCRF. That is, time since ARDS will not be computed for patients not already diagnosed with ARDS at screening.

# 12. MEDICAL HISTORY

Medical history is defined as any medical conditions/diseases that started and stopped before screening as well as any medical conditions/diseases that started before screening AND were ongoing at the time of screening.

Medical history will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 23.1 or later and will be summarized by System Organ Class and PT overall and by treatment arm based on the FAS. The control arm of a candidate agent (refer to Section 4.5) will be further broken down by sub-protocol. A patient having more than one medical condition/disease within the same System Organ Class or PT will be counted only once for that System Organ Class or PT. In the summary, System Organ Classes will be sorted in alphabetical order and within each System Organ Class, PTs will be sorted in decreasing order of total frequency.

Additionally, for each of the following COVID-19 comorbidities, the number and percentage of patients, as captured on the *Medical History* page of the eCRF, will be reported overall and by treatment arm based on the FAS. The control arm of a candidate agent (refer to Section 4.5) will be further broken down by sub-protocol.

Any comorbidity, defined as having any of the comorbidities listed below;



- Obesity (refer to Sections 7.7 and 10.1);
- Diabetes;
- Cardiovascular disease;
- Hypertension;
- Chronic lung disease;
- Chronic liver disease;
- Kidney disease;
- Immunosuppressive/immunodeficiency disorder.

# 13. PRIOR AND CONCOMITANT MEDICATIONS

All medications collected on the Concomitant Medications page of the eCRF will be classified as either:

• Prior medications, defined as any medication that started and stopped prior to the date of Study Day 1 (refer to Section 6.1);

or

- Concomitant medications, defined as:
  - Any medication that started before the date of Study Day 1 AND ended on or after the date of Study Day 1, or were ongoing at that time;
  - O Any medication that started on or after the date of Study Day 1.

Partially or completely missing medication start and stop dates will be handled as described in Appendix 1.

All medications will be coded using the World Health Organization (WHO) Drug Global dictionary, version September 2020 B3 or later.

Concomitant medications will be summarized by Anatomical Therapeutic Class (ATC) level 2 and preferred drug name overall and by treatment arm based on the FAS. A patient having more than one medication within the same ATC level 2 or preferred drug name will be counted only once for that ATC level 2 or preferred drug name. Further,



for each sub-protocol, separate summaries will also be presented for patients randomized to the sub-protocol placebo plus SoC treatment group.

Additionally, the number and percentages of patients receiving following medications of interest will be summarized overall and by treatment arm based on the FAS. For each sub-protocol, summaries will also be presented for the subset of patients randomized to the Placebo to the candidate agent plus SoC treatment group of the sub-protocol.

- Remdesivir use at baseline (yes or no) based on data collected on the *Concomitant Medications* page of the eCRF (i.e., medications that were being taken by a patient on the day the patient was randomized to a subprotocol);
- Concomitant use of remdesivir at any time during the period of the analysis being performed (yes or no; refer to Section 7.7);
- Dexamethasone use at baseline (yes or no) based on data collected on the *Concomitant Medications* page of the eCRF (i.e., medications that were being taken by a patient on the day the patient was randomized to a subprotocol);
- Concomitant use of dexamethasone at any time during the period of the analysis being performed (yes or no; refer to Section 7.7);
- Steroid use at baseline (yes or no) based on data collected on the *Concomitant Medications* page of the eCRF (i.e., medications that were being taken by a patient on the day the patient was randomized to a sub-protocol);
- Concomitant steroid use at any time during the period of the analysis being performed (yes or no; refer to Section 7.7).

All medications (prior and concomitant) will be listed.

# 14. EXPOSURE TO STUDY DRUG

Each candidate agent included within the study will have a sub-protocol that will provide details of that treatment, including route and mode of administration, dose, dosage regimen, and duration of treatment. The derivations for study drug exposure as well as summaries and analyses of exposure are therefore not covered in this master protocol SAP but will be covered in the SAP for each sub-protocol.



# 15. COMPLIANCE WITH STUDY DRUG

Similar to study drug exposure, derivations of compliance to study drug as well as summaries and analyses of study drug compliance, are not covered in this master protocol SAP, but will be covered in the SAP for each sub-protocol.

## 16. EFFICACY ENDPOINTS

Unless otherwise indicated, all efficacy summaries and figures will be presented by treatment arm and visit, when appropriate, based on the FAS. Listings will be provided for all efficacy data.

## 16.1. PRIMARY EFFICACY

Unless otherwise indicated, all efficacy summaries and analyses will be presented based on the FAS.

# 16.1.1. TIME TO CONFIRMED CLINICAL RECOVERY THROUGH DAY 29, WITHOUT RE-HOSPITALIZATION THROUGH DAY 29

The primary efficacy endpoint is the time to confirmed clinical recovery through Day 29, i.e., fit for discharge (defined by achieving a score of 6, 7, or 8 on the 8-point ordinal scale for clinical severity), without being rehospitalized through Day 29.

It is to be noted that:

- The re-hospitalization-free requirement does not apply to patients who achieved an ordinal scale score of 6 that were never discharged from the hospital before Day 29. For such patients, the re-hospitalization-free requirement is superseded by not having a subsequent worsening on the ordinal scale score (i.e., a score < 6 on the ordinal scale for clinical severity) that would remain until Day 29;
- Patients achieving a score of 7 on the ordinal scale for clinical severity discharged to hospice care will be considered as not fit for discharge in the analysis.

The ordinal scale for clinical severity is as follows:

- 1. Death;
- 2. Hospitalized, on invasive mechanical ventilation or ECMO;
- 3. Hospitalized, on non-invasive ventilation or high-flow oxygen devices;



- 4. Hospitalized, requiring supplemental oxygen;
- 5. Hospitalized, not requiring supplemental oxygen, requiring ongoing medical care (COVID-19 related or otherwise);
- 6. Hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care;
- 7. Not hospitalized, limitation on activities and/or requiring home oxygen;
- 8. Not hospitalized, no limitations on activities.

Time to confirmed clinical recovery through Day 29, without re-hospitalization through Day 29, will be measured in days from the date of Study Day 1 (refer to Section 6.1):

• Time to confirmed clinical recovery through Day 29, without re-hospitalization through Day 29 (days) = (Date of event – Date of Study Day) + 1

Refer to Section 6.1 for the definition of Study Day 1.

The following algorithm will be followed to determine if a patient met the event (i.e., confirmed clinical recovery through Day 29, without rehospitalization through Day 29) or should be censored:

- 1. First, the patient's alive status by Day 29 will be verified as per data collected on the *Death Details* page of the eCRF. If the patient died before or on Day 29, he/she will be censored at Day 29. If the patient has not died by Day 29, then go to step 2;
- 2. Second, the patient's study discontinuation status by Day 29 will be verified as per data collected on the *Disposition* page of the eCRF. If the patient discontinued from the study before or on Day 29, he/she will be censored at date of discontinuation from study. If the patient was still ongoing in the study at Day 29, then go to step 3;
- 3. Last, it will be verified if a patient had a score of 6, 7 or 8 on the 8-point ordinal scale (as captured on the *Ordinal Scale for Clinical Severity* page of the eCRF) before or on Day 29:
  - a. For patients who had a score of 6 on the 8-point ordinal scale and were never discharged from the hospital before Day 29, it will be checked if patient worsened on the 8-point ordinal scale (i.e., had a score < 6) before or on Day 29:
    - i. If so (i.e., patient worsened) and patient never subsequently re-reached a score of 6 before or on Day 29, the patient will be censored at Day 29;
    - ii. If so (i.e., patient worsened) but patient subsequently re-reached a score of 6 before or on

Day 29, the patient will be considered as having the event and the date of the event will be the earliest date on which the patient re-reached a score of 6;

- iii. If not (i.e., patient did not worsen), the patient will be considered as having the event and the date of the event will be the earliest date on which the patient had a score of 6 before or on Day 29;
- b. For patients who had a score of 7 on the 8-point ordinal scale, it will first be verified if patient was discharged to hospice care as per data captured on the *Hospitalization* page of the eCRF.
  - i. If so (i.e., patient was discharged to hospice care), the patient will be considered as not fit for discharge and will be censored at Day 29;
  - ii. If not (i.e., patient was discharged, but not to hospice care), then go to step c.
- c. For patients who had a score of 7 (discharged, but not to hospice care) or 8 on the 8-point ordinal scale, it will be verified if patient was re-hospitalized before or on Day 29 as per data captured on the *Hospitalization* page of the eCRF. To do so, it will be checked if a patient had at least one record where the hospitalization start date is after the earliest date on which the patient had a score of 7 or 8 but before or on Day 29.
  - i. If so (i.e., patient was re-hospitalized), the patient will be censored at Day 29;
  - ii. If not (i.e., patient was not re-hospitalized), the patient will be considered as having the event and the date of the event will be the earliest date on which patient had a score ≥ 6 before or on Day 29;
- d. Patients who never had a score of 6, 7 or 8 on the 8-point ordinal scale, did not discontinue from the study or died before or on Day 29 will be censored at Day 29

Refer to Figure 2 for a schematic of the primary endpoint determination of date of event and censoring.

Figure 2 Schematic of Determination of Primary Efficacy Endpoint Date of Event or Censoring



\* For patients who had a score of 6, worsened, *re*-reached a score of 6, and were never discharged from the hospital before or on Day 29, earliest date on which the patient *re*-reached a score of 6.




#### 16.1.2. MISSING DATA IMPUTATION METHOD FOR PRIMARY EFFICACY ENDPOINT

For the time to confirmed clinical recovery (days) through Day 29, without re-hospitalization through Day 29, missing ordinal scale for clinical severity scores and missing hospitalization data will not be imputed before applying the censoring rules for the main analysis of the primary efficacy endpoint (refer to Section 16.1.1).

#### 16.1.3. MAIN ANALYSIS OF PRIMARY EFFICACY ENDPOINT

For the time to confirmed clinical recovery through Day 29, without re-hospitalization through Day 29, as defined in Section 16.1.1, the number and percentage of patients with and without the event will be presented by randomized treatment arm. For patients who did not meet the event, the main reason for censoring (refer to Section 16.1.1) will be summarized similarly.

Kaplan-Meier curves (product-limit estimate) will be provided by treatment arm for the time to confirmed clinical recovery though Day 29, without re-hospitalization through Day 29. Kaplan-Meier estimate of the time to confirmed clinical recovery through Day 29, without re-hospitalization through Day 29, in days, will be provided at the 25<sup>th</sup>, 50<sup>th</sup> (median), and 75<sup>th</sup> percentiles time along with their corresponding two-sided 95% CIs. The estimates of the SEs will be computed using the Greenwood's formula, the CI for the median will be calculated according to Brookmeyer and Crowley (1982), and the CIs for the survival function estimates at above mentioned time points will be derived from the Kaplan-Meier estimates using the log-log transformation. Kaplan-Meier estimates of the probability of having the event will also be provided at Day 29 along with the number of patients with the event and the number of patients at risk at that time.

The difference between a candidate agent plus SoC arm and its control arm will be compared using a stratified log-rank test. The stratification factor will be the baseline clinical severity of 2 on the 8-point ordinal scale (yes or no) stratification variable, remdesivir use at baseline (yes or no) stratification variable, both as captured on the IWRS, and country (region; refer to Section 7.5). The p-value associated with the stratified log-rank test statistic will be provided and compared at the two-sided 0.05 alpha level at the time of the primary analysis of a candidate agent. The p-value will also be compared to the specified boundaries at the IAs for futility in order to serve as guidance for the IDMC to make recommendations based on the totality of available information at the time of the IAs (refer to Section 16.5).

Additionally, a Cox proportional hazards model will be performed including the baseline clinical severity of 2 on the 8-point ordinal scale (yes or no) stratification variable, remdesivir use at baseline (yes or no) stratification variable, both as captured on the IWRS, country (region), and treatment arm as factors. Ties will be handled using the exact

Version Number: Amendment 1, v1.0 Version Date: 23Apr2021

method. The HR (candidate agent plus SoC vs. placebo plus SoC) and corresponding two-sided 95% CI will be provided.

For the methods to control the overall alpha level of a sub-protocol at the two-sided 0.05 level, refer to Section 7.4.

#### 16.1.4. SENSITIVITY ANALYSES FOR PRIMARY EFFICACY ENDPOINT

The following sensitivity analyses to the main analysis of the primary efficacy endpoint will be performed:

- Sensitivity to stratification variables: The main analysis to the primary efficacy endpoint (refer to Section 16.1.3) may be repeated but stratification variables as derived based on the eCRF data (refer to Section 7.6) will be included in the model instead of the stratification variables as captured on the IWRS. This analysis will be performed only if at least 10% of patients are mis-stratified at the time of randomization for a stratification variable;
- Sensitivity to censoring assumptions #1: The main analysis of the primary efficacy endpoint will be repeated but patients who discontinued early from the study before or on Day 29 will be censored at Day 29;
- Sensitivity to censoring assumptions #2: The main analysis of the primary efficacy endpoint will be repeated but, for patients who discontinued early from the study before or on Day 29, the last patients' known event status will be carried forward to Day 29 before applying the censoring rules for the main analysis of the primary efficacy endpoint (refer to Section 16.1.1).
- Sensitivity to censoring assumptions #3: The primary analysis assumes that censoring is at random (CAR) for patients who discontinued early from the study before or on Day 29 (refer to Section 16.1.3). For this sensitivity analysis, the time to event (refer to Section 16.1.1) will be imputed only for these patients using a model that assumes censoring not at random (CNAR). The model will assume that these patients would have hazard following discontinuation from study that is reduced by some factor delta ( $\delta$ ) compared with hazard of remaining patients in their group who have similar key baseline characteristics (Lipkovich et al, 2016), where reduced hazard rate indicates a longer time to event (confirmed clinical recovery through Day 29, without rehospitalization through Day 29). In order to stress-test the assumption of CAR with an assumption that is less favorable to a candidate agent plus SoC treatment arm, a  $\delta$  < 1 will be used for the candidate agent plus SoC treatment arm while a  $\delta$  = 1 will be used for the concurrent shared placebo plus SoC control arm as  $\delta$  = 1, which corresponds to the CAR assumption.

Multiple imputation method using covariates-adjusted and delta-adjusted piecewise exponential survival model



Amgen Inc Master Protocol COV-01 

Master Statistical Analysis Plan

as suggested in Lipkovich et al, 2016, will be used as the imputation method separately for each treatment arm. For each sub-protocol, the prior distribution and pieces used in this covariates-adjusted and delta-adjusted piecewise exponential survival model will be determined in a blinded fashion prior to the DBL for a sub-protocol Primary Analysis. The model will include the baseline clinical severity of 2 on the 8-point ordinal scale stratification variable (yes or no), remdesivir use at baseline stratification variable (yes or no), both as captured on the IWRS, and country (region; refer to Section 7.5) as covariates.

If the imputed event time exceeds Day 29, the patient will be censored at Day 29. Multiple imputation (MI) method will be used where 100 imputed datasets will be generated using above model and a seed of 2102.

Each of the multiply-imputed datasets will then be analyzed using the same stratified log-rank test and Cox regression model as for the main analysis to the primary efficacy endpoint (refer to Section 16.1.3). The survival distribution quartiles (25<sup>th</sup>, 50<sup>th</sup> [median], and 75<sup>th</sup> percentiles), log-rank statistics, and hazard ratios will be combined as suggested in Moscovici and Ratitch, 2017. The combined statistics and p-value associated with the combined log-rank statistic will be presented.

A tipping point analysis will be implemented where the above described MI will first be performed using a  $\delta$  = 0.95 for the candidate agent plus SoC treatment arm and then repeated but decreasing the  $\delta$ -adjustment applied to the candidate agent plus SoC treatment arm gradually by reduction of 0.05 (i.e., 0.95, 0.90, 0.85, etc.) until the study conclusion is not significant anymore. For each of these analyses, the  $\delta$  used for the concurrent shared placebo plus SoC control arm will always remain 1. The  $\delta$  when the study conclusion becomes non-significant will be referred to as the tipping point.

Additional sensitivity analyses might be specified in the sub-protocol SAPs.

## 16.1.5. SUPPLEMENTARY ANALYSES FOR PRIMARY EFFICACY ENDPOINT

The following supplementary analyses to the main analysis of the primary efficacy endpoint will be performed:

- The main analysis to the primary efficacy endpoint will be repeated (refer to Section 16.1.3) but without country (region; refer to Section 7.5) included as stratification variable;
- The main analysis of the primary efficacy endpoint will be repeated but without the requirement for follow-up confirmation. That is, for this analysis, patients will be considered as having met the event as soon as they reach a score of 6, 7 or 8 on the 8-point ordinal scale, regardless of if they subsequently worsened or were rehospitalized before or on Day 29, exception of patients with a score of 7 discharged to hospice care who will

| CCI | | |
|-----|----------------------------------|--------------------------------|
| PPD | Version Number:<br>Version Date: | Amendment 1, v1.0<br>23Apr2021 |
| CCI | | |

still be considered as not having the event;

• The main analysis of the primary efficacy endpoint will be repeated for each subgroup defined in Section 7.7. For subgroups corresponding to one of the factors included in the main model, the corresponding factor will be excluded from the model. For example, the remdesivir use at baseline (yes/no) stratification variable as captured on the IWRS will not be included in the model for the analysis of the patients who received remdesivir at randomization as captured on the IWRS subgroup, and analysis of the patients who did not receive remdesivir at randomization as captured on the IWRS subgroup.

# 16.2. SECONDARY EFFICACY

## 16.2.1. SECONDARY EFFICACY ENDPOINTS

#### 16.2.1.1. Incidence of Patients with Oxygen-Free Recovery at Day 29

The first key secondary efficacy endpoint is the incidence of patients with oxygen-free recovery at Day 29, defined as the proportion of patients who were alive, discharged, and not receiving supplemental oxygen at Day 29.

- 1. The alive status of a patient at Day 29 (yes or no) will be determined as follows based on data captured on the *Death Details* page of the eCRF: patients who died before or on Day 29 will be considered as not being alive at Day 29 while patients without any data captured on this page of the eCRF before or on Day 29 but with some data captured on any other page of the eCRF on or after Day 29 will be considered to be alive at Day 29;
- 2. The patient's discharge status (yes or no) at Day 29 will be established as follows based on data collected on the *Ordinal Scale for Clinical Severity* page of the eCRF: a patient will be considered as being discharged at Day 29 if 1) their ordinal scale score is 7 at Day 29 and patient was not discharged to hospice care or 2) their ordinal scale score is 8 at Day 29. Discharge to hospice care status will be verified based on data collected on the *Hospitalization* page of the eCRF. To do so, the outcome of the hospitalization record with the latest stop date before or on Day 29 will be examined. The hospitalization outcome of that record should not be 'Home: Hospice Care' or 'Hospice Medical Facility' for a patient with an ordinal scale score of 7 at Day 29 to be considered as discharged at that time. Patients who discontinued early from study before Day 29 will be considered as having a missing discharged status at Day 29;
- 3. The patient's oxygen-free status (yes or no) at Day 29 will be determined as follows: data collected on the



Supplemental Oxygen and Mechanical Ventilation page of the eCRF will be examined to verify if the patient has a record where the start date of supplemental oxygen/mechanical ventilation is before or on Day 29 and stop date of supplemental oxygen/mechanical ventilation is after Day 29\* or is ongoing at Day 29. Patients without such record will be considered as being oxygen-free at Day 29 while patient with such record will be considered as being not oxygen-free at Day 29. Patients who discontinued early from study before Day 29 will be considered as having a missing oxygen-free status at Day 29.

\* That is, patients who stopped receiving supplemental oxygen/mechanical ventilation on Day 29 will be considered as being oxygen-free at Day 29.

All three criteria (alive, discharged, and not receiving supplemental oxygen at Day 29) must be fulfilled for a patient to be considered as having an oxygen-free recovery at Day 29. That is, as soon as a patient does not fulfill at least one of the three criteria, he/she will be considered as not having an oxygen-free recovery at Day 29, regardless of the status of the other criteria. Should the status of one of the three criteria be missing while the two other criteria are fulfilled or missing, patients' oxygen-free recovery at Day 29 will be considered as missing.

| Scenario | Alive at Day 29<br>(as per step 1) | Discharge at Day 29 (as per step 2) | Oxygen-free at Day 29 (as per step 3) | Oxygen-free Recovery at Day 29 |
|---|---|---|---|---|
| 1 | Alive | Yes | Yes | Yes |
| 2 | Dead | Yes, No, Missing | Yes, No, Missing | No |
| 3 | Alive, Dead, Missing | No | Yes, No, Missing | No |
| 4 | Alive, Dead, Missing | Yes, No, Missing | No | No |
| 5 | Missing | Yes, Missing | Yes, Missing | Missing |
| 6 | Alive, Missing | Missing | Yes, Missing | Missing |
| 7 | Alive, Missing | Yes, Missing | Missing | Missing |

Refer to Section 16.2.2.1 for handling of missing oxygen-free recovery at Day 29 status.

# 16.2.1.2. Incidence of Patients with ≥ 2-point Improvement from Baseline or Fit for Discharge on the Ordinal Scale at Day 29

The second key secondary efficacy endpoint is the incidence of patients with  $\geq$  2-point improvement from baseline or fit for discharge on the 8-point ordinal scale for clinical severity (refer to Section 16.1.1) at Day 29, where fit for discharge is defined as having a score of 6, 7 or 8 on the ordinal scale for clinical severity. Patients with an ordinal scale score of 7 must not have been discharged to hospice care to be considered as fit for discharge.

By endpoint definition, patients with an ordinal scale score of 6, 7 (but not discharged to hospice care) or 8 at Day 29 will be considered as having met the event (yes) at Day 29, regardless of their change from baseline in ordinal



scale score, while patients with a score of 7 discharged to hospice care will be considered as not having met the event, also regardless of their change from baseline in ordinal scale score. For patients hospitalized and not considered as fit for discharge at Day 29 i.e., patients with an ordinal scale score < 6, the ' $\geq$  2-point improvement from baseline' requirement (yes or no) will be established based on the patient's change from baseline in the ordinal scale at Day 29, where change from baseline will be computed as defined in Section 6.5.

Refer to Section 16.2.2.1 for handling of missing  $\geq$  2-point improvement from baseline or fit for discharge on the 8-point ordinal scale for clinical severity status.

#### 16.2.1.3. Incidence of All-Cause Mortality through Day 29

The third key secondary efficacy endpoint is the incidence of all-cause mortality through Day 29, defined as the proportion of patients having died due to any cause before or on Day 29. Patients' alive/death status by Day 29 will be determined based on data captured on the *Death Details* page of the eCRF. If a patient does not have any data captured on the *Death Details* page of the eCRF by Day 29 but his/her 'subject status' captured on the *Contact* page of the eCRF at Day 29 is alive or he/she had some data captured on any other page of the eCRF on or after Day 29, he/she will be considered alive on Day 29.

Refer to Section 16.2.2.1 for handling of missing alive/death through Day 29 status.

# 16.2.1.4. Distribution of Patients across the Categories of the 8-point Ordinal Scale for Clinical Severity at Days 8, 15, and 29

An 'other secondary efficacy endpoint' is the distribution of patients across the categories of the 8-point ordinal scale for clinical severity at Days 8, 15, and 29 i.e., the proportion of patients in each category of the 8-point ordinal scale for clinical severity at Days 8, 15, and 29. It is to be noted that patients with a score of 7 discharged to hospice care will be pooled with patients with a score of 1 (death) for this 'other secondary efficacy endpoint'.

Refer to Section 16.1.1 for the description of the 8-point ordinal scale and to Section 16.2.2.1 for handling of missing ordinal scale scores.

#### 16.2.1.5. Worst Post-Baseline Score on 8-point Ordinal Scale from Baseline to Day 29

An 'other secondary efficacy endpoint' is the worst post-baseline score (lower scores are worse) through Day 29 in the 8-point ordinal scale (refer to Section 16.1.1), derived from all scores recorded after baseline up to and including Day 29. It is to be noted that patients with a score of 7 discharged to hospice care will be considered as having a


score of 1 (death) instead of a score of 7 for this 'other secondary efficacy endpoint.

Refer to Section 16.2.2.2 for handling of missing ordinal scale scores.

#### 16.2.1.6. Number of ICU Days from Day 1 through Day 29

An 'other secondary efficacy endpoint' is the number of ICU days from Day 1 through Day 29. This endpoint will be considered as an ordinal endpoint.

For each patient, the number of ICU days from Day 1 through Day 29 will be derived based on the sum of the duration of any episodes of ICU admission between Day 1 and Day 29, inclusively, for patients who were alive on Day 29. Episodes of ICU admission will be identified based on data recorded on the *Hospitalization* page of the eCRF, where *Hospitalization Status* is recorded as *ICU/HDU*. For patients who were discharged to hospice care or died before or on Day 29, the number of ICU days from Day 1 through Day 29 will be set to 30 (worst possible scenario).

The duration, in days, of an episode of ICU admission will be derived as follows:

• Duration of an episode of ICU admission (days) = (Date of ICU discharge – Date of ICU admission) + 1

If the start date of an episode of ICU admission is prior to Day 1, it will be set to the date of Study Day 1 (refer to Section 6.1) when deriving ICU duration for that episode.

If an episode of ICU admission is ongoing at Day 29 or at the time of analysis, the stop date of the admission will be set to the minimum of:

- The start date of any subsequent ICU admission;
- Day 29;
- The data cut-off date for the analysis.

If there are any overlapping dates of ICU admission, a Day will only be counted once when deriving the overall number of ICU days for a patient. For example, if a patient has a record where the start and stop Study Days of the ICU/HDU admission are Day 3 and Day 10, respectively, and another record where the start and stop Study Days of ICU/HDU admission are Day 9 and Day 12, respectively, Days 9 and 10 will be counted only once in the overall number of ICU days for that patient.

Refer to Section 16.2.2.2 for handling of missing number of ICU days from Day 1 through Day 29.



#### 16.2.1.7. Number of Invasive Mechanical Ventilator Days from Day 1 through Day 29

For each patient, the 'other secondary efficacy endpoint' of the number of invasive mechanical ventilator days from Day 1 through Day 29, inclusively, will be considered as an ordinal endpoint and derived similarly to the number of ICU days from Day 1 through Day 29 (refer to Section 16.2.1.6) but using the data collected on the *Supplemental Oxygen and Mechanical Ventilation* page of the eCRF where *Type of supplemental oxygen* is recorded as *Invasive Mechanical Ventilation*.

Refer to Section 16.2.2.2 for handling of missing number of invasive mechanical ventilation days from Day 1 through Day 29.

#### 16.2.1.8. Incidence of Patients with Clinical Recovery by Days 8, 15, and 29

An 'other secondary efficacy endpoint' is the incidence of patients with clinical recovery at Days 8, 15, and 29, defined as the proportion of patients being fit for discharge (i.e., patients achieving a score of 6, 7, or 8 on the 8-point ordinal scale for clinical severity; refer to Section 16.1.1) at Days 8, 15, and 29, respectively, as per data recorded on the *Ordinal Scale for Clinical Severity* page of the eCRF. It is to be noted that patients with a score of 7 discharged to hospice care will not be considered as being fit for discharge for this 'other secondary efficacy endpoint'.

Refer to Section 16.2.2.1 for handling of missing clinical recovery status by Days 8, 15, and 29.

# 16.2.1.9. Incidence of Patients with Sustained Clinical Recovery as Confirmed by Day 60 Follow-up

An 'other secondary efficacy endpoint' is the incidence of patients with sustained clinical recovery as confirmed by Day 60 follow-up, defined as the proportion of patients considered as being fit for discharge (i.e., achieving a score of 6, 7, or 8 on the 8-point ordinal scale for clinical severity) through Day 29, without re-hospitalization by Day 60 (refer to Section 16.1.1), as per the *Ordinal Scale for Clinical Severity* and *Hospitalization* pages of the eCRF. It is to be noted that patients with a score of 7 discharged to hospice care before or on Day 29 will not be considered as being fit for discharge for this 'other secondary efficacy endpoint'.

Similarly to the primary efficacy endpoint, patients achieving a score of 6 on the ordinal scale for clinical severity before or on Day 29 will be considered as having sustained clinical recovery if they have no worsening of their ordinal scale score by Day 60 (i.e., a score < 6 on the ordinal scale for clinical severity) or were discharged from the hospital after Day 29 and were not re-hospitalized by Day 60.

PPD


CCI

Refer to Section 16.2.2.1 for handling of missing sustained clinical recovery as confirmed by Day 60 status.

## 16.2.2. MISSING DATA IMPUTATION METHOD FOR SECONDARY EFFICACY ENDPOINTS

## 16.2.2.1. Binary Endpoints

For the *incidence of oxygen-free recovery at Day 29* endpoint, the algorithm defined in Section 16.2.1.1 will first be applied. Then, patients with a missing oxygen-free recovery status at Day 29 will considered as not having met the event for this key secondary efficacy endpoint.

For the *incidence of patients with*  $\geq$  2-point improvement from baseline or fit for discharge on the ordinal scale at Day 29 endpoint (refer to Section 16.2.1.2), patients with a missing ordinal scale score at Day 29 due to patient's death, discontinuation from study before or on Day 29 or for any other reason (with the following exception) will be considered as not having met the event at Day 29 for that key secondary endpoint. The only exception is for patients with a missing ordinal scale score at Day 29 for which the latest non-missing ordinal scale score before Day 29 was 7 (but not discharge to hospice care) or 8. These patients will be assumed to be fit for discharge at Day 29 and so, as having met the event.

For the *incidence of all-cause mortality through Day 29* endpoint (refer to Section 16.2.1.3), patients with an unknown alive/death status at Day 29 due to discontinuation from study for a reason other than death or missing data will be considered as alive in the analysis, exception of patients for who the last-missing ordinal scale score was 7 and that have been discharged to hospice care before discontinuing from study before Day 29. These patients will be considered as dead at Day 29 for the main analysis of this key secondary efficacy endpoint.

For the *clinical recovery by Day 8* endpoint (refer to Section 16.2.1.8), any patient who died before or on Day 8, discontinued from study before or on Day 8 or with missing clinical recovery status at Day 8 will be considered as not having clinical recovery by Day 8. Missing *clinical recovery by Days 15 and 29* will be handled similarly.

For the *sustained clinical recovery as confirmed by Day 60* follow-up endpoint (refer to Section 16.2.1.9), any patient who died before or on Day 60, discontinued study before Day 60 or with a missing 8-point ordinal scale score at Day 60 will be counted as not having sustained clinical recovery.

## 16.2.2.2. Ordinal Endpoints

Missing *ordinal scale scores* will be imputed as follows for the distribution of patients across the categories of the 8-point ordinal scale for clinical severity at Day 8 endpoints (refer to Section 16.2.1.4):



- Patients who died prior to Day 8 will have a score of 1 used for Day 8;
- For all other occurrences of patient with missing ordinal score at Day 8 (e.g., patients who discontinued from the study before Day 8, etc.), the last non-missing post-baseline ordinal scale score before Day 8 (included data collected at unscheduled post-baseline visits) will be used to impute the missing ordinal scale score at Day 8 exception of patients for who the last non-missing post-baseline ordinal scale score before Day 8 is 7 that were discharged to hospice care. For these patients, the missing ordinal scale score at Day 8 will be imputed to 1.

Missing ordinal scale score at Days 15 and 29 will be imputed similarly.

For the *worst post-baseline score on the 8-point ordinal scale from baseline to Day 29* endpoint(refer to Section 16.2.1.5), patients who have died prior to Day 29 will have their worst post-baseline ordinal scale score from Day 1 to Day 29 set to a score of 1. For patients who are alive at Day 29, no imputation of missing post-baseline ordinal scale scores will be performed. The worst post-baseline ordinal scale score will be identifying among the non-missing post-baseline ordinal scale scores (including data collected at unscheduled post-baseline visits).

For the *number of ICU days and number of invasive mechanical ventilation days* endpoints (refer to Sections 16.2.1.6 and 16.2.1.7, respectively), missing data will not be imputed.

#### 16.2.3. MAIN ANALYSIS OF SECONDARY EFFICACY ENDPOINTS

Refer to Section 7.4 for more information about the hierarchical testing procedure that will be used to test the three key secondary hypotheses. Only nominal p-values will be provided for the non-key secondary endpoints.

#### 16.2.3.1. Binary Endpoints

For the incidence of patients with oxygen-free recovery at Day 29 (refer to Section 16.2.1.1), incidence of patients with ≥ 2-point improvement from baseline or fit for discharge on the ordinal scale at Day 29 (refer to Section 16.2.1.2), incidence of all-cause mortality through Day 29 (refer to Section 16.2.1.3), incidence of patients with clinical recovery at Days 8, 15 and 29 (refer to Section 16.2.1.8), and incidence of patients with sustained clinical recovery as confirmed by Day 60 follow-up (refer to Section 16.2.1.9), the number and percentage of patients with and without the event will be provided by treatment arm. For the incidence of all-cause mortality, primary reason of death will also be summarized by treatment arm.

For each of these endpoints, a logistic regression will be performed to test the difference between a candidate agent plus SoC and placebo plus SoC treatment arms, including the baseline clinical severity of 2 on the 8-point ordinal

PPD


CCI

scale for clinical severity (yes or no) stratification variable, remdesivir use at baseline (yes or no) stratification variable, both as captured on the IWRS, country (region; refer to Section 7.5), and treatment arm as factors. The estimate of the relative risk (risk difference) between the two treatment arms, the corresponding two-sided 95% Wald CI, and the p-value obtained from the logistic regression model will be provided.

The odds ratio (of candidate agent plus SoC vs. placebo plus SoC) for having the event at the specified Day and its two-sided 95% CI will also be presented.

### 16.2.3.2. Ordinal Endpoints

For the incidence of patients in each category of the 8-point ordinal scale for clinical severity at Days 8, 15, and 29 endpoints (refer to Section 16.2.1.4), the number and percentage of patients in each ordinal scale category will be provided at each specified Day for each treatment arm and will be analyzed using a proportional odds model, including the baseline clinical severity of 2 on the 8-point ordinal scale for clinical severity (yes or no) stratification variable, remdesivir use at baseline (yes or no) stratification variable, both as captured on the IWRS, country (region; refer to Section 7.5), and treatment arm as factors.

The odds ratio (candidate agent plus SoC vs. placebo plus SoC) of having a higher score than any given category k of the ordinal scale at Days 8, 15, and 29, their two-sided 95% CI, and associated p-value will be presented for each specified Day, where it is assumed that the odds ratio does not differ depending upon k.

The worst post-baseline score on the 8-point ordinal scale for clinical severity from randomization to Day 29 (refer to Section 16.2.1.5) and each "number of days" endpoint (refer to Sections 16.2.1.6 and 16.2.1.7) will be summarized and analyzed similarly.

Shift tables from baseline to each post-baseline day up to Day 29 as well as to the worst post-baseline score will also be provided for the 8-point ordinal scale for clinical severity.

#### 16.2.4. SENSITIVITY ANALYSES FOR SECONDARY EFFICACY ENDPOINTS

The following sensitivity analyses to the main analysis of each key secondary efficacy endpoint will be performed. No sensitivity analyses will be performed for the non-key secondary efficacy endpoints.

• Sensitivity to stratification variables: The main analysis of each key secondary efficacy endpoint will be repeated but the stratification variables as derived based on the eCRF data (refer to Section 7.6) will be included in the model instead of the stratification variables as captured on the IWRS if at least 10% of patients are mis-



stratified at the time of randomization for a stratification variable.

#### • Sensitivity analysis to missing data assumption #1:

o For the incidence of patients with oxygen-free recovery at Day 29 (refer to Section 16.2.1.1), a multiple imputation approach will be applied to impute the missing oxygen-free recovery status (yes or no) at Day 29 for subjects who discontinued from study before or on Day 29 using a logistic regression including effects for the treatment arm, baseline clinical severity of 2 on the 8-point ordinal scale for clinical severity stratification variable (yes or no), remdesivir use at baseline stratification variable (yes or no), both as captured on the IWRS, and country (or region; refer to Section 7.5). One hundred (100) imputed datasets will be generated using a seed of 2504.

Each imputed dataset will then be analyzed using the same model as for the main analysis of this key secondary efficacy endpoint (refer to Section 16.2.3.1).

The relative risks and parameter estimates for the effects of the logistic regression model and their SEs will then be combined using the Rubin's rule to obtain a combined estimate of the treatment arm effect and its SE, and the associated p-value will be provided. The relative risks and odds ratios will first be log transformed and then combined to obtain a combined relative risk and combined odds ratio, and their associated 95% CI. The combined relative risk and combined odds ratio, and associated 95% CI, will be back-transformed before being displayed;

- o For the incidence of patients with ≥ 2-point improvement from baseline or fit for discharge on the ordinal scale at Day 29 (refer to Section 16.2.1.2), the same sensitivity analysis using multiple imputation as described above as for the key secondary efficacy endpoint of incidence of patients with oxygen-free recovery at Day 29 will be performed for this key secondary efficacy endpoint, but using a seed of 1228:
- For the incidence of all-cause mortality through Day 29 (refer to Section 16.2.1.3), the same sensitivity analysis using multiple imputation as described above as for the key secondary efficacy endpoint of incidence of patients with oxygen-free recovery at Day 29 will be performed for this key secondary efficacy endpoint, but using a seed of 2007.

## • Sensitivity analysis to missing data assumption #2:

For the incidence of all-cause mortality through Day 29, a tipping point analysis will be performed. For patients who discontinued early from the study, all possible combinations of the number of patients



dead or alive at Day 29 will be considered and the main analysis of this key secondary efficacy endpoint will be repeated for each combination.

A dot plot will be produced with number of patients with unknown death status at Day 29 imputed to death for the shared placebo plus SoC treatment arm reported on the x-axis and number of patients with unknown death status at Day 29 imputed to death for the candidate agent plus SoC treatment arm reported on the y-axis, and distinguishing between combination that results in statistically significant treatment effect (a dot is displayed for the combination) vs. not statistically significant treatment effect (no dot is displayed for the combination). The clinical plausibility of the combinations on the boundary will be discussed in the clinical study report (CSR) to evaluate robustness of study conclusions to missing data.

#### 16.2.5. SUPPLEMENTARY ANALYSES FOR SECONDARY EFFICACY ENDPOINTS

The main analysis of each key secondary efficacy endpoint will be repeated for each subgroup defined in Section 7.7. For subgroups corresponding to one of the factors included in the main model, the corresponding factor will be excluded from the model. For example, the remdesivir use at baseline (yes/no) stratification variable, as captured on the IWRS, will not be included in the analysis of the patients who received remdesivir at randomization subgroup, as captured on the IWRS, and analysis of the patients who did not receive remdesivir at randomization subgroup, as captured on the IWRS.

The following supplementary analyses will also be performed for the incidence to all-cause mortality key secondary efficacy endpoint:

- For the incidence of all-cause mortality through Day 29, the time to all-cause death, in days, will be derived as follows:
  - Time to all-cause mortality (days) =

(Date of all-cause death/Date of censoring - Date of Study Day 1 [refer to Section 6.1]) + 1.

The date of death will be taken from data captured on the *Death Details* page of the eCRF.

For patients who were alive on Day 29, time to all cause-mortality will be censored at Day 29. For patients with an unknown alive status at the time of the analysis due to missing data, time to all-cause mortality will be censored at the latest date on which the patient was known to be alive before or on the data cut-off date of the analysis. The last date the patient was known to be alive will be the latest date



Amgen Inc Master Protocol COV-01 

collected on any page of the eCRF. For patients who discontinued from the study before the time of the analysis, time to all-cause mortality will be censored at the date of study discontinuation, as captured on the *Disposition* page of the eCRF.

Number and percentage of patients with and without the event will be presented by randomized treatment arm. For patients who did not meet the event, the main reason for censoring will be summarized similarly.

The incidence of all-cause mortality through Day 29 along with its two-sided 95% CI by treatment arm will then be estimated using Kaplan-Meier survival curves of the time to all-cause mortality. Kaplan-Meier survival curves by treatment arm will also be provided.

The 25<sup>th</sup> percentile, 50<sup>th</sup> percentile (median), and 75<sup>th</sup> percentile of time to all-cause mortality (days) with the corresponding two-sided 95% CIs based on the Kaplan-Meier survival curves (refer to Section 16.2.4) for each treatment arm will also be presented. The estimate of the SEs will be computed using Greenwood's formula, the CI for the median will be calculated according to Brookmeyer and Crowley (1982) and the other CIs will be derived from the Kaplan-Meier estimates using the log-log transformation.

A Cox proportional hazard model will be performed, including the baseline clinical severity of 2 on the 8-point ordinal scale for clinical severity (yes or no), remdesivir use at baseline (yes or no) stratification variables, both as captured on the IWRS, country (region), and treatment arm as factors. Ties will be handled using the exact method. The hazard ratio of the candidate agent plus SoC vs. placebo plus SoC, its associated two-sided 95% CI, and p-value will be provided.

No supplementary analyses will be performed for the non-key secondary efficacy endpoints.

# 16.3. EXPLORATORY EFFICACY

#### 16.3.1. EXPLORATORY EFFICACY ENDPOINTS









Amgen Inc Master Protocol COV-01 

Master Statistical Analysis Plan





CCI

Amgen Inc Master Protocol COV-01 

Master Statistical Analysis Plan



PPD Version Number: Amendment 1, v1.0 Version Date: 23Apr2021

CCI

Amgen Inc Master Protocol COV-01 

Master Statistical Analysis Plan







Master Statistical Analysis Plan  CCI Amendment 1, v1.0 23Apr2021 Version Number: PPD Version Date:

Master Statistical Analysis Plan

 CCI Amendment 1, v1.0 Version Number: PPD Version Date: 23Apr2021

CCI

Amgen Inc Master Protocol COV-01 

Master Statistical Analysis Plan



Master Statistical Analysis Plan



#### 16.3.4. SENSITIVITY ANALYSES FOR EXPLORATORY EFFICACY ENDPOINTS

CCI

#### 16.3.5. SUPPLEMENTARY ANALYSES FOR EXPLORATORY EFFICACY ENDPOINTS

CCI

# 16.4. ADDITIONAL EFFICACY

#### 16.4.1. ADDITIONAL EFFICACY ENDPOINT

#### 16.4.1.1. Incidence of All-Cause Mortality through Day 60

An additional efficacy endpoint is the incidence of all-cause mortality through Day 60, defined as the proportion of patients having died due to any cause before or on Day 60. Patients death before or at Day 60 will be based on data captured on the *Death Details* page of the eCRF.

#### 16.4.2. MISSING DATA IMPUTATION METHOD FOR ADDITIONAL EFFICACY ENDPOINT

Patients with an unknown alive/death status at Day 60 will be considered as alive at Day 60.

#### 16.4.3. ANALYSIS OF ADDITIONAL EFFICACY ENDPOINT

The number and percentage of patients alive and dead through Day 60 (refer to Section 16.4.1.1) along with the two-sided 95% CI for the percentage of patients dead through Day 60 will be provided by treatment arm. Primary reason of death will also be summarized by treatment arm. No statistical inference will be performed for this endpoint but treatment effect estimate (i.e., relative risk, odds ratio) and two-sided 95% CI will be provided.

## 16.4.4. SENSITIVITY ANALYSES FOR ADDITIONAL EFFICACY ENDPOINT

No sensitivity analyses will be performed for the additional efficacy endpoint.

PPD


#### 16.4.5. SUPPLEMENTARY ANALYSES FOR ADDITIONAL EFFICACY ENDPOINT

The time to all-cause death through Day 60, in days, will be derived as follows:

• Time to all-cause mortality through Day 60 (days) =

(Date of death / Date of censoring - Date of Study Day 1 [refer to Section 6.1]) + 1.

The date of death will be taken from data captured on the *Death Details* page of the eCRF.

For patients who were alive or patients with an unknown alive status at the time of the analysis due to missing data, time to all-cause mortality will be censored at the latest date on which the patient was known to be alive before or on Day 60. The last date the patient was known to be alive will be the latest date collected on any page of the eCRF. For patients who discontinued from the study before Day 60, time to all-cause mortality will be censored at the date of study discontinuation, as captured on the *Disposition* page of the eCRF.

Number and percentage of patients with and without the event will be presented by randomized treatment arm. For patients who did not meet the event, the main reason for censoring (refer to Section 16.1.1) will be summarized similarly.

The incidence of all-cause mortality through Day 60 along with its two-sided 95% CI by treatment arm will then be estimated using Kaplan-Meier survival curves of the time to all-cause mortality through Day 60. Kaplan-Meier survival curves by treatment arm will also be provided.

The 25<sup>th</sup> percentile, 50<sup>th</sup> percentile (median), and 75<sup>th</sup> percentile of time to all-cause mortality (days) with the corresponding two-sided 95% CIs based on the Kaplan-Meier survival curves for each treatment arm will be presented. The estimate of the SEs will be computed using Greenwood's formula, the CI for the median will be calculated according to Brookmeyer and Crowley (1982) and the CIs for the survival function estimates at above mentioned time points will be derived from the Kaplan-Meier estimates using the log-log transformation.

Finally, a Cox proportional hazard model will be performed, including the baseline clinical severity of 2 on the 8-point ordinal scale for clinical severity (yes or no), remdesivir use at baseline (yes or no) stratification variables, both as captured on the IWRS, country (region), and treatment arm as factors. Ties will be handled using the exact method. The hazard ratio of the candidate agent plus SoC vs. placebo plus SoC and its associated two-sided 95% CI will be provided.

Version Number: Amendment 1, v1.0 Version Date: 23Apr2021

# 16.5. INTERIM ANALYSIS

## 16.5.1. INTERIM ANALYSIS FOR FUTILITY

Each candidate agent may be evaluated for futility at up to two IAs.

The IAs will be based on analyses of the primary efficacy endpoint (refer to Section 16.1.1), using the analysis methods described in Section 16.1.3.

The IAs are planned at information fractions of approximately 25% and 55% of expected number of confirmed clinical recoveries (refer to Table 1), i.e., after approximately 123 and 270 patients have met the primary endpoint of confirmed clinical recovery on a particular candidate agent plus SoC and its contemporaneous placebo plus SoC, respectively. However, the timing of these IAs may be adjusted due to operational considerations, e.g., actual enrollment rate.

For the IAs, a Pocock beta spending function will be used for non-binding futility boundary specification. This strategy will allow for ineffective agents to be identified early for discontinuation of further evaluation. Assuming no treatment effect for a candidate agent plus SoC arm compared with placebo plus SoC patients included in the control arm of the candidate agent, there is a 49.7% chance that enrolment to this agent is stopped at the first IA and 34.6% chance at the second IA. Under the scenario that treatment has a negative effect on outcome (refer to Table 2), these probabilities become 72.3% and 24.7%, respectively.

The primary analysis for a candidate agent will occur after 350 patients have been randomized to a particular candidate agent plus SoC and have had the opportunity to complete the Day 29 visit, when approximately 490 confirmed clinical recovery events are expected to have been observed in total across the candidate plus SoC arm and placebo plus SoC patients included in the control arm of the candidate agent, unless a candidate agent is stopped early for futility. The final analysis of a candidate agent will occur after all patients randomized to that candidate agent plus Soc and the concurrent placebo plus SoC controls have had the opportunity to complete the Day 60 visit.

Table 1 and Table 2 present a summary of futility incremental probabilities at the first interim and second interim analyses together with Pocock futility boundaries in the scenario of 88.3% estimated power when the IAs occur at information fraction of 25% and 55% of expected number of recoveries, respectively.

Version Number: Amendment 1, v1.0 Version Date: 23Apr2021

Table 1 Summary of Futility Probabilities and Boundaries with 88.3% Power using Pocock Futility Boundaries

| Analysis | Total Number of<br>Events<br>(Information<br>Fraction) | Boundary of<br>Futility,<br>Non-binding<br>(HR) | Boundary of<br>Futility,<br>Non-binding<br>(p-value) | Incremental Probability to Declare Futility under the Null (HR=1) |
|---|---|---|---|---|
| First Interim | 123 (25%) | ≤ 0.998 | 0.503 | 0.497 |
| Second Interim | 270 (55%) | ≤ 1.121 | 0.175 | 0.346 |

HR=hazard ratio.

Assume 1-sided  $\alpha$  of 0.025.

Interim analyses using Pocock futility boundaries at 25% and 55% information fraction.

HR boundaries are translated from p-values, dependent of relative timing, and will be re-calculated for IDMC.

Table 2 Summary of Futility Probabilities and Boundaries with 88.3% Power using Pocock Futility Boundaries for the Negative Treatment Scenario (HR=0.9)

| Analysis | Total Number of<br>Events<br>(Information<br>Fraction) | Boundary of<br>Futility,<br>Non-binding<br>(HR) | Boundary of<br>Futility, Non-<br>binding<br>(p-value) | Incremental Probability to Declare Futility under the Negative Treatment Effect Scenario (HR=0.9) |
|---|---|---|---|---|
| First Interim | 123 (25%) | ≤ 0.998 | 0.503 | 0.723 |
| Second Interim | 270 (55%) | ≤ 1.121 | 0.175 | 0.247 |

HR=hazard ratio.

Assume 1-sided  $\alpha$  of 0.025.

Interim analyses using Pocock futility boundaries at 25% and 55% information fraction.

HR boundaries are translated from p-values, dependent of relative timing, and will be re-calculated for IDMC.

PPD Version Number: Amendment 1, v1.0 Version Date: 23Apr2021

## 17. SAFETY ENDPOINTS

All safety summaries will be presented by treatment arm based on the safety analysis set. Further, for each sub-protocol, separate summaries will also be presented for patients randomized to the placebo plus SoC treatment group of the sub-protocol.

There will be no statistical comparisons between the treatment arms for safety data.

## 17.1. ADVERSE EVENTS

Each AE will be classified as either:

- Prior, defined as any AE that started or worsened in severity on or after the date of signed informed consent but before the first dose of study drug;
- Treatment-emergent, defined as any AE that started or worsened in severity on or after the first dose of study drug.

If time of the first dose of study drug and time of start of AEs are available, then the times will be taken into account for determining TEAEs. Refer to Appendix 1 for handling of partial and completely missing dates for AEs. In the case where it is not possible to define an AE as treatment emergent or not, the AE will be classified by the worst case; i.e. treatment emergent.

AEs will be coded using the MedDRA dictionary, version 23.1 or later. Summaries by System Organ Class and PT will be sorted as follows: System Organ Classes will be sorted in alphabetical order and within each System Organ Class, PTs will be sorted by decreasing order to total frequency.

An overall summary of number and percentage of patients within each of the categories described in the subsections below will be provided by treatment arm. Should a patient experience multiple events within a category, the patient will be counted only once for that category. Additionally, the risk difference of the overall incidence rates of serious TEAEs and overall incidence rates of AESIs (when applicable for a sub-protocol) between treatment and control arms will be presented along with its 95% two-sided Wald CI.

All AEs (prior and TEAE) will be listed.

Version Number: Amendment 1, v1.0 Version Date: 23Apr2021


#### **17.1.1. ALL TEAES**

Number and percentage of patients with at least one TEAE will be presented by System Organ Class and PT. Should a patient experience multiple events within a System Organ Class or PT, the patient will be counted only once for that System Organ Class or PT.

Number and percentage of patients with at least one TEAE will be broken down further separately by maximum severity (CTCAE Grades 1-5), CTCAE Grade ≥3, relationship to study drug (not related and related), and relationship to non-study drug (not related and related).

#### 17.1.1.1. CTC Grading for AEs

Toxicity will be classified as mild (Grade 1), moderate (Grade 2), severe (Grade 3), life-threatening (Grade 4) or fatal (Grade 5) according to the CTCAE, version 5:

https://ctep.cancer.gov/protocoldevelopment/electronic applications/docs/CTCAE v5 Quick Reference 5x7.pdf

Should a patient experience multiple events within a System Organ Class or PT, only the patient's worst CTCAE grade will be counted for that System Organ Class or PT.

#### 17.1.1.2. Relationship to Study Drug, Non-Study Drug, and Study Procedure

Relationship to study drug, relationship to non-study drug, and relationship to study procedure, as indicated by the Investigator, will be classified as unrelated or related.

Should a patient experience multiple events within a System Organ Class or PT, only the patient's worst relationship (i.e., related) will be counted for that System Organ Class or PT.

TEAEs will not be summarized by the relationship to study procedure, but relationship to study procedure will be listed.

#### 17.1.2. FATAL ADVERSE EVENTS

Fatal TEAEs are those events which are recorded as *Fatal* or with a CTCAE grade of 5 on the *Adverse Events* page of the eCRF. A summary of fatal TEAEs by System Organ Class and PT will be prepared.

A listing of all fatal AEs will be provided.




#### 17.1.3. SERIOUS ADVERSE EVENTS

SAEs are those events recorded as *Serious* on the *Adverse Events* page of the eCRF. A summary of serious TEAEs by System Organ Class and PT will be prepared. Should a patient experience multiple events within a System Organ Class or PT, the patient will be counted only once for that System Organ Class or PT.

A listing of all SAEs will be provided

#### 17.1.4. Most Common Non-Serious Adverse Events

Number and percentage of patients with at least one most common non-serious TEAE will be presented by PT, where most common is defined as a PT with at least 5% of patients in at least one treatment arm. Should a patient experience multiple events within a PT, the patient will be counted only once for that PT.

## 17.1.5. TEAES LEADING TO DOSE MODIFICATIONS

TEAEs leading to dose modification are those events recorded with "Action Taken with study treatment" on the Adverse Events pages of the eCRF of any of the following: Dose increased, Dose reduced, Dose rate reduced, or Drug interrupted. A summary of TEAEs leading to dose modification by System Organ Class and PT will be prepared. Should a patient experience multiple events within a System Organ Class or PT, the patient will be counted only once for that System Organ Class or PT.

#### 17.1.6. TEAES LEADING TO DISCONTINUATION OF STUDY TREATMENT

TEAEs leading to permanent discontinuation of study treatment are those events recorded with *Action Taken with study treatment* of *Drug withdrawal* on the *Adverse Events* page of the eCRF. A summary of TEAEs leading to permanent discontinuation of study drug by System Organ Class and PT will be prepared. Should a patient experience multiple events within a System Organ Class or PT, the patient will be counted only once for that System Organ Class or PT.

A listing of all AEs leading to permanent discontinuation of study drug will be provided.

#### 17.1.7. **AESIS**

For applicable sub-protocols, refer to sub-protocol SAP for more details.



## 17.2. LABORATORY EVALUATIONS

A serum or urine pregnancy test will be performed at screening. Hematology, coagulation, and chemistry (including cardiac enzymes and liver function tests) laboratory tests will be performed as per the schedule of events (refer to the example schedule of events in Section 1.3 of the master protocol but note that each sub-protocol will have its own schedule of events).

A list of laboratory tests to be included in the outputs is included in Appendix 5. It is to be noted that additional laboratory tests might be collected in a sub-protocol.

Results of quantitative laboratory tests reported as "< X", i.e. below the lower limit of quantification (BLQ) or "> X", i.e. above the upper limit of quantification (ULQ), will be converted to X for the purpose of quantitative summaries, but will be presented as recorded, i.e. as "< X" or "> X" in the listings. Observed values will then be normalized (refer to Section 17.2.1) before being summarized and changes from baseline will be computed based on the normalized observed values.

The following summaries will be provided by treatment arm for each hematology, coagulation, and chemistry test:

- Observed, change, and percent change from baseline values in Standard International (SI) units by visit (for quantitative tests)
- Box and whisker plots over time in SI units (for selected quantitative tests at IDMC safety data review meetings and IAs only)
- Shift from baseline to the worst post-baseline observed value according to the CTCAE toxicity grades (for quantitative tests with available CTCAE toxicity grades; refer to Section 17.2.2)
- Listing of patients with at least one laboratory observed value meeting a CTCAE toxicity grade ≥ 3 (for quantitative tests with available CTCAE toxicity grades; refer to Section 17.2.2)
- Shifts from baseline to the maximum/minimum post-baseline observed value according to reference range criteria (for quantitative tests without CTCAE toxicity grades; refer to Section 17.2.3)
- Listing of patients with at least one abnormal laboratory observed value outside the reference range criteria (for quantitative tests without CTCAE toxicity grades; refer to Section 17.2.3)
- Maximum post-baseline ALT/AST observed value categorized as < 3 x upper limit of normal (ULN), ≥ 3 to < 5</li>
   x ULN, ≥ 5 to < 10 x ULN or ≥ 10 ULN by maximum post-baseline total bilirubin observed value categorized</li>

PPD Version Number: Amendment 1, v1.0 Version Date: 23Apr2021

as 
$$< 2 \times ULN \text{ or } \ge 2 \times ULN$$

- Scatter plots of the maximum post-baseline observed value in ALT value by the maximum post-baseline observed value in TBL value, both expressed as multiple of ULN
- Scatter plots of the maximum post-baseline observed value in AST value by the maximum post-baseline observed value in TBL value, both expressed as multiple of ULN
- A listing of patients with at least one observed value in ALT value > 3 x ULN, AST value > 3 x ULN or TBL value ≥ 2 x ULN will be provided

#### 17.2.1. LABORATORY NORMALIZATION

If a laboratory test has different reference ranges in the database, observed values of all patients will first be standardized to a common standard unit and then, normalized to a common set of standardized reference range using the location-scale normalization formula (Chuang-Stein, 1992):

$$\bullet \quad y = L_y + (x - L_X) \frac{(U_Y - L_Y)}{(U_X - L_X)}$$

where:

- $\circ$  y = normalized and standardized observed value;
- $\circ$  x = standardized observed value;
- $L_{\rm Y}$  = Lower limit of the reference range chosen to be the common standardized reference range;
- $\circ$  U<sub>Y</sub> = Upper limit of the reference range chosen to be the common standardized reference range;
- o L<sub>X</sub> = Lower limit of the reference range associated with the standardized observed value;
- $\circ$  U<sub>X</sub> = Upper limit of the reference range associated with the standardized observed value.

It is to be noted that the choice of the common standardized reference range is arbitrary.

#### 17.2.2. CTCAE TOXICITY GRADES

Quantitative laboratory tests with available CTCAE toxicity grades will be categorized as follows where higher grades representing a more severe toxicity (refer to Appendix 6 for each test toxicity grade criteria):


- Grade 1 (i.e., mild);
- Grade 2 (i.e., moderate);
- Grade 3 (i.e., severe);
- Grade 4 (i.e., life-threatening);
- Grade 5 (i.e., death).

Although not defined in the CTCAE toxicity grading system, version 5, non-missing laboratory test results not meeting any of the 5 grades defined in the CTCAE toxicity grading system will be categorized as 'No Event' for the purpose of the shift from baseline summaries.

#### 17.2.3. LABORATORY REFERENCE RANGES

Quantitative laboratory tests will be compared with the relevant laboratory reference ranges in SI units and categorized as:

- Low: Below the lower limit of the laboratory reference range
- Normal: Within the laboratory reference range (upper and lower limit included)
- High: Above the upper limit of the laboratory reference range

## 17.3. VITAL SIGNS

The following vital sign parameters will be collected as per the schedule of events (refer to the example schedule of events in Section 1.3 of the master protocol, but note that each sub-protocol will have its own schedule of events):

- Systolic blood pressure (SBP) (mmHg);
- Diastolic blood pressure (DBP) (mmHg);
- Pulse rate (beats per minute [bpm]);
- Oxygen saturation (%);
- FiO<sub>2</sub> (%);



- Respiratory rate (breaths/min);
- Body temperature (°C).

The following summaries will be provided by treatment arm for each vital sign parameter:

- Observed and change from baseline values by visit;
- Number and percentages of patients with at least one markedly abnormal post-baseline observed value/change from baseline (refer to Section 17.3.1);
- Listing of patients with at least one markedly abnormal observed value/change from baseline (refer to Section 17.3.1).

## 17.3.1. VITAL SIGNS MARKEDLY ABNORMAL CRITERIA

Markedly abnormal vital sign observed values and/or change from baseline will be identified in accordance with the following predefined markedly abnormal criteria:

| Variable | Unit | Low | High |
|---|---|---|---|
| SBP | mmHg | ≤ 90 mmHg AND change from Baseline ≤ -20 mmHg | ≥ 180 mmHg AND change from Baseline ≥ 20 mmHg |
| DBP | mmHg | ≤ 50 mmHg AND change from Baseline ≤ -15 mmHg | ≥ 105 mmHg AND change from Baseline ≥ 15 mmHg |
| Pulse rate | bpm | ≤ 50 bpm AND change from Baseline ≤ -15 bpm | ≥ 120 bpm AND change from Baseline ≥ 15 bpm |
| Oxygen saturation | % | < 94 % | Not applicable |
| Body<br>temperature | °C | Not applicable | ≥ 38.3 °C AND change from Baseline ≥ 1.1 °C |

Version Number: Amendment 1, v1.0 Version Date: 23Apr2021

# 17.4. ECG EVALUATIONS

12-lead electrocardiograms (ECGs) will be performed at screening only to assess exclusion criteria 3 of the master protocol. As such ECG data will not be assessed as a safety parameter.

# 17.5. PHYSICAL EXAMINATION

A general physical examination will be performed at screening only. As such, physical examination will not be assessed as a safety parameter.

# 18. DATA NOT SUMMARIZED OR PRESENTED

Data that will not be summarized or listed are:

- Reason for screen failure;
- Inclusion/exclusion criteria;
- SARS-CoV-2 test results;
- Pharmacogenetics sampling;
- Pregnancy test results;
- Screening ECG parameters;
- Screening physical examination;
- Contact information;
- Comments.

These data will be available in the Study Data Tabulation Model (SDTM) datasets.

# 19. REFERENCES

Brookmeyer R, Crowley J. A (1982) Confidence Interval for the Median Survival Time. Biometrics 38:29-41.

Chuang-Stein C (1992). Summarizing laboratory data with different reference ranges in multi-center clinical trials. Drug Information Journal 26(1);77-84.

Lipkovich I, Ratitch B, and O'Kelly M (2016). Sensitivity to censored-at-random assumption in the analysis of time-to-event endpoints. Pharmaceutical Statistics 15;216-229. DOI:10.1002/pst.1738

Moscovici J and Ratitch B (2017). Combining Survival Analysis Results after Multiple Imputation of Censored Event Times. PharmaSUG-Paper SP05.

Royal College of Physicians (2017). National Early Warning Score (NEWS) 2: Standardizing the Assessment of Acute-illness Severity in the NHS – Updated Report of a Working Party. London. <a href="https://www.rcplondon.ac.uk/file/8504/download">https://www.rcplondon.ac.uk/file/8504/download</a> [accessed 08 May 2020].

Rubin DB (1987). Multiple Imputations for Nonresponse in Surveys. New York, NY: John Wiley & Sons, Inc.

# **APPENDIX 1 PARTIAL DATE CONVENTIONS**

# ALGORITHM FOR TREATMENT EMERGENCE OF ADVERSE EVENTS

| START DATE | END DATE | ACTION |
|---|---|---|
| Known | Known/Partial/<br>Missing | If AE start date/time < date/time of first dose of study drug, then not a TEAE; Otherwise, TEAE. |
| Partial, but known components show that AE started before date of first dose of study drug | Known/Partial/<br>Missing | Not TEAE. |
| Partial and known components show that AE started on or after date of first dose of study drug | Known/Partial/<br>Missing | Assume TEAE. |
| | Known | If AE end date/time < date/time of first dose of study drug, then not TEAE; Otherwise, TEAE. |
| Missing | Partial | If known components of AE end date/time show that AE stopped before date/time of first dose of study drug, then not TEAE; Otherwise, TEAE. |
| | Missing | Assume TEAE. |

Note: If an AE started prior to first dose of study drug but worsened after the first dose of study drug, it will be reported as a separate adverse event with new AE start date/time.



# **ALGORITHM FOR PRIOR / CONCOMITANT MEDICATIONS**

| START DATE | STOP DATE | ACTION |
|---|---|---|
| | Known | If medication stop date < date of first dose of study drug, assign as prior; |
| | | Otherwise, assign as concomitant |
| Known, Partial or Missing Partial | | If known components of medication stop date show that medication stopped before date of first dose of study drug, assign as prior; |
| | | Otherwise, assign as concomitant |
| | Missing, or | Can never be assigned as prior, therefore assign as concomitant. |
| | ongoing | |

CCI PPD


# **APPENDIX 2 PROGRAMMING CONVENTIONS FOR OUTPUTS**

# **DATES & TIMES**

Depending on data available, dates and times will take the form yyyy-mm-dd hh:mm.

# **SPELLING FORMAT**

English US.

# PAPER SIZE, ORIENTATION, AND MARGINS

The size of paper will be letter and the page orientation will be landscape. Margins will provide at least 1 inch (2.54 centimeters) of white space all around the page.

## **FONTS**

The font type 'Courier New' will be used, with a font size of 8. The font color will be black with no bolding, underlining, italics or subscripting.

## PRESENTATION OF TREATMENT ARMS

For outputs, treatment arms will be represented as follows and in the given order:

| Treatment arm | Tables and Graphs | Listings |
|------------------------------------|-------------------|----------|
| < <agent>&gt;&gt; plus SoC</agent> | 1 | 1 |
| Placebo plus SoC | 2 | 2 |
| Total [1] | 3 | n/a |
| Screen Failure | n/a | 3 |

[1] Not applicable for efficacy tables, safety tables and graphs.



## PRESENTATION OF NOMINAL VISITS

For outputs, nominal visits will be represented as follows and in that order:

| Long Name (default) | Short Name |
|----------------------------|--------------------------|
| Screening | Scrn |
| Baseline | Base |
| Day x, where $x = 1$ to 29 | Day x, where $x=1$ to 29 |
| Day 60 | Day 60 |

### **DESCRIPTIVE STATISTICS**

If the original data has N decimal places, then the summary statistics will have the following number of decimal places:

- Minimum and maximum: N;
- Mean, Q1, median, Q3, lower and upper bounds of two-sided 95% CI: N + 1;
- SD and SE: N + 2

## **PERCENTAGES**

Percentages will be reported to one decimal place. Rounding will be applied, except for percentages < 0.1 but > 0.0 which will be presented as '< 0.1' and percentages < 100.0 but > 99.9 which will be presented as '> 99.9'.

Where counts are zero, no percentages will appear in the output.

#### **P-VALUES**

p-values will be reported to three decimal places. Rounding will be applied, except for the p-values < 0.001 which will be presented as '< 0.001' and p-values < 1.000 but > 0.999 which will be presented as '> 0.999'.




# **LISTINGS**

All listings will be ordered by the following (unless otherwise indicated in the output template):

- Randomized treatment arm (or treatment received if it's a safety output)
- Patient ID
- Parameter, when applicable
- Date/Time, when applicable
- Timepoint, when applicable

CCI

Master Statistical Analysis Plan

Amgen Inc Master Protocol COV-01 



PPD


CCI

# APPENDIX 4 VASOPRESSOR DRUG CODES AS PER THE WHO DRUG GLOBAL DICTIONARY, SEPTEMBER 2020, VERSION B3

| Drug code | Product Name | <b>Active Ingredients</b> |
|-------------|---------------------------------|---------------------------|
| 00360702173 | 3-hydroxytyramine HCL | Dopamine hydrochloride |
| 00360702174 | 3-hydroxytyramine hydrochloride | Dopamine hydrochloride |
| 00493402134 | 46236 | Dobutamine hydrochloride |
| 00360702138 | A si ke ding | Dopamine hydrochloride |
| 00360702012 | Abbodop | Dopamine hydrochloride |
| 00493402057 | Abbott dobutamine hydrochloride | Dobutamine hydrochloride |
| 00360702103 | Abbott dopamine hcl | Dopamine hydrochloride |
| 00360702024 | Actopamin | Dopamine hydrochloride |
| 00493402099 | Adregotec | Dobutamine hydrochloride |
| 00003902019 | Adreject | Epinephrine hydrochloride |
| 00003902041 | Adren | Epinephrine hydrochloride |
| 00003901075 | Adrenaclick | Epinephrine |
| 00003901055 | Adrenal | Epinephrine |
| 00003901002 | Adrenalin | Epinephrine |
| 00003902015 | Adrenalin | Epinephrine hydrochloride |
| 00003903015 | Adrenalin | Epinephrine bitartrate |
| 00003903051 | Adrenalin aguettant | Epinephrine bitartrate |
| 00003901069 | Adrenalin apotek ab | Epinephrine |
| 00003903057 | Adrenalin bradex | Epinephrine bitartrate |
| 00003901063 | ADRENALIN Carino | Epinephrine |
| 00003901027 | Adrenalin chl sankyo | Epinephrine |
| 00003902052 | Adrenalin chloride | Epinephrine hydrochloride |
| 00003902031 | Adrenalin cl | Epinephrine hydrochloride |
| 00003901103 | Adrenalin galen | Epinephrine |
| 00003902026 | Adrenalin hcl | Epinephrine hydrochloride |
| 00003902063 | Adrenalin hydrochloride | Epinephrine hydrochloride |
| 00003903031 | Adrenalin hydrotar | Epinephrine bitartrate |
| 00003902018 | Adrenalin IMS | Epinephrine hydrochloride |

CCI

PPD




| Drug code | Product Name | Active Ingredients |
|-------------|-----------------------------|---------------------------|
| 00003903040 | Adrenalin Infectopharm | Epinephrine bitartrate |
| 00003901062 | Adrenalin Injeel | Epinephrine |
| 00003903038 | Adrenalin Jenapharm | Epinephrine bitartrate |
| 00003901101 | Adrenalin labatec | Epinephrine |
| 00003903010 | Adrenalin Leiras | Epinephrine bitartrate |
| 00003903048 | Adrenalin Martindale Pharma | Epinephrine bitartrate |
| 00003901026 | Adrenalin medica | Epinephrine |
| 00003903008 | Adrenalin medihal | Epinephrine bitartrate |
| 00003903014 | Adrenalin Merck NM | Epinephrine bitartrate |
| 00003903042 | Adrenalin mylan | Epinephrine bitartrate |
| 00003901106 | Adrenalin osel | Epinephrine |
| 00003901107 | Adrenalin solofarm | Epinephrine |
| 00003903052 | Adrenalin stragen | Epinephrine bitartrate |
| 00003901022 | Adrenalin streuli | Epinephrine |
| 00003903033 | Adrenalin Tartrate | Epinephrine bitartrate |
| 00003903024 | Adrenalina | Epinephrine bitartrate |
| 00003902037 | Adrenalina | Epinephrine hydrochloride |
| 00003901019 | Adrenalina | Epinephrine |
| 00003903054 | Adrenalina Aguettant | Epinephrine bitartrate |
| 00003902042 | Adrenalina apolo | Epinephrine hydrochloride |
| 00003901047 | Adrenalina biol | Epinephrine |
| 00003902057 | Adrenalina braun | Epinephrine hydrochloride |
| 00003902048 | Adrenalina clorhidrato | Epinephrine hydrochloride |
| 00003901048 | Adrenalina fada | Epinephrine |
| 00003901066 | Adrenalina galenica senese | Epinephrine |
| 00003902013 | Adrenalina level | Epinephrine hydrochloride |
| 00003902007 | Adrenalina llorente | Epinephrine hydrochloride |
| 00003902014 | Adrenalina miro | Epinephrine hydrochloride |
| 00003902065 | Adrenalina ogna | Epinephrine hydrochloride |
| 00003902028 | Adrenalina pisa | Epinephrine hydrochloride |
| 00003901021 | Adrenalina sintetica | Epinephrine |
| 00003903045 | Adrenalina wzf | Epinephrine bitartrate |
| 00003903005 | Adrenaline | Epinephrine bitartrate |

<u>CCI</u>

PPD




| Drug code | Product Name | Active Ingredients |
|---|---|---|
| 00003902047 | Adrenaline | Epinephrine hydrochloride |
| 00003901003 | Adrenaline | Epinephrine |
| 00003903055 | Adrenaline (Epinephrine) Injection BP 1:1000 | Epinephrine bitartrate |
| 00003902060 | Adrenaline (HCl) Sterop | Epinephrine hydrochloride |
| 00003901089 | Adrenaline (tartrate) Aguettant | Epinephrine |
| 00003903037 | Adrenaline (Tartrate) Sterop | Epinephrine bitartrate |
| 00003903026 | Adrenaline acid tartrate | Epinephrine bitartrate |
| 00003901040 | Adrenaline aguettant | Epinephrine |
| 00003901094 | Adrenaline aurum | Epinephrine |
| 00003901041 | Adrenaline b.braun | Epinephrine |
| 00003901042 | Adrenaline cooper | Epinephrine |
| 00003903036 | Adrenaline Demo | Epinephrine bitartrate |
| 00003903056 | Adrenaline fresenius | Epinephrine bitartrate |
| 00003902025 | Adrenaline hcl | Epinephrine hydrochloride |
| 00003902053 | Adrenaline hydrochloride | Epinephrine hydrochloride |
| 00003901098 | Adrenaline jr mylan | Epinephrine |
| 00003901072 | Adrenaline Lavois | Epinephrine |
| 00003902072 | Adrenaline life | Epinephrine hydrochloride |
| 00003903046 | Adrenaline link | Epinephrine bitartrate |
| 00003901091 | Adrenaline martindale | Epinephrine |
| 00003901099 | Adrenaline mylan | Epinephrine |
| 00003902062 | Adrenaline Parke-Davis | Epinephrine hydrochloride |
| 00003901058 | Adrenaline pch | Epinephrine |
| 00003903049 | Adrenaline renaudin | Epinephrine bitartrate |
| 00003901100 | Adrenaline solopharm | Epinephrine |
| 00003901093 | Adrenaline sophar | Epinephrine |
| 00003903043 | Adrenaline tartrate | Epinephrine bitartrate |
| 00003901102 | Adrenaline/ariti | Epinephrine |
| 00003902059 | Adrenalini | Epinephrine hydrochloride |
| 00003903029 | Adrenalini bitartras | Epinephrine bitartrate |
| 00003902068 | Adrenalini hcl | Epinephrine hydrochloride |
| 00003902069 | Adrenalini hydrochloridum | Epinephrine hydrochloride |
| 00003902056 | Adrenalini hydrotartras | Epinephrine hydrochloride |

CCI

PPD





| Drug code | Product Name | Active Ingredients |
|-------------|-------------------------|------------------------------|
| 00003903030 | Adrenalini hydrotartras | Epinephrine bitartrate |
| 00003903032 | Adrenalini tartras | Epinephrine bitartrate |
| 00003904003 | Adrenalin-neutrale | Epinephryl borate |
| 00003903016 | Adrenalinum | Epinephrine bitartrate |
| 00003901081 | Adrenalinum | Epinephrine |
| 00003901087 | Adrenol | Epinephrine |
| 00127502065 | Adrenor | Norepinephrine bitartrate |
| 00003903027 | Adrenotone | Epinephrine bitartrate |
| 00003901051 | Adrine | Epinephrine |
| 00003901076 | Adrinor | Epinephrine |
| 00127501007 | ADS-Noltron | Norepinephrine |
| 00003901097 | Adyphren amp kit | Epinephrine |
| 00003901085 | Allerject | Epinephrine |
| 00003901061 | Altellus | Epinephrine |
| 00493402104 | An chang | Dobutamine hydrochloride |
| 00003902051 | Anaguard | Epinephrine hydrochloride |
| 00003902012 | Ana-guard | Epinephrine hydrochloride |
| 00003901045 | Anahelp | Epinephrine |
| 00003901044 | Anakit | Epinephrine |
| 00003901031 | Anapen | Epinephrine |
| 00003902045 | Anapen | Epinephrine hydrochloride |
| 01872201012 | Antidiuretic hormone | Vasopressin |
| 00493402085 | Ao wan yuan | Dobutamine hydrochloride |
| 00493402067 | Ao wang yan | Dobutamine hydrochloride |
| 00360702128 | Aprical dopamida | Dopamine hydrochloride |
| 01872201024 | Argipresina | Vasopressin |
| 01872201016 | Argipressin | Vasopressin |
| 00127503002 | Arterenol | Norepinephrine hydrochloride |
| 01872201018 | Arterina | Vasopressin |
| 00360702175 | Asl-279 | Dopamine hydrochloride |
| 00003903035 | Aspen Adrenaline | Epinephrine bitartrate |
| 00003903004 | Asthmahaler | Epinephrine bitartrate |
| 00003901028 | Asthsedan | Epinephrine |

CCI

PPD





| Drug code | Product Name | Active Ingredients |
|-------------|--------------------------|---------------------------|
| 00003901073 | Auvi q | Epinephrine |
| 00360702159 | Bagotropin | Dopamine hydrochloride |
| 00127502064 | Biemefrin | Norepinephrine bitartrate |
| 00003902005 | Bosmin | Epinephrine hydrochloride |
| 00003901029 | Bosmin | Epinephrine |
| 00003901009 | Bronkaid | Epinephrine |
| 00003902032 | Bronkaid | Epinephrine hydrochloride |
| 00493402010 | Bubucin | Dobutamine hydrochloride |
| 00493402112 | Butamine | Dobutamine hydrochloride |
| 00493402143 | Cardease | Dobutamine hydrochloride |
| 00127502063 | Cardenor | Norepinephrine bitartrate |
| 00127502040 | Cardiamed | Norepinephrine bitartrate |
| 00493402118 | Cardiforce | Dobutamine hydrochloride |
| 00493402050 | Cardiject | Dobutamine hydrochloride |
| 00493402056 | Cardiomin | Dobutamine hydrochloride |
| 00360702105 | Cardiopal | Dopamine hydrochloride |
| 00493402149 | Cardiotrex | Dobutamine hydrochloride |
| 00493402160 | Cardob | Dobutamine hydrochloride |
| 00493402120 | Cardomin | Dobutamine hydrochloride |
| 00360702144 | Cardopa | Dopamine hydrochloride |
| 00360702016 | Catabon | Dopamine hydrochloride |
| 00360702152 | Catherine | Dopamine hydrochloride |
| 00360702038 | Catherine amel | Dopamine hydrochloride |
| 00003903058 | CCM Adrenaline Injection | Epinephrine bitartrate |
| 00360702109 | Cetadop | Dopamine hydrochloride |
| 00003901088 | Chenpen | Epinephrine |
| 00360702187 | Clorhidrat de dopamina | Dopamine hydrochloride |
| 00360702131 | Clorhidrato dopamina | Dopamine hydrochloride |
| 00493402037 | Cloridrato de dobutamina | Dobutamine hydrochloride |
| 00360702081 | Cloridrato de dopamina | Dopamine hydrochloride |
| 00360702066 | Clorpamina | Dopamine hydrochloride |
| 00360702151 | Constriction | Dopamine hydrochloride |
| 00493402152 | Corbusin | Dobutamine hydrochloride |

CCI

PPD




| Drug code | Product Name | Active Ingredients |
|-------------|--------------------|--------------------------|
| 00360702167 | Cordodopa | Dopamine hydrochloride |
| 00360702170 | Cordodopa Forte | Dopamine hydrochloride |
| 00360702052 | Corskool | Dopamine hydrochloride |
| 01872201020 | Cpressin p | Vasopressin |
| 00360702013 | Critpan | Dopamine hydrochloride |
| 00493402025 | Cryobutol | Dobutamine hydrochloride |
| 00493402126 | Dasomin | Dobutamine hydrochloride |
| 00360702045 | Dasomin | Dopamine hydrochloride |
| 00003901049 | Davinefrina | Epinephrine |
| 00003901064 | Denolin Adrenaline | Epinephrine |
| 00493401002 | Dobaden | Dobutamine |
| 00493402093 | Dobamin | Dobutamine hydrochloride |
| 00493402044 | Dobamine | Dobutamine hydrochloride |
| 00493402088 | Dobcard | Dobutamine hydrochloride |
| 00493402052 | Dobicard | Dobutamine hydrochloride |
| 00493402147 | Dobier s | Dobutamine hydrochloride |
| 00493402109 | Dobine | Dobutamine hydrochloride |
| 00493402036 | Dobtan | Dobutamine hydrochloride |
| 00493402140 | Dobuca | Dobutamine hydrochloride |
| 00493402133 | Dobucard | Dobutamine hydrochloride |
| 00493402053 | Dobucef | Dobutamine hydrochloride |
| 00493402054 | Dobucin | Dobutamine hydrochloride |
| 00493402034 | Dobucor | Dobutamine hydrochloride |
| 00493402077 | Dobuha | Dobutamine hydrochloride |
| 00493402005 | Dobuject | Dobutamine hydrochloride |
| 00493402125 | Dobulex | Dobutamine hydrochloride |
| 00493402157 | Dobulon | Dobutamine hydrochloride |
| 00493402161 | Dobumarc | Dobutamine hydrochloride |
| 00493402151 | Dobumean | Dobutamine hydrochloride |
| 00493402045 | Dobumin | Dobutamine hydrochloride |
| 00493402137 | Dobumine | Dobutamine hydrochloride |
| 00493402116 | Dobunex pf | Dobutamine hydrochloride |
| 00493402021 | Dobupum | Dobutamine hydrochloride |

<u>CCI</u>

PPD




Master Statistical Analysis Plan

| Drug code | Product Name | Active Ingredients |
|-------------|-------------------------|--------------------------|
| 00493402017 | Doburack | Dobutamine hydrochloride |
| 00493402079 | Doburak | Dobutamine hydrochloride |
| 00493402043 | Doburan | Dobutamine hydrochloride |
| 00493402087 | Dobusol | Dobutamine hydrochloride |
| 00493402094 | Dobustat | Dobutamine hydrochloride |
| 00493402078 | Dobutal | Dobutamine hydrochloride |
| 00493402048 | Dobutam | Dobutamine hydrochloride |
| 00493402004 | Dobutamin | Dobutamine hydrochloride |
| 00493402012 | Dobutamin abbott | Dobutamine hydrochloride |
| 00493402089 | Dobutamin Admeda | Dobutamine hydrochloride |
| 00493402159 | Dobutamin carinopharm | Dobutamine hydrochloride |
| 00493402102 | Dobutamin ebewe | Dobutamine hydrochloride |
| 00493402013 | Dobutamin Fresenius | Dobutamine hydrochloride |
| 00493402059 | Dobutamin giulini | Dobutamine hydrochloride |
| 00493402130 | Dobutamin hameln | Dobutamine hydrochloride |
| 00493402022 | Dobutamin hexal | Dobutamine hydrochloride |
| 00493402106 | Dobutamin ratiopharm | Dobutamine hydrochloride |
| 00493401004 | Dobutamina | Dobutamine |
| 00493402040 | Dobutamina | Dobutamine hydrochloride |
| 00493402032 | Dobutamina abbott | Dobutamine hydrochloride |
| 00493402086 | Dobutamina Aps | Dobutamine hydrochloride |
| 00493402098 | Dobutamina bioindustria | Dobutamine hydrochloride |
| 00493402146 | Dobutamina Claris | Dobutamine hydrochloride |
| 00493402041 | Dobutamina fabra | Dobutamine hydrochloride |
| 00493402115 | Dobutamina fu | Dobutamine hydrochloride |
| 00493402138 | Dobutamina Generis | Dobutamine hydrochloride |
| 00493402141 | Dobutamina genthon | Dobutamine hydrochloride |
| 00493402024 | Dobutamina gi pisa | Dobutamine hydrochloride |
| 00493402026 | Dobutamina gi tecn | Dobutamine hydrochloride |
| 00493402139 | Dobutamina gray | Dobutamine hydrochloride |
| 00493402035 | Dobutamina inibsa | Dobutamine hydrochloride |
| 00493402023 | Dobutamina kendric | Dobutamine hydrochloride |
| 00493402132 | Dobutamina Norgreen | Dobutamine hydrochloride |

CCI

PPD




Master Statistical Analysis Plan

| Drug code | Product Name | Active Ingredients |
|-------------|-------------------------------|--------------------------|
| 00493402156 | Dobutamina panpharma | Dobutamine hydrochloride |
| 00493402033 | Dobutamina rovi | Dobutamine hydrochloride |
| 00493402103 | Dobutamina sanderson | Dobutamine hydrochloride |
| 00493401001 | Dobutamine | Dobutamine |
| 00493402007 | Dobutamine | Dobutamine hydrochloride |
| 00493402062 | Dobutamine abbott | Dobutamine hydrochloride |
| 00493402075 | Dobutamine Aguettant | Dobutamine hydrochloride |
| 00493402063 | Dobutamine antigen | Dobutamine hydrochloride |
| 00493402047 | Dobutamine baxter | Dobutamine hydrochloride |
| 00493402068 | Dobutamine CF | Dobutamine hydrochloride |
| 00493402122 | Dobutamine Claris | Dobutamine hydrochloride |
| 00493402030 | Dobutamine dakota | Dobutamine hydrochloride |
| 00493402097 | Dobutamine EG | Dobutamine hydrochloride |
| 00493402155 | Dobutamine fresenius | Dobutamine hydrochloride |
| 00493402111 | Dobutamine hameln | Dobutamine hydrochloride |
| 00493402028 | Dobutamine hel | Dobutamine hydrochloride |
| 00493402073 | Dobutamine hel DBL | Dobutamine hydrochloride |
| 00493402072 | Dobutamine hexal | Dobutamine hydrochloride |
| 00493402001 | Dobutamine Hydrochloride | Dobutamine hydrochloride |
| 00493403001 | Dobutamine lactobionate | Dobutamine lactobionate |
| 00493402046 | Dobutamine mayne pharma (ben) | Dobutamine hydrochloride |
| 00493402029 | Dobutamine merck | Dobutamine hydrochloride |
| 00493402108 | Dobutamine mylan | Dobutamine hydrochloride |
| 00493402076 | Dobutamine Panpharma | Dobutamine hydrochloride |
| 00493402113 | Dobutamine Qualimed | Dobutamine hydrochloride |
| 00493402136 | Dobutamine sdz | Dobutamine hydrochloride |
| 00493402092 | Dobutamine winthrop | Dobutamine hydrochloride |
| 00493402049 | Dobutamine-abbott | Dobutamine hydrochloride |
| 00493402066 | Dobutamine-bc | Dobutamine hydrochloride |
| 00493402091 | Dobutamin-hameln | Dobutamine hydrochloride |
| 00493402135 | Dobutamini hydrochloridum | Dobutamine hydrochloride |
| 00493401003 | Dobutaminum | Dobutamine |
| 00493402039 | Dobutamol | Dobutamine hydrochloride |

CCI

PPD





| Drug code | Product Name | Active Ingredients |
|-------------|-----------------|--------------------------|
| 00493402090 | Dobutan | Dobutamine hydrochloride |
| 00493402107 | Dobutanil | Dobutamine hydrochloride |
| 00493402144 | Dobutasel | Dobutamine hydrochloride |
| 00493402061 | Dobutel | Dobutamine hydrochloride |
| 00493402150 | Dobuthaver | Dobutamine hydrochloride |
| 00493402038 | Dobutil | Dobutamine hydrochloride |
| 00493402121 | Dobutin | Dobutamine hydrochloride |
| 00493402127 | Dobutina | Dobutamine hydrochloride |
| 00493402002 | Dobutrex | Dobutamine hydrochloride |
| 00493402080 | Dobutrex k | Dobutamine hydrochloride |
| 00493402096 | Dobutrim | Dobutamine hydrochloride |
| 00493402158 | Dobutrust | Dobutamine hydrochloride |
| 00493402071 | Dobux | Dobutamine hydrochloride |
| 00493402019 | Dobux nichiiko | Dobutamine hydrochloride |
| 00493402058 | Dobuxin | Dobutamine hydrochloride |
| 00493402124 | Dobuzef | Dobutamine hydrochloride |
| 00360702101 | Docard | Dopamine hydrochloride |
| 00360702064 | Dofamin | Dopamine hydrochloride |
| 00360702186 | Dofamine | Dopamine hydrochloride |
| 00360702172 | Dofamine Ferein | Dopamine hydrochloride |
| 00493402119 | Dofuse | Dobutamine hydrochloride |
| 00360702040 | Dolpamil | Dopamine hydrochloride |
| 00360702116 | Domin | Dopamine hydrochloride |
| 00360702093 | Domine | Dopamine hydrochloride |
| 00493402128 | Dominic | Dobutamine hydrochloride |
| 00360702014 | Dominin | Dopamine hydrochloride |
| 00360702162 | Domins | Dopamine hydrochloride |
| 00360702050 | Donapan | Dopamine hydrochloride |
| 00360702044 | Doncal | Dopamine hydrochloride |
| 00360702058 | Dopa kit | Dopamine hydrochloride |
| 00360702082 | Dopabane | Dopamine hydrochloride |
| 00360702185 | Dopabas | Dopamine hydrochloride |
| 00360702113 | Dopac | Dopamine hydrochloride |

<u>CCI</u>

PPD




| Drug code | Product Name | Active Ingredients |
|-------------|----------------------|------------------------|
| 00360702161 | Dopacef | Dopamine hydrochloride |
| 00360702147 | Dopacin | Dopamine hydrochloride |
| 00360702083 | Dopacris | Dopamine hydrochloride |
| 00360702140 | Dopadren | Dopamine hydrochloride |
| 00360702178 | Dopaglan | Dopamine hydrochloride |
| 00360702143 | Dopamax | Dopamine hydrochloride |
| 00360702117 | Dopamex | Dopamine hydrochloride |
| 00360702003 | Dopamin | Dopamine hydrochloride |
| 00360702136 | Dopamin Admeda | Dopamine hydrochloride |
| 00360702030 | Dopamin braun | Dopamine hydrochloride |
| 00360702065 | Dopamin ebewe | Dopamine hydrochloride |
| 00360702029 | Dopamin fresenius | Dopamine hydrochloride |
| 00360702025 | Dopamin giulini | Dopamine hydrochloride |
| 00360702114 | Dopamin hausmann | Dopamine hydrochloride |
| 00360702070 | Dopamin natter | Dopamine hydrochloride |
| 00360702150 | Dopamin Sintetica | Dopamine hydrochloride |
| 00360702126 | Dopamin solvay | Dopamine hydrochloride |
| 00360701004 | Dopamina | Dopamine |
| 00360702080 | Dopamina | Dopamine hydrochloride |
| 00360702165 | Dopamina 3m | Dopamine hydrochloride |
| 00360702076 | Dopamina abbott | Dopamine hydrochloride |
| 00360702182 | Dopamina basi | Dopamine hydrochloride |
| 00360702168 | Dopamina clorhidrato | Dopamine hydrochloride |
| 00360702194 | Dopamina cloridrato | Dopamine hydrochloride |
| 00360702087 | Dopamina duncan | Dopamine hydrochloride |
| 00360702164 | Dopamina exakta | Dopamine hydrochloride |
| 00360702130 | Dopamina fides | Dopamine hydrochloride |
| 00360702160 | Dopamina fu | Dopamine hydrochloride |
| 00360702069 | Dopamina gi zafiro | Dopamine hydrochloride |
| 00360702181 | Dopamina grifols | Dopamine hydrochloride |
| 00360702068 | Dopamina kendrick | Dopamine hydrochloride |
| 00360702163 | Dopamina northia | Dopamine hydrochloride |
| 00360702078 | Dopamina pht | Dopamine hydrochloride |

<u>CCI</u>

PPD




Master Statistical Analysis Plan

| Drug code | Product Name | Active Ingredients |
|-------------|----------------------------------|------------------------|
| 00360702077 | Dopamina salf | Dopamine hydrochloride |
| 00360702183 | Dopamina surar pharma | Dopamine hydrochloride |
| 00360701001 | Dopamine | Dopamine |
| 00360702007 | Dopamine | Dopamine hydrochloride |
| 00360702119 | Dopamine abbott | Dopamine hydrochloride |
| 00360702074 | Dopamine aguettant | Dopamine hydrochloride |
| 00360702095 | Dopamine fresenius | Dopamine hydrochloride |
| 00360702071 | Dopamine hel | Dopamine hydrochloride |
| 00360702111 | Dopamine hel abbott | Dopamine hydrochloride |
| 00360702102 | Dopamine hel-fresenius | Dopamine hydrochloride |
| 00360702096 | Dopamine hycrochloride | Dopamine hydrochloride |
| 00360702001 | Dopamine hydrochloride | Dopamine hydrochloride |
| 00360702115 | Dopamine hydrochloride dbl | Dopamine hydrochloride |
| 00360702124 | Dopamine hydrochloride kobayashi | Dopamine hydrochloride |
| 00360702134 | Dopamine Hydrochloride Mochida | Dopamine hydrochloride |
| 00360702133 | Dopamine Hydrochloride Shionogi | Dopamine hydrochloride |
| 00360702073 | Dopamine lucien | Dopamine hydrochloride |
| 00360702075 | Dopamine merck | Dopamine hydrochloride |
| 00360702193 | Dopamine mylan | Dopamine hydrochloride |
| 00360702127 | Dopamine nativelle | Dopamine hydrochloride |
| 00360702146 | Dopamine PCH | Dopamine hydrochloride |
| 00360702072 | Dopamine pierre fabre | Dopamine hydrochloride |
| 00360702062 | Dopamine premix | Dopamine hydrochloride |
| 00360702135 | Dopamine Renaudin | Dopamine hydrochloride |
| 00360702057 | Dopamine towa | Dopamine hydrochloride |
| 00360702190 | Dopamine/anfarm | Dopamine hydrochloride |
| 00360702099 | Dopamine-p | Dopamine hydrochloride |
| 00360702100 | Dopaminex | Dopamine hydrochloride |
| 00360702176 | Dopamini hydrochloridum | Dopamine hydrochloride |
| 00360701003 | Dopaminum | Dopamine |
| 00360702129 | Dopaminum hydrochloricum | Dopamine hydrochloride |
| 00360702085 | Dopamol | Dopamine hydrochloride |
| 00360702094 | Dopan | Dopamine hydrochloride |

CCI

PPD




| Drug code | Product Name | <b>Active Ingredients</b> |
|-------------|-------------------|---------------------------|
| 00360702098 | Dopaplus | Dopamine hydrochloride |
| 00360702166 | Dopaqard | Dopamine hydrochloride |
| 00360702041 | Doparalmin | Dopamine hydrochloride |
| 00360702192 | Dopasel | Dopamine hydrochloride |
| 00360702092 | Dopasin | Dopamine hydrochloride |
| 00360702191 | Dopasunny | Dopamine hydrochloride |
| 00360702180 | Dopatropin | Dopamine hydrochloride |
| 00360702123 | Dopavate | Dopamine hydrochloride |
| 00360702195 | Dopazef | Dopamine hydrochloride |
| 00360702110 | Doperba | Dopamine hydrochloride |
| 00360702063 | Dophamin | Dopamine hydrochloride |
| 00360702120 | Dopin | Dopamine hydrochloride |
| 00360702106 | Dopina | Dopamine hydrochloride |
| 00360702097 | Dopinga | Dopamine hydrochloride |
| 00360702033 | Dopmin | Dopamine hydrochloride |
| 00360701002 | Dopmin | Dopamine |
| 00493402016 | Dopmin | Dobutamine hydrochloride |
| 00493402081 | Dopmin-k | Dobutamine hydrochloride |
| 00360702179 | Dopnax | Dopamine hydrochloride |
| 00360702088 | Dopramine | Dopamine hydrochloride |
| 00360702139 | Dopress | Dopamine hydrochloride |
| 00360702196 | Doprina | Dopamine hydrochloride |
| 00493402082 | Doputamin | Dobutamine hydrochloride |
| 00493402100 | Doputamin Fuji | Dobutamine hydrochloride |
| 00493402020 | Doputamin h hexal | Dobutamine hydrochloride |
| 00493402083 | Doputamin k | Dobutamine hydrochloride |
| 00493402101 | Dotamin | Dobutamine hydrochloride |
| 00493402055 | Dotrex | Dobutamine hydrochloride |
| 00493402145 | Dotropina | Dobutamine hydrochloride |
| 00003901079 | Drenalin | Epinephrine |
| 00127502068 | Drenorep | Norepinephrine bitartrate |
| 00493402148 | Dubuject | Dobutamine hydrochloride |
| 00493402114 | Duvig | Dobutamine hydrochloride |

CCI

PPD





| Drug code | Product Name | Active Ingredients |
|-------------|---------------------------|---------------------------|
| 00360702079 | Dynatra | Dopamine hydrochloride |
| 00360702021 | Dynatra dopamine | Dopamine hydrochloride |
| 00360702020 | Dynos | Dopamine hydrochloride |
| 00003902039 | Dyspne inhalante | Epinephrine hydrochloride |
| 00003901039 | Dyspne-inhal | Epinephrine |
| 00493402142 | E.m.c. dobutamina | Dobutamine hydrochloride |
| 00493402123 | Easydobu | Dobutamine hydrochloride |
| 00360702149 | Easydopa | Dopamine hydrochloride |
| 00003901065 | Efrinalin | Epinephrine |
| 00360702047 | Elebumin | Dopamine hydrochloride |
| 00003903047 | Emerade | Epinephrine bitartrate |
| 00003903044 | Enatrate | Epinephrine bitartrate |
| 01872201008 | Encrise | Vasopressin |
| 00003901096 | Ephedrix | Epinephrine |
| 00003902033 | Epi e-z | Epinephrine hydrochloride |
| 00003902034 | Epi e-z pen jr. | Epinephrine hydrochloride |
| 00003902071 | Epibbas | Epinephrine hydrochloride |
| 00003903034 | Epifrin | Epinephrine bitartrate |
| 00003902022 | Epifrin | Epinephrine hydrochloride |
| 00003904004 | Epinal | Epinephryl borate |
| 00003902049 | Epinefrina | Epinephrine hydrochloride |
| 00003901050 | Epinefrina | Epinephrine |
| 00003901001 | Epinephrine | Epinephrine |
| 00003902030 | Epinephrine | Epinephrine hydrochloride |
| 00003903006 | Epinephrine | Epinephrine bitartrate |
| 00003903001 | Epinephrine bitartrate | Epinephrine bitartrate |
| 00003902070 | Epinephrine HCL | Epinephrine hydrochloride |
| 00003902001 | Epinephrine hydrochloride | Epinephrine hydrochloride |
| 00003901070 | Epinephrine minijet | Epinephrine |
| 00003901108 | Epinephrine professional | Epinephrine |
| 00003901105 | Epinephrinesnap v | Epinephrine |
| 00003901077 | Epinephrinum | Epinephrine |
| 00003904001 | Epinephryl borate | Epinephryl borate |

CCI

PPD




Master Statistical Analysis Plan


| Drug code | Product Name | Active Ingredients |
|-------------|-------------------|---------------------------------------|
| 00127504004 | Epinor | Norepinephrine bitartrate monohydrate |
| 00003901014 | Epipen | Epinephrine |
| 00003901082 | Epipen 2-pak | Epinephrine |
| 00003901084 | Epipen jr | Epinephrine |
| 00003901037 | Epipen jr 2-pak | Epinephrine |
| 00003901104 | Epipen junior | Epinephrine |
| 00003901020 | Epiquick | Epinephrine |
| 00003902043 | Epiren | Epinephrine hydrochloride |
| 00003902054 | Epirenamin | Epinephrine hydrochloride |
| 00003902064 | Epirenin | Epinephrine hydrochloride |
| 00003901086 | Episnap | Epinephrine |
| 00003901071 | Epista | Epinephrine |
| 00003903003 | Epitrate | Epinephrine bitartrate |
| 00003902073 | Epix | Epinephrine hydrochloride |
| 00003901024 | Ерру | Epinephrine |
| 00003904002 | Ерру п | Epinephryl borate |
| 00003901013 | Eppy plus | Epinephrine |
| 00360702022 | Evetant | Dopamine hydrochloride |
| 00360702059 | Evetant hexal | Dopamine hydrochloride |
| 00360702056 | Evetant towa | Dopamine hydrochloride |
| 00003902011 | Fastjekt | Epinephrine hydrochloride |
| 00003902038 | Fastjekt junior | Epinephrine hydrochloride |
| 00127502036 | Fioritina | Norepinephrine bitartrate |
| 00127502073 | Forefrin | Norepinephrine bitartrate |
| 00360702042 | Gabans | Dopamine hydrochloride |
| 00493402065 | Gendobu | Dobutamine hydrochloride |
| 00360702004 | Giludop | Dopamine hydrochloride |
| 00003902066 | Gingi pak z twist | Epinephrine hydrochloride |
| 00003901012 | Gingipak | Epinephrine |
| 00360702156 | Gipamine | Dopamine hydrochloride |
| 00003902027 | Glaucon | Epinephrine hydrochloride |
| 00003903011 | Glaucon | Epinephrine bitartrate |
| 00003902010 | Glaufrin | Epinephrine hydrochloride |

CCI

PPD






| Drug code | Product Name | Active Ingredients |
|-------------|--------------------------------|---------------------------|
| 00003901015 | Glauposine | Epinephrine |
| 00127502028 | Hemitartarato de Norepinefrina | Norepinephrine bitartrate |
| 00493402015 | Hercarenone d | Dobutamine hydrochloride |
| 00360702086 | Hettytropin | Dopamine hydrochloride |
| 00003901046 | Hydren | Epinephrine |
| 00127502014 | Hyponor | Norepinephrine bitartrate |
| 00493402153 | Imatim | Dobutamine hydrochloride |
| 00003902023 | Ims adrenaline | Epinephrine hydrochloride |
| 00360702061 | Ims dopamine | Dopamine hydrochloride |
| 00360702112 | Indop | Dopamine hydrochloride |
| 00003902055 | Infectokrupp | Epinephrine hydrochloride |
| 00003903053 | Infectokrupp | Epinephrine bitartrate |
| 00127502034 | Infunor | Norepinephrine bitartrate |
| 00493402095 | Inocard | Dobutamine hydrochloride |
| 00493402131 | Inodex | Dobutamine hydrochloride |
| 00493402117 | Inoject | Dobutamine hydrochloride |
| 00360702090 | Inophan | Dopamine hydrochloride |
| 00360702118 | Inopin | Dopamine hydrochloride |
| 00493402027 | Inotop | Dobutamine hydrochloride |
| 00493402003 | Inotrex | Dobutamine hydrochloride |
| 00493402060 | Inotrop | Dobutamine hydrochloride |
| 00360702067 | Inotropin | Dopamine hydrochloride |
| 00360702084 | Inotropisa | Dopamine hydrochloride |
| 00360702005 | Inovan | Dopamine hydrochloride |
| 00360702002 | Intropin | Dopamine hydrochloride |
| 00360702060 | Intropin ahs | Dopamine hydrochloride |
| 00003901032 | Isopto ephinal | Epinephrine |
| 00003901025 | Isopto epinal | Epinephrine |
| 00003901007 | Isoptoepinal | Epinephrine |
| 00003903039 | Jext | Epinephrine bitartrate |
| 00360702031 | Kakodin | Dopamine hydrochloride |
| 00360702137 | Kakodin D | Dopamine hydrochloride |
| 00493402051 | Kardia | Dobutamine hydrochloride |

<u>CCI</u>

PPD




Master Statistical Analysis Plan

| Drug code | Product Name | Active Ingredients |
|-------------|----------------------------|------------------------------|
| 00127502049 | L noradrenalina braun | Norepinephrine bitartrate |
| 00003901035 | L-adrenalin | Epinephrine |
| 00003901078 | L-epinephrine | Epinephrine |
| 00127501003 | Levarterenol | Norepinephrine |
| 00127502038 | Levarterenol bitartrate | Norepinephrine bitartrate |
| 00127503007 | Levarterenol HCL | Norepinephrine hydrochloride |
| 00127503008 | Levarterenol hydrochloride | Norepinephrine hydrochloride |
| 00003902008 | Levocon | Epinephrine hydrochloride |
| 00127502005 | Levonor | Norepinephrine bitartrate |
| 00127502002 | Levophed | Norepinephrine bitartrate |
| 00127502023 | Levophed bitartrat | Norepinephrine bitartrate |
| 00127502003 | Levophed bitartrate | Norepinephrine bitartrate |
| 00127501009 | Levophrine | Norepinephrine |
| 00003903019 | Liadren | Epinephrine bitartrate |
| 00360702177 | Loxin | Dopamine hydrochloride |
| 00003903009 | Lyophrin | Epinephrine bitartrate |
| 00360702043 | Martburn | Dopamine hydrochloride |
| 00003902024 | Mediastman | Epinephrine hydrochloride |
| 00003903020 | Medihaler | Epinephrine bitartrate |
| 00003903002 | Medihaler-epi | Epinephrine bitartrate |
| 00360702169 | Medopa | Dopamine hydrochloride |
| 00360702158 | Megadose | Dopamine hydrochloride |
| 00493402162 | Mekard | Dobutamine hydrochloride |
| 00127502081 | Mephrin | Norepinephrine bitartrate |
| 00003901030 | Mf adrenalin | Epinephrine |
| 00360702148 | Micro Dopamine | Dopamine hydrochloride |
| 00003903028 | Micro-adrenaline | Epinephrine bitartrate |
| 00003902004 | Micronefrin | Epinephrine hydrochloride |
| 00003901059 | Min-I-Jet Adrenalin | Epinephrine |
| 00360702141 | Miocina | Dopamine hydrochloride |
| 00493402031 | Miozac | Dobutamine hydrochloride |
| 00360702051 | Mitasmin | Dopamine hydrochloride |
| 00493402129 | Mobitil | Dobutamine hydrochloride |

<u>CCI</u>

PPD




| Drug code | Product Name | Active Ingredients |
|---|---|---|
| 00360702104 | Myocard | Dopamine hydrochloride |
| 00360702184 | Myofast | Dopamine hydrochloride |
| 00360702171 | Myomine | Dopamine hydrochloride |
| 00360702189 | Myotil | Dopamine hydrochloride |
| 00127502058 | N Epi | Norepinephrine bitartrate |
| 00003901004 | Nebulogenum hectalini | Epinephrine |
| 00127502086 | Nefrinor | Norepinephrine bitartrate |
| 00003902058 | Neosynephrine Badrial | Epinephrine hydrochloride |
| 00127502090 | Nevoleen | Norepinephrine bitartrate |
| 00127502083 | Nobify | Norepinephrine bitartrate |
| 00127502008 | Nor adrenalin | Norepinephrine bitartrate |
| 00127501010 | Nor adrenalin | Norepinephrine |
| 00127502020 | Norad | Norepinephrine bitartrate |
| 00127502087 | Norad 4 | Norepinephrine bitartrate |
| 00127502041 | Noradrec | Norepinephrine bitartrate |
| 00127502013 | Noradren | Norepinephrine bitartrate |
| 00127501005 | Noradrenalin | Norepinephrine |
| 00127502006 | Noradrenalin | Norepinephrine bitartrate |
| 00127503005 | Noradrenalin | Norepinephrine hydrochloride |
| 00127503006 | Nor-Adrenalin | Norepinephrine hydrochloride |
| 00127502017 | Nor-adrenalin | Norepinephrine bitartrate |
| 00127502051 | Noradrenalin Abcur | Norepinephrine bitartrate |
| 00127502084 | Noradrenalin aguettant | Norepinephrine bitartrate |
| 00127502010 | Noradrenalin Bichsel | Norepinephrine bitartrate |
| 00127502045 | Noradrenalin Hospira | Norepinephrine bitartrate |
| 00127502094 | Noradrenalin ligula pharma | Norepinephrine bitartrate |
| 00127502011 | Noradrenalin mayrhofer | Norepinephrine bitartrate |
| 00127502042 | Noradrenalin naf sykehusapoteket | Norepinephrine bitartrate |
| 00127502061 | Noradrenalin orpha | Norepinephrine bitartrate |
| 00127502007 | Noradrenalin sad | Norepinephrine bitartrate |
| 00127502098 | Noradrenalin sintetica | Norepinephrine bitartrate |
| 00127503004 | Noradrenalina | Norepinephrine hydrochloride |
| 00127502043 | Noradrenalina | Norepinephrine bitartrate |

CCI

PPD




| Drug code | Product Name | Active Ingredients |
|---|---|---|
| 00127501006 | Noradrenalina | Norepinephrine |
| 00127502071 | Noradrenalina basi | Norepinephrine bitartrate |
| 00127502015 | Noradrenalina biol | Norepinephrine bitartrate |
| 00127502025 | Noradrenalina braun | Norepinephrine bitartrate |
| 00127502050 | Noradrenalina Combino pharm | Norepinephrine bitartrate |
| 00127502067 | Noradrenalina Generis | Norepinephrine bitartrate |
| 00127501008 | Noradrenalina Max vision | Norepinephrine |
| 00127502029 | Noradrenalina Normon | Norepinephrine bitartrate |
| 00127502089 | Noradrenalina novophar | Norepinephrine bitartrate |
| 00127502016 | Noradrenalina richet | Norepinephrine bitartrate |
| 00127502033 | Noradrenalina tartrato | Norepinephrine bitartrate |
| 00127502092 | Noradrenalina tartrato aguettant | Norepinephrine bitartrate |
| 00127501002 | Noradrenaline | Norepinephrine |
| 00127502021 | Noradrenaline | Norepinephrine bitartrate |
| 00127504003 | Noradrenaline | Norepinephrine bitartrate monohydrate |
| 00127502097 | Noradrenaline (Norpinephrine) | Norepinephrine bitartrate |
| 00127502055 | Noradrenaline acid tartrate anhydrous | Norepinephrine bitartrate |
| 00127502012 | Noradrenaline aguettant | Norepinephrine bitartrate |
| 00127502079 | Noradrenaline bnm | Norepinephrine bitartrate |
| 00127503009 | Noradrenaline dl-form hydrochloride | Norepinephrine hydrochloride |
| 00127502046 | Noradrenaline Hospira | Norepinephrine bitartrate |
| 00127503010 | Noradrenaline hydrochloride | Norepinephrine hydrochloride |
| 00127503011 | Noradrenaline hydrochloride, dl-form | Norepinephrine hydrochloride |
| 00127502088 | Noradrenaline kabi | Norepinephrine bitartrate |
| 00127502078 | Noradrenaline medis | Norepinephrine bitartrate |
| 00127502026 | Noradrenaline Merck | Norepinephrine bitartrate |
| 00127502085 | Noradrenaline mylan | Norepinephrine bitartrate |
| 00127502072 | Noradrenaline myx | Norepinephrine bitartrate |
| 00127502037 | Noradrenaline PCH | Norepinephrine bitartrate |
| 00127502027 | Noradrenaline Renaudin | Norepinephrine bitartrate |
| 00127502059 | Noradrenaline saiph | Norepinephrine bitartrate |
| 00127502091 | Noradrenaline Sintetica | Norepinephrine bitartrate |
| 00127502074 | Noradrenaline tartrate renaudin | Norepinephrine bitartrate |

<u>CCI</u>

PPD




Master Statistical Analysis Plan

| Drug code | Product Name | Active Ingredients |
|---|---|---|
| 00127502056 | Noradrenalini tartras | Norepinephrine bitartrate |
| 00127501012 | Noradrenalinum | Norepinephrine |
| 00127502053 | Noradria | Norepinephrine bitartrate |
| 00127502047 | Norages | Norepinephrine bitartrate |
| 00127502060 | Noraline | Norepinephrine bitartrate |
| 00127502069 | Norbit | Norepinephrine bitartrate |
| 00127502077 | Norene | Norepinephrine bitartrate |
| 00127502044 | Norepin | Norepinephrine bitartrate |
| 00127502039 | Norepine | Norepinephrine bitartrate |
| 00127502035 | Norepinefrina | Norepinephrine bitartrate |
| 00127501014 | Norepinefrina | Norepinephrine |
| 00127502048 | Norepinefrina northia | Norepinephrine bitartrate |
| 00127502075 | Norepinefrina vitalis | Norepinephrine bitartrate |
| 00127502024 | Norepinefrine | Norepinephrine bitartrate |
| 00127503003 | Norepinephrine | Norepinephrine hydrochloride |
| 00127502004 | Norepinephrine | Norepinephrine bitartrate |
| 00127501001 | Norepinephrine | Norepinephrine |
| 00127502001 | Norepinephrine Bitartrate | Norepinephrine bitartrate |
| 00127504001 | Norepinephrine bitartrate monohydrate | Norepinephrine bitartrate monohydrate |
| 00127503012 | Norepinephrine HCL | Norepinephrine hydrochloride |
| 00127503001 | Norepinephrine hydrochloride | Norepinephrine hydrochloride |
| 00127502093 | Norepinephrine sopharma | Norepinephrine bitartrate |
| 00127502057 | Norepinephrine tartrate | Norepinephrine bitartrate |
| 00127501013 | Norepinephrinum | Norepinephrine |
| 00127502019 | Norepirin | Norepinephrine bitartrate |
| 00127502082 | Noreprin | Norepinephrine bitartrate |
| 00127502052 | Norphed | Norepinephrine bitartrate |
| 00127501011 | Norpin | Norepinephrine |
| 00127502018 | Norpine | Norepinephrine bitartrate |
| 00127502096 | Northix | Norepinephrine bitartrate |
| 01872201009 | Novopressina-V | Vasopressin |
| 00003902061 | Oboi Epinephrine | Epinephrine hydrochloride |
| 00003901034 | Oftan adrenalin | Epinephrine |

CCI

PPD




Master Statistical Analysis Plan

| Drug code | Product Name | <b>Active Ingredients</b> |
|-------------|--------------------------|---------------------------|
| 00003901011 | Oftan-adrenalin | Epinephrine |
| 00360702107 | Oridop | Dopamine hydrochloride |
| 00003902009 | Orostat | Epinephrine hydrochloride |
| 00003901095 | Penepin | Epinephrine |
| 00003903041 | Pharma Q Adrenaline | Epinephrine bitartrate |
| 00360702188 | Pharma q dopamine | Dopamine hydrochloride |
| 00003903050 | Pharma-q adrenaline | Epinephrine bitartrate |
| 00003902050 | Phenylephrin | Epinephrine hydrochloride |
| 00003901080 | Phinev | Epinephrine |
| 00127502032 | Pidram | Norepinephrine bitartrate |
| 00003901036 | Pinadrina | Epinephrine |
| 01872202006 | Pitressin | Vasopressin tannate |
| 01872201002 | Pitressin | Vasopressin |
| 01872201006 | Pitressin aqueous | Vasopressin |
| 01872201013 | Pitressin tanato | Vasopressin |
| 01872202004 | Pitressin Tannat in Oil | Vasopressin tannate |
| 01872202002 | Pitressin tannate | Vasopressin tannate |
| 01872201011 | Pitressin tannate | Vasopressin |
| 01872202007 | Pitressin tannate in oil | Vasopressin tannate |
| 01872201015 | Pitressin tannate in oil | Vasopressin |
| 01872202003 | Pitressin tannate oil | Vasopressin tannate |
| 00493402008 | Posiject | Dobutamine hydrochloride |
| 00003901056 | Posumin | Epinephrine |
| 00360702032 | Predopa | Dopamine hydrochloride |
| 00360702132 | Predopa Kyowa | Dopamine hydrochloride |
| 00360702125 | Predopa merck hoei | Dopamine hydrochloride |
| 01872201003 | Pressyn | Vasopressin |
| 01872201007 | Pressyn ar | Vasopressin |
| 00127502009 | Pridam | Norepinephrine bitartrate |
| 00003901067 | Primatene | Epinephrine |
| 00003901060 | Primatene mist | Epinephrine |
| 00360702108 | Proinfark | Dopamine hydrochloride |
| 00493402154 | Pusogard | Dobutamine hydrochloride |

<u>CCI</u>

PPD




| Drug code | Product Name | Active Ingredients |
|---|---|---|
| 00127502066 | Q phrine | Norepinephrine bitartrate |
| 00003903021 | Racepinephrine | Epinephrine bitartrate |
| 00003902006 | Racord | Epinephrine hydrochloride |
| 00127502062 | Radline | Norepinephrine bitartrate |
| 00127504002 | Raivas | Norepinephrine bitartrate monohydrate |
| 00493402110 | Retamex | Dobutamine hydrochloride |
| 00360702006 | Revimine | Dopamine hydrochloride |
| 00360702015 | Revivan | Dopamine hydrochloride |
| 00003903017 | S2 | Epinephrine bitartrate |
| 00003902036 | S-2 | Epinephrine hydrochloride |
| 00360702018 | Sabax dopamine | Dopamine hydrochloride |
| 00127502080 | Sandine | Norepinephrine bitartrate |
| 00003903012 | Sanepi | Epinephrine bitartrate |
| 00127502070 | Seladrenalin | Norepinephrine bitartrate |
| 00360702153 | Seminiet | Dopamine hydrochloride |
| 00003901008 | Simplene | Epinephrine |
| 00127502076 | Sinora | Norepinephrine bitartrate |
| 00127502095 | Softamicid | Norepinephrine bitartrate |
| 00003902067 | Spinefe | Epinephrine hydrochloride |
| 00493402084 | Starzen | Dobutamine hydrochloride |
| 00127502054 | Stenor | Norepinephrine bitartrate |
| 00127502031 | Steradin | Norepinephrine bitartrate |
| 00360702157 | Sterile dopamine concentrate | Dopamine hydrochloride |
| 01872201014 | Stimate | Vasopressin |
| 00003901090 | Supradin | Epinephrine |
| 00003901005 | Suprarenin | Epinephrine |
| 00003902029 | Suprarenin | Epinephrine hydrochloride |
| 00003901074 | Surgident | Epinephrine |
| 00003902002 | Sus-phrine | Epinephrine hydrochloride |
| 00003901038 | Sus-phrine | Epinephrine |
| 00003901092 | Symjepi | Epinephrine |
| 00360702055 | Taiadopa | Dopamine hydrochloride |
| 00360702017 | Tensamin | Dopamine hydrochloride |

CCI

PPD




| Drug code | Product Name | Active Ingredients |
|-------------|----------------------------|---------------------------|
| 00493402042 | Toburex | Dobutamine hydrochloride |
| 00003901023 | Tonogen | Epinephrine |
| 00360702154 | Tronjin | Dopamine hydrochloride |
| 00360702089 | Tropin | Dopamine hydrochloride |
| 00360702046 | Tsurudopami | Dopamine hydrochloride |
| 00127502099 | Turktipsan noradrenalin | Norepinephrine bitartrate |
| 00003901057 | Twinject | Epinephrine |
| 00360702091 | Udopa | Dopamine hydrochloride |
| 00360702145 | Upamine | Dopamine hydrochloride |
| 00360702121 | Uramin | Dopamine hydrochloride |
| 00493402064 | Utamine | Dobutamine hydrochloride |
| 00003902003 | Vaponefrin | Epinephrine hydrochloride |
| 00003902020 | Vaponefrin hisamitsu | Epinephrine hydrochloride |
| 00003902021 | Vaponefrin tokyo mi shokai | Epinephrine hydrochloride |
| 01872201023 | Vascel | Vasopressin |
| 00127502022 | Vascon | Norepinephrine bitartrate |
| 00003903025 | Vasocon | Epinephrine bitartrate |
| 01872201025 | Vasopar | Vasopressin |
| 01872201017 | Vasopin | Vasopressin |
| 01872201001 | Vasopressin | Vasopressin |
| 01872201010 | Vasopressin injection | Vasopressin |
| 01872201022 | Vasopressin sandoz | Vasopressin |
| 01872201005 | Vasopressin tannat | Vasopressin |
| 01872202005 | Vasopressin tannat | Vasopressin tannate |
| 01872202001 | Vasopressin tannate | Vasopressin tannate |
| 01872201019 | Vasopressina | Vasopressin |
| 01872201004 | Vasopressine | Vasopressin |
| 01872202008 | Vasopressini tannas | Vasopressin tannate |
| 01872201021 | Vasostrict | Vasopressin |
| 00360702122 | Vidopa | Dopamine hydrochloride |
| 00003901053 | Weradren | Epinephrine |
| 00360702155 | Yaelista | Dopamine hydrochloride |
| 00360702049 | Yaelista mita | Dopamine hydrochloride |

CCI

PPD






Amgen Inc Master Protocol COV-01 

Master Statistical Analysis Plan

| Drug code | Product Name | Active Ingredients |
|-------------|--------------|------------------------|
| 00360702142 | Zetarina | Dopamine hydrochloride |

### **APPENDIX 5 LABORATORY ASSESSMENTS**

### Hematology (SI unit)

- Platelets count (x10E9/L)
- Hemoglobin (g/L)
- White blood cell (WBC) count total (x10E9/L)
- Absolute neutrophils count (x10E9/L)
- Absolute lymphocyte count (x10E9/L)
- Absolute monocyte count (x10E9/L)
- Absolute eosinophils count (x10E9/L)
- Absolute basophils count (x10E9/L)

- Relative neutrophils count (%)
- Relative lymphocyte count (%)
- Relative monocyte count (%)
- Relative eosinophils count (%)
- Relative basophils count (%)

### Coagulation (SI unit)

- D-dimer (mg/Lmg/L)
- Fibrinogen (g/L)
- Activated partial thromboplastin time (s)
- Prothrombin time (PT) (s)
- International normalized ratio (INR)

- C-reactive protein (CRP) (mg/L)
- Ferritin (μg/L)
- Lactate dehydrogenase (LDH) (IU/L)
- Procalcitonin (μg/L)

PPD




o Triglycerides (mmol/L)

| Ch | emi | stry (SI unit) | | |
|---|---|---|---|---|
| • | Ge | neral | | |
| | 0 | Potassium (mmol/L) | 0 | Phosphate (mmol/L) |
| | 0 | Sodium (mmol/L) | 0 | Bicarbonate (mmol/L) |
| | 0 | Calcium (mmol/L) | 0 | Creatinine (µmol/L) |
| | 0 | Magnesium (mmol/L) | 0 | Glucose (mmol/L) |
| • | Liv | ver Function Tests | | |
| | 0 | Alkaline phosphatase (ALP) (IU/L) | 0 | Alanine transaminase (ALT) (IU/L) |
| | 0 | Total bilirubin (µmol/L) | 0 | Gamma glutamyl transferase (GGT) (IU/L) |
| | 0 | Aspartate transaminase (AST) (IU/L) | | |
| • | Ca | rdiac Panel | | |
| | 0 | Creatine kinase (CK) (IU/L) | 0 | Troponin I (μg/L) |
| | 0 | CK MB isoenzyme fraction of CK (IU/L) | 0 | Troponin T (μg/L) |

## APPENDIX 6 CTCAE TOXICITY GRADE, VERSION 5.0

https://ctep.cancer.gov/protocolDevelopment/electronic applications/ctc.htm (accessed on 22-Apr-2020)

| CTCAE Term | Laboratory Test | No Event | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|---|---|
| Platelet count decreased | Platelet count (x10E9/L) | ≥LLN | ≥ 75 x 10E9/L<br>- < LLN | ≥ 50 -<br>< 75 x 10E9/L | ≥ 25 -<br>< 50 x 10E9/L | < 25 x 10E9/L | n/a |
| Anemia | Hemoglobin (g/L) | ≥LLN | ≥ 100 g/L -<br>< LLN | ≥ 80 -<br>< 100 g/L | < 80 g/L | n/a | n/a |
| Hemoglobin increased | Hemoglobin (g/L) | No increase from baseline | Increase from baseline > 0 - ≤ 20 g/L | Increase from baseline > 20 - $\leq$ 40 g/L | Increase from baseline > 40 g/L | n/a | n/a |
| White blood cell (WBC) decreased | WBC (x 10E9/L) | ≥LLN | ≥ 3.0 x 10E9/L<br>- < LLN | ≥ 2.0 - < 3.0 x 10E9/L | ≥ 1.0 - < 2.0 x<br>10E9/L | < 1.0 x 10E9/L | n/a |
| Leukocytosis | WBC (x 10E9/L) | ≤ 100 x<br>10E9/L | n/a | n/a | > 100 x 10E9/L | n/a | n/a |
| Absolute neutrophils count decreased | Absolute neutrophils count (x 10E9/L) | ≥LLN | ≥ 1.5 x 10E9/L<br>- < LLN | ≥ 1.0 -<br>< 1.5 x 10E9/L | ≥ 0.5 - < 1.0 x<br>10E9/L | < 0.5 x 10E9/L | n/a |

PPD




| CTCAE Term | Laboratory Test | No Event | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|---|---|
| Absolute lymphocytes count decreased | Absolute lymphocytes count (x 10E9/L) | ≥LLN | ≥ 0.8 x 10E9/L<br>-< LLN | ≥ 0.5 -<br>< 0.8 x 10E9/L | ≥ 0.2 -<br>< 0.5 x 10E9/L | < 0.2 x 10E9/L | n/a |
| Absolute lymphocytes count increased | Absolute lymphocytes count (x 10E9/L) | ≤ 4 x 10E9/L | n/a | > 4 -<br>≤ 20 x 10E9/L | > 20 x 10E9/L | n/a | n/a |
| Eosinophilia | Absolute eosinophils count (x 10E9/L) | ≤ ULN or<br>≤ Baseline | > ULN and<br>> Baseline | n/a | n/a | n/a | n/a |
| Fibrinogen decreased | Fibrinogen (g/L) | ≥ LLN if baseline normal; no decrease from baseline if baseline abnormal | ≥ 0.75 - < 1 x LLN if baseline normal; > 0 - < 25% decrease from baseline if baseline abnormal | ≥ 0.5 - < 0.75 x LLN if baseline normal; ≥ 25 - < 50% decrease from baseline if baseline abnormal | ≥ 0.25 - < 0.5 x LLN if baseline normal; ≥ 50 - < 75% decrease from baseline if baseline abnormal | < 0.25 x LLN if baseline normal; ≥ 75% decrease from baseline if baseline abnormal | |
| Activated partial thromboplastin time (aPTT) prolonged | aPTT (s) | ≤ULN | > ULN −<br>≤ 1.5 x ULN | > 1.5 −<br>≤ 2.5 x ULN | > 2.5 ULN | n/a | n/a |




| CTCAE Term | Laboratory Test | No Event | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|---|---|
| International normalized ratio (INR) increased | INR | ≤ 1.2 if not on anticoagulant; ≤ baseline if on anticoagulant | > 1.2 -≤1.5 if<br>not on<br>anticoagulant;<br>> baseline -<br>≤1.5 x baseline<br>if on<br>anticoagulant | > $1.5 - \le 2.5$ if<br>not on<br>anticoagulant;<br>> $1.5 - \le 2.5$ x<br>baseline if on<br>anticoagulant | > 2.5 if not on<br>anticoagulant;<br>> 2.5 x baseline<br>if on<br>anticoagulant | n/a | n/a |
| Blood lactate<br>dehydrogenase (LDH)<br>increased | LDH (IU/L) | ≤ULN | > ULN | n/a | n/a | n/a | n/a |
| Hyperkalemia | Potassium (mmol/L) | ≤ULN | > ULN –<br>≤ 5.5 mmol/L | > 5.5 –<br>≤ 6.0 mmol/L | > 6.0 –<br>≤ 7.0 mmol/L | > 7.0 mmol/L | n/a |
| Hypokalemia | Potassium (mmol/L) | ≥LLN | ≥ 3.0 mmol/L −<br>< LLN;<br>asymptomatic;<br>no intervention<br>indicated | ≥ 3.0 mmol/L −<br>< LLN;<br>symptomatic;<br>intervention<br>indicated | ≥ 2.5 - < 3.0 mmol/L | < 2.5 mmol/L | n/a |




| CTCAE Term | Laboratory Test | No Event | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|---|---|
| Hypernatremia | Sodium (mmol/L) | ≤ULN | > ULN - ≤ 150<br>mmol/L | > 150 −<br>≤ 155 mmol/L | > 155 −<br>≤ 160 mmol/L | > 160 mmol/L | n/a |
| Hyponatremia | Sodium (mmol/L) | ≥LLN | ≥ 130 mmol/L<br>- < LLN | ≥ 125 -<br>< 130 mmol/L<br>and<br>asymptomatic | $\geq$ 120 -<br>< 125 mmol/L<br>or<br>$\geq$ 125 -<br>< 130 mmol/L<br>and<br>symptomatic | < 120 mmol/L | n/a |
| Hypermagnesemia | Magnesium (mmol/L) | ≤ULN | > ULN −<br>≤ 1.23 mmol/L | n/a | > 1.23 −<br>≤ 3.30 mmol/L | > 3.30 mmol/L | n/a |
| Hypomagnesemia | Magnesium (mmol/L) | ≥LLN | ≥ 0.5 mmol/L − < LLN | ≥ 0.4 -<br>< 0.5 mmol/L | ≥ 0.3 -<br>< 0.4 mmol/L | < 0.3 mmol/L | n/a |
| Blood bicarbonate decreased | Bicarbonate (mmol/L) | ≥LLN | < LLN | n/a | n/a | n/a | n/a |


| CTCAE Term | Laboratory Test | No Event | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|---|---|
| Creatinine increased | Creatinine (µmol/L) | ≤ULN | > ULN –<br>≤ 1.5 x ULN | > $1.5 - $<br>$\leq 3.0 \text{ x ULN}$<br>or<br>> $1.5 - \leq 3.0 \text{ x}$<br>baseline | > 3.0 -<br>≤ 6.0 x ULN<br>or<br>> 3.0 x baseline | > 6.0 x ULN | n/a |
| Hypoglycemia | Glucose (mmol/L) | ≥LLN | ≥ 3.0 mmol/L − < LLN | ≥ 2.2 - < 3.0 mmol/L | ≥ 1.7 - < 2.2 mmol/L | < 1.7 mmol/L | n/a |
| Alkaline phosphatase (ALP) increased | ALP (U/L) | ≤ ULN if baseline normal; ≤ 2.0 x baseline if baseline abnormal | > ULN -<br>≤ 2.5 x ULN if<br>baseline<br>normal;<br>> 2.0 -<br>≤ 2.5 x baseline<br>if baseline<br>abnormal | > 2.5 −<br>≤ 5.0 x ULN if<br>baseline<br>normal;<br>> 2.5 −<br>≤ 5.0 x baseline<br>if baseline<br>abnormal | > 5.0 -<br>$\le 20.0 \text{ x ULN if}$<br>baseline<br>normal;<br>$> 5.0 - \le 20.0 \text{ x}$<br>baseline if<br>baseline<br>abnormal | > 20.0 x ULN if baseline normal; > 20.0 x baseline if baseline abnormal | n/a |


| CTCAE Term | Laboratory Test | No Event | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|---|---|
| Blood bilirubin | Total bilirubin | ≤ULN if | > ULN - | > 1.5 - | $> 3.0 - \le 10.0 \text{ x}$ | > 10.0 x ULN if | n/a |
| increased | (µmol/L) | baseline | $\leq$ 1.5 x ULN if | $\leq$ 3.0 x ULN if | ULN if baseline | baseline | |
| | | normal; | baseline | baseline | normal; | normal; | |
| | | ≤ baseline if | normal; | normal; | $> 3.0 - \le 10.0 \text{ x}$ | > 10.0 x | |
| | | baseline | > baseline - ≤ | $> 1.5 - \le 3.0 \text{ x}$ | baseline if | baseline if | |
| | | abnormal | 1.5 x baseline | baseline if | baseline | baseline | |
| | | | if baseline | baseline | abnormal | abnormal | |
| | | | abnormal | abnormal | | | |
| Aspartate transaminase | AST (U/L) | ≤ULN if | > ULN - | > 3.0 - | $> 5.0 - \le 20.0 \text{ x}$ | > 20.0 x ULN if | n/a |
| (AST) increased | | baseline | $\leq$ 3.0 x ULN if | $\leq$ 5.0 x ULN if | ULN if baseline | baseline | |
| | | normal; | baseline | baseline | normal; | normal; | |
| | | ≤ 1.5 x | normal; | normal; | $> 5.0 - \le 20.0 \text{ x}$ | > 20.0 x | |
| | | baseline if | $> 1.5 - \le 3.0 \text{ x}$ | $> 3.0 - \le 5.0 \text{ x}$ | baseline if | baseline if | |
| | | baseline | baseline if | baseline if | baseline | baseline | |
| | | abnormal | baseline | baseline | abnormal | abnormal | |
| | | | abnormal | abnormal | | | |


| CTCAE Term | Laboratory Test | No Event | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|---|---|
| Alanine transaminase | ALT (U/L) | ≤ULN if | > ULN - | > 3.0 - | $> 5.0 - \le 20.0 \text{ x}$ | > 20.0 x ULN if | n/a |
| (ALT) increased | | baseline | $\leq$ 3.0 x ULN if | $\leq$ 5.0 x ULN if | ULN if baseline | baseline | |
| | | normal; | baseline | baseline | normal; | normal; | |
| | | ≤ 1.5 x | normal; | normal; | $> 5.0 - \le 20.0 \text{ x}$ | > 20.0 x | |
| | | baseline if | $> 1.5 - \le 3.0 \text{ x}$ | $> 3.0 - \le 5.0 \text{ x}$ | baseline if | baseline if | |
| | | baseline | baseline if | baseline if | baseline | baseline | |
| | | abnormal | baseline | baseline | abnormal | abnormal | |
| | | | abnormal | abnormal | | | |
| Gamma glutamyl | GGT (U/L) | ≤ULN if | > ULN - | > 2.5 - | $> 5.0 - \le 20.0 \text{ x}$ | > 20.0 x ULN if | n/a |
| transferase (GGT) | | baseline | $\leq$ 2.5x ULN if | $\leq$ 5.0 x ULN if | ULN if baseline | baseline | |
| increased | | normal; | baseline | baseline | normal; | normal; | |
| | | ≤ 2.0 x | normal; | normal; | $> 5.0 - \le 20.0 \text{ x}$ | > 20.0 x | |
| | | baseline if | > 2.0 - | > 2.5 - | baseline if | baseline if | |
| | | baseline | $\leq$ 2.5 x baseline | $\leq$ 5.0 x baseline | baseline | baseline | |
| | | abnormal | if baseline | if baseline | abnormal | abnormal | |
| | | | abnormal | abnormal | | | |
| CPK increased | Creatine kinase (U/L) | ≤ULN | > ULN - | > 2.5 - | > 5 - | > 10 x ULN | n/a |
| | | | ≤ 2.5 x ULN | ≤5 x ULN | ≤ 10 x ULN | | |




Amgen, Inc. Master Protocol COV-01 

Master Statistical Analysis Plan

| CTCAE Term | Laboratory Test | No Event | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|---|---|
| Hypertriglyceridemia | Triglycerides | ≤ 1.71 mmol/L | > 1.71 – | > 3.42 - | > 5.70 - | > 11.40 mmol/L | n/a |
| | (mmol/L) | | $\leq$ 3.42 mmol/L | $\leq$ 5.70 mmol/L | $\leq 11.40 \text{ mmol/L}$ | | |

CCI PPD

Version Number: Version Date: Amendment 1, v1.0 23Apr2021

CCI



| Certificate Of Completion | | |
|---|---|---|
| PPD | | Status: Completed |
| PPD | | |
| Record Tracking | | |
| Status: Original<br>4/23/2021 4:13:46 PM | Holder: PPD | Location: DocuSign |
| Signer Events | Signature | Timestamp |

| Signer Events | Signature | Timestamp |
|---------------|-----------|-----------|
| PPD | | |

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent Certified Delivered Signing Complete Completed | Hashed/Encrypted Security Checked Security Checked Security Checked | 4/23/2021 4:15:59 PM<br>4/23/2021 9:22:08 PM<br>4/23/2021 9:23:12 PM<br>4/23/2021 9:23:12 PM |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disclosure | | |

### CONSENT TO ELECTRONIC DELIVERY AND EXECUTION OF DOCUMENTS

From time to time, ("we" or "us") may provide you certain written contracts, notices, disclosures, authorizations, acknowledgements or other documents (collectively, the "Documents") electronically. Please read this consent form carefully. It explains the terms and conditions under which such Documents are provided by us and executed by you electronically through your DocuSign, Inc. ("DocuSign") user account. If you consent to the delivery and execution of such Documents electronically, please click the "I Agree" button.

### **Documents** will be sent to you electronically

If you consent to electronic delivery, Documents will be sent to your DocuSign user account. You may request a paper copy of documents previously made available through your DocuSign user account, but an additional charge may be incurred. Alternatively, you can download and print documents sent to your DocuSign user account. Unless otherwise noted, you can access a Document up to 30 days from the date we first sent the Document to you.

### Withhold Consent or Withdrawing Consent to Electronic Delivery

If you withhold consent to electronic delivery or execution, or withdraw your consent at a later date, all Documents will be sent to your mailing address following our receipt of notice of such action. The following sections explain the consequences of withholding or withdrawing your consent to electronic delivery and execution of Documents, and also the procedures you must follow in order to effectuate delivery to your mailing address.

### **Consequences of Withdrawing Consent**

By electing to only receive and execute Documents sent to your mailing address, we will not be able to carry out transactions or services as efficiently. For instance, some transactions or services require your express consent. We can perform these transaction or services only if we first receive an acknowledgement that indicates you received and consent to the Document related to the proposed transaction or service.

To withhold consent now or withdraw consent at a later date, please sign DocuSign's "Withdraw Consent" form on the signing page of your DocuSign user account. This will indicate that you have withdrawn your consent to receive Documents electronically. Once you sign the "Withdraw Consent" form, you will no longer be able to use your DocuSign user account to execute Documents electronically and we will send Documents to your mailing address. Withdrawal of consent does not affect the validity of any Documents previously executed electronically prior to such withdrawal of Consent. In addition, should you execute any Documents electronically, your execution of such Documents shall indicate your continued consent to execute such Documents electronically.

### How to contact **CC**

If you would like us to send the Documents to a different e-mail address, request paper copies of Documents you have previously received electronically, or withdraw your consent to receive electronic documents, please follow the instructions below. If you have any other questions, please contact: CCI

### 1. To advise ccl of your new e-mail address

If you would like your Documents sent to a different e-mail address, you must send an e-mail message to column and the send and e-mail please state the following: (i) your previous e-mail address, and (ii) your new e-mail address. No other information is required.

In addition, you must notify DocuSign of your new e-mail address. Please log into your DocuSign user account, and follow the instructions to update your e-mail address.

### 2. To request paper copies from CCI

To request paper copies of Documents you have received previously through your DocuSign user account, send an e-mail to CCI

In the body of the e-mail please state the following: (i) your e-mail address, (ii) full name, (iii) U.S. Postal address, and (iv) telephone number. Additional charges may apply for such paper copies.

### 3. To withdraw your consent with CC

To withdraw your consent to receiving and executing Documents in an electronic format, you may do one of the following:

i. decline to sign a document from within your DocuSign user account, and on the subsequent page, select the check-box indicating you wish to withdraw your consent; or ii. send us an e-mail to CCI and and in the body of such request you must state your e-mail, full name, US Postal Address, telephone number, and account number. No additional information is necessary.

### Required hardware and software

| Operating Systems: | Windows® 2000, Windows® XP, Windows Vista®; Mac OS® X |
|---|---|
| Browsers: | <ul> <li>Internet Explorer (Windows Only) 8.0 or above – compatibility mode is supported only for 9.0 and above.</li> <li>Windows Edge Current Version</li> <li>Mozilla Firefox Current Version</li> <li>Safari (Mac OS only) 6.2 or above</li> <li>Google Chrome Current Version</li> </ul> |
| PDF Reader: | Acrobat® or similar software may be required to view and print PDF files |
| Screen Resolution: | 1024 x 768 Recommended |
| Enabled Security Settings: | Allow per session cookies |
| Mobile Signing: | <ul><li>Apple iOS 7.0 or above</li><li>Android 4.0 or above</li></ul> |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, we will provide you with an e-mail message at the e-mail address we have on file for you at the time the hardware and software requirements are revised.

Pre-release (e.g. beta) versions of operating systems and browsers are not supported.

### Acknowledging your access and consent to receive materials electronically

To confirm you can access this information electronically and that you consent to receiving and executing Documents electronically on the terms and conditions described above, please let us know by clicking the "I Agree" button.

By clicking the "I Agree" button, you confirm that

- You can access and read this Consent To Electronic Delivery and Execution of Documents; and
- You can print on paper the disclosure or save or send the disclosure to a place where you can print it, for future reference and access; and
- Until or unless you notify occur as described above, you consent to the delivery and execution of Documents electronically.

## COV-01-001 STATISTICAL ANALYSIS PLAN

INDUSTRY ALLIANCE PLATFORM TRIAL TO ASSESS THE EFFICACY AND SAFETY OF MULTIPLE CANDIDATE AGENTS FOR THE TREATMENT OF COVID-19 IN HOSPITALIZED PATIENTS

**SUB-PROTOCOL NUMBER: COV-01-001** 

SUB-PROTOCOL FOR CANDIDATE AGENT: LANADELUMAB-IV

**AUTHOR: PPD** 

VERSION NUMBER AND DATE: AMENDMENT 3 v1.0, 23-Jul-2021



# TAKEDA SUB-PROTOCOL STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

Takeda sub-protocol COV-01-001 Statistical Analysis Plan (SAP) Amendment 3 v1.0 (dated 23-Jul-2021).

| | Name | Signature | Date (DD-Mmm-YYYY) |
|-----------|------|-----------|--------------------|
| Author: | PPD | PPD | |
| Position: | PPD | | |
| Company: | CCI | | |

Upon review of this document, the undersigned approves this version of the sub-protocol COV-01-001 SAP, authorizing that the content is acceptable for the reporting specific to this sub-protocol.

| | Name | Signature | Date (DD-Mmm-YYYY) |
|---------------|--------|-----------|--------------------|
| Approved by: | PPD | PPD | |
| Position: | PPD | | |
| Company: | CCI | | |
| On behalf of: | PPD | | |
| Position: | PPD | | |
| Company: | CCI | | |
| Approved by: | PPD | PPD | |
| Position: | PPD | | |
| Company: | Takeda | | |

| CCI | | |
|-----|----------------------------------|----------------------------------|
| PPD | Version Number:<br>Version Date: | Amendment 3, v1.0<br>23-Jul-2021 |
| CCI | | |

## **MODIFICATION HISTORY**

| Unique<br>Identifier for<br>this Version | Date of the<br>Document<br>Version | Author | Significant Changes from Previous Version |
|---|---|---|---|
| Final, v1.0 | 14-Dec-2020 | PPD | Not Applicable – First Version |
| Amendment 1, v1.0 | 27-Apr-2021 | PPD | Updated COV-01-001 sub-protocol version on which this subprotocol SAP is based from version 1.2, dated 26Oct2020, to version 2.0, dated 14Apr2021 Update title of Sections 11 and 13 to be in line with Master SAP; Added a subgroup that will be used to perform supportive analysis for selected safety data and related additional supportive analysis; Added the risk difference of the overall incidence rates of having any treatmentemergent AESI between the treatment groups will be presented along with its 95% two-sided Wald CI; Added Appendices 1 and 2. |



| Unique<br>Identifier for<br>this Version | Date of the<br>Document<br>Version | Author | Significant Changes from Previous Version |
|---|---|---|---|
| Amendment 2, v1.0 | 24-Jun-2021 | PPD | Specified that the two Interim Analyses (IAs) and Primary Analysis at Day 29 will not be performed for this sub-protocol since enrollment into COV-01-001 sub-protocol was early terminated by the Sponsor on 03-May-2021 i.e., before the trigger of each of these analyses was met. Exception of summary statistics for the primary efficacy, key secondary, and other secondary efficacy endpoints, removed all planned efficacy analyses given that 1) enrollment into COV-01-001 sub-protocol was early terminated by the Sponsor on 03-May-2021, 2) number of patients to be included in COV-01-001 sub-protocol final analysis, and 3) an abbreviated Clinical Study Report will be created for this sub-protocol. Added two-sided 95% exact binomial Confidence Interval within each treatment arm, when applicable. Removed the additional subgroup analyses that were to be performed as supportive analysis for selected safety data. |
| Amendment 3, v1.0 | 23-Jul-2021 | PPD | Updated the definition of the Shared Placebo<br>Arm |



## **TABLE OF CONTENTS**

| 1. | INTRODUCTION | 9 |
|---|---|---|
| 2. | STUDY OBJECTIVES | 9 |
| 3. | STUDY DESIGN | 9 |
| 3.1. | General Description | 9 |
| 3.2. | Schedule of Activities | 9 |
| 3.3. | Changes to Planned Analyses from Master Protocol and Sub-Protocol COV-01-001 | 9 |
| 4. | PLANNED ANALYSES | 10 |
| 4.1. | IDMC Safety Analyses | 10 |
| 4.2. | Interim Analyses | 10 |
| 4.3. | Primary Analysis | 10 |
| 4.4. | Final Analysis | 11 |
| <b>4.5.</b> 4.5. 4.5. | 12 112 2 20100 1 111001 2 2 2 | 11 |
| 5. | ANALYSIS SETS | 12 |
| 5.1. | Primary Analysis Set | 12 |
| 5.2. | Pharmacokinetic Analysis Set | 12 |
| 5.3. | Pharmacodynamic Analysis Set | 12 |
| 5.4. | Plasma Anti-Drug Antibody Analysis Set | 13 |
| 5.5. | Process for Analysis Set Assignment | 13 |
| CCL | | |

PPD

Version Number: Amendment 3, v1.0 Version Date: 23-Jul-2021

| 6. | GENERAL CONSIDERATIONS | 13 |
|---|---|---|
| 7. | STATISTICAL CONSIDERATIONS | 13 |
| 7.1. | Sample Size Calculation | 13 |
| 7.2. | Missing data | 13 |
| 7.3. | Statistical Tests | 14 |
| 7.4. | Multiple Comparisons/ Multiplicity | 14 |
| 7.5. | Multicenter Studies | 14 |
| 7.6. | Adjustments for Covariates and Factors to be Included in Analyses | 14 |
| 7.7. | Examination of Subgroups | 14 |
| 7.8. | Software Version | 14 |
| 8. | OUTPUT PRESENTATIONS | 14 |
| 9. | DISPOSITION AND WITHDRAWALS | 15 |
| 10. | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 15 |
| 11. | DISEASE HISTORY | 15 |
| 12. | MEDICAL HISTORY | 15 |
| 13. | PRIOR AND CONCOMITANT MEDICATIONS | 15 |
| 14. | EXPOSURE TO STUDY DRUG | 15 |
| 14.1. | Derivations | 17 |
| 15. | COMPLIANCE WITH STUDY DRUG | 17 |
| CCI<br>PPD | Version Number: A Version Date: | mendment 3, v1.0<br>23-Jul-2021 |

| 15.1. | Derivations | 18 |
|---|---|---|
| 16. EI | FFICACY ENDPOINTS | 19 |
| 16.1. | Primary Efficacy | 19 |
| 16.1.1. | Time to Confirmed Clinical Recovery through Day 29, without Re-Hospitalization Th | |
| | Day 29 | 19 |
| 16.1.2. | Missing Data Imputation Method for Primary Efficacy Endpoint | 19 |
| 16.1.3. | Main Analysis of Primary Efficacy Endpoint | |
| 16.1.4. | Sensitivity Analyses for Primary Efficacy Endpoint | |
| 16.1.5. | Supplementary Analyses for Primary Efficacy Endpoint | 20 |
| 16.2. | Secondary Efficacy | 20 |
| 16.2.1. | Secondary Efficacy Endpoints | |
| 16.2. | | |
| 16.2. | | |
| | Ordinal Scale at Day 29 | |
| 16.2. | 1.3. Incidence of All-Cause Mortality through Day 29 | 21 |
| 16.2. | | |
| | at Days 8, 15, and 29 | |
| 16.2.1 | 1 | |
| 16.2.1 | | |
| 16.2.1 | | |
| 16.2.1<br>16.2.1 | | |
| 16.2.2. | | |
| 16.2.2. | Missing Data Imputation Method for Secondary Efficacy Endpoints | |
| 16.2.2 | <b>7</b> 1 | |
| 16.2.3. | Main Analysis of Secondary Efficacy Endpoints | |
| 16.2.3 | | |
| 16.2.3 | | |
| 16.2.4. | Sensitivity Analyses for Secondary Efficacy Endpoints | |
| 16.2.5. | Supplementary Analyses for Secondary Efficacy Endpoints | |
| 16.3. | Exploratory Efficacy | 23 |
| 16.4. | Additional Efficacy | 23 |
| 16.5. | Interim Analysis | 23 |
| | · | |
| 17. SA | AFETY ENDPOINTS | 23 |
| 17.1. | Adverse Events | 24 |
| 17.1.1. | Adverse Events of Special Interest | |
| CCI | | |
| PPD | Version Number: Amendme | |
| | Version Date: 23 | -Jul-2021 |

| 17.2. | Laboratory Evaluations | 24 |
|-------|------------------------------------------|----|
| 17.3. | Vital Signs | 24 |
| 17.4. | ECG Evaluation | 24 |
| 17.5. | Physical Examination | 25 |
| 18. | PHARMACOKINETICS | 25 |
| 19. | PHARMACODYNAMICS | 26 |
| 20. | PLASMA ANTI-DRUG ANTIBODY TESTING | 26 |
| 21. | DATA NOT SUMMARIZED OR PRESENTED | 26 |
| APP | ENDIX 1 HYPERSENSITIVITY REACTIONS | 27 |
| APP | ENDIX 2 EVENTS OF DISORDERED COAGULATION | 28 |

CCI

PPD

Version Number: An Version Date:

Amendment 3, v1.0 23-Jul-2021

CC

### 1. Introduction

This statistical analysis plan (SAP) describes the rules and conventions to be used in the presentation and analysis of data specific to sub-protocol COV-01-001 of master protocol COV-01. It describes the specific data to be summarized and analyzed, including specifics of the statistical analyses to be performed.

This sub-protocol SAP is based on version 2.0 of the sub-protocol COV-01-001, dated 14-Apr 2021.

For the rules and conventions to be used in the presentation and analysis of data common across all sub-protocols, refer to the Master COV-01 SAP.

### 2. STUDY OBJECTIVES

The study objectives are described in the Master COV-01 SAP.

### 3. STUDY DESIGN

### 3.1. GENERAL DESCRIPTION

The general description is available in the Master COV-01 SAP.

### 3.2. SCHEDULE OF ACTIVITIES

The schedule of activities can be found in Section 1.2 of the sub-protocol COV-01-001.

# 3.3. CHANGES TO PLANNED ANALYSES FROM MASTER PROTOCOL AND SUB-PROTOCOL COV-01-001

Enrollment into sub-protocol COV-01-001 was prematurely terminated by the Sponsor on 03-May-2021 due issues with the administration of the study drug. In conformance with the Food and Drug Administration (FDA) Guidance for Submission of Abbreviated Report and Synopsis in Support of Marking Application, an abbreviated Clinical Study Report (CSR) will be written for this sub-protocol. As such, not all analyses planned in the master protocol



will be performed for sub-protocol COV-01-001 (refer to Section 4 for more details concerning the analyses to be performed for this sub-protocol).

Definition of the control arm (i.e., the shared placebo + standard of care [SoC] arm) was updated for this sub-protocol to minimize the randomization imbalance issue noted by the CC Unblinded Biostatistician and IDMC members at the time of CC (refer to Section 4.5).

### 4. PLANNED ANALYSES

The analyses initially planned to be performed are listed and described in the Master COV-01 SAP. However, the two Interim Analyses (IAs) for futility and Primary Analysis will not be performed for this sub-protocol since enrollment into sub-protocol COV-01-001 was early terminated by the Sponsor on 03-May-2021 (refer to Section 3.3 for additional details) i.e., before the trigger for each of these analyses was met. That is, the only analysis that will be performed, in addition to the monthly IDMC Safety analyses, is the final analysis after all patients who were ongoing at the time Sponsor early terminated this sub-protocol completed the study (Day 60 visit) or discontinued early from the study, whichever occurs first.

All outputs described in this sub-protocol SAP will be produced at the time of sub-protocol COV-01-001 final analysis.

### 4.1. IDMC SAFETY ANALYSES

Details are provided in the Master COV-01 SAP.

### 4.2. INTERIM ANALYSES

No IAs will be performed for this sub-protocol (refer to Section 4).

### 4.3. PRIMARY ANALYSIS

No primary analysis will be performed for this sub-protocol (refer to Section 4).



### 4.4. FINAL ANALYSIS

The final analysis for this sub-protocol will take place after:

- Sponsor Authorization of this SAP.
- Final database lock of the database including data from screen failed patients.
- Final database lock of the database of each sub-protocol contributing to the control arm of this sub-protocol (refer to Section 4.5).
- Final database lock of the database of this sub-protocol.

All planned analyses identified in this sub-protocol SAP will be performed by Biostatistics at the time of the final analysis of this sub-protocol.

### 4.5. SELECTION OF THE CONTROL ARM FOR AN ANALYSIS

### 4.5.1. IDMC SAFETY ANALYSES

Details are provided in Master SAP Section 4.5.

### 4.5.2. FINAL ANALYSIS

For final analysis of this sub-protocol, the control arm (also referred to as shared placebo + SoC arm) will include all patients randomized to the placebo arm of any sub-protocol before this sub-protocol was early terminated (refer to section 3.3) at a site at which:

- This sub-protocol was opened for enrollment.
- At least one patient was randomized to either this sub-protocol active (Lanadelumab- intra-venous [IV] + SoC) or placebo (placebo to Lanadelumab-IV + SoC) arms.

That is, patients that satisfy these criteria will be included in the control arm of this sub-protocol regardless of 1) whether patients was randomized before this sub-protocol was opened for enrollment at the site (that is, patients randomized after enrollment into COV-01-001 sub-protocol was early terminated will be excluded from the control



arm of this sub-protocol) and 2) patient's eligibility to this sub-protocol specific inclusion/exclusion criteria.

The purpose of this change from the Master SAP control arm definition (Master SAP Section 4.5) is to minimize the randomization imbalance issue noted by the CCI Unblinded Biostatistician and IDMC members at the time of

time this sub-protocol SAP was finalized, the randomization imbalance was estimated to be approximately 7:1 between this sub-protocol active and control arms, should the original control arm definition would have been retained for the final analysis of this sub-protocol.

### 5. ANALYSIS SETS

Analysis sets are described in the COV-01 Master SAP.

Additional analysis sets that are specific to sub-protocol COV-01-001 are described below:

### 5.1. PRIMARY ANALYSIS SET

The primary analysis set will include all randomized patients with a baseline clinical severity status of Grade 3 to 5 on the 8-point ordinal scale for clinical severity.

For displays and analyses based on the primary analysis set, patients will be classified according to the randomized treatment.

The main analyses of all efficacy endpoints will be performed on the primary analysis set.

### 5.2. PHARMACOKINETIC ANALYSIS SET

The pharmacokinetic (PK) analysis set will include patients from the safety analysis set (refer to Master COV-01 SAP Section 5.2) randomized to the Lanadelumab-(IV + SoC arm who have at least one measured concentration post dose of Lanadelumab-IV.

### 5.3. PHARMACODYNAMIC ANALYSIS SET

The pharmacodynamic (PD) analysis set will include patients from the safety analysis set (refer to Master COV-01



SAP Section 5.2) randomized to COV-01-001 sub-protocol (i.e., Lanadelumab-IV + Standard of Care (SoC) arm or Placebo to Lanadelumab-IV + SoC) who have at least one measured biomarker level post dose of Lanadelumab-IV (e.g., cHMWk, pKAL, etc.).

### 5.4. PLASMA ANTI-DRUG ANTIBODY ANALYSIS SET

The plasma anti-drug antibody (ADA) analysis set will include patients from the safety analysis set (refer to Master COV-01 SAP Section 5.2) randomized to COV-01-001 sub-protocol (i.e., Lanadelumab- IV + Standard of Care (SoC) arm or Placebo to Lanadelumab-IV + SoC) who have at least one evaluated ADA response.

### 5.5. PROCESS FOR ANALYSIS SET ASSIGNMENT

As the primary, PK, PD and ADA analysis sets are defined based on objective criteria only, the authorization of this sub-protocol SAP will stand for the agreement and authorization of the inclusion/exclusion of each patient in the primary, PK, PD and ADA analysis sets.

### 6. GENERAL CONSIDERATIONS

Details are provided in the Master COV-01 SAP.

### 7. STATISTICAL CONSIDERATIONS

### 7.1. SAMPLE SIZE CALCULATION

Details are provided in the Master COV-01 SAP.

### 7.2. MISSING DATA

Details are provided in the Master COV-01 SAP.



### 7.3. STATISTICAL TESTS

Not applicable since no statistical inferences will be performed for the final analysis of this sub-protocol (refer to Section 16).

### 7.4. MULTIPLE COMPARISONS/ MULTIPLICITY

Not applicable since no statistical inferences will be performed for the final analysis of this sub-protocol (refer to Section 16).

### 7.5. MULTICENTER STUDIES

Details are provided in the Master COV-01 SAP.

# 7.6. ADJUSTMENTS FOR COVARIATES AND FACTORS TO BE INCLUDED IN ANALYSES

Not applicable since no statistical inferences will be performed for the final analysis of this sub-protocol (refer to Section 16).

### 7.7. EXAMINATION OF SUBGROUPS

No subgroup analyses will be performed for the final analysis of this sub-protocol.

### 7.8. SOFTWARE VERSION

Details are provided in Master COV-01 SAP.

### 8. OUTPUT PRESENTATIONS

Output presentations are described in the Master COV-01 SAP.



### 9. DISPOSITION AND WITHDRAWALS

Analysis of disposition and withdrawals will be presented as described in the Master COV-01 SAP.

### 10. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Demographic characteristics and other baseline characteristics data will be presented as described in the Master COV-01 SAP.

### 11. DISEASE HISTORY

Analysis of disease history will be performed as described in the Master COV-01 SAP.

### 12. MEDICAL HISTORY

Analysis of medical history will be performed as described in the Master COV-01 SAP.

### 13. PRIOR AND CONCOMITANT MEDICATIONS

Analysis of prior and concomitant medications will be performed as described in the Master COV-01 SAP.

### 14. EXPOSURE TO STUDY DRUG

### Patients randomized to sub-protocol COV-01-001

Patients randomized to the Lanadelumab-IV + SoC or Placebo + SoC treatment groups of COV-01-001 sub-protocol will receive an IV injection of either Lanadelumab-IV 300 mg diluted in normal saline or placebo (normal saline), as applicable, in a double-blind manner, one dose on Day 1 and a second dose on Day 4, along with SoC.

Reason for dose modification of study drug (i.e., dose increased, dose reduced, drug interrupted and drug withdrawal) will be captured on the *Exposure* page of the eCRF.



# <u>Patients included in the control arm of COV-01-001 sub-protocol who were randomized to the Placebo + SoC</u> group of a sub-protocol other than COV-01-001

It is to be noted that the planned duration of exposure to a study drug, planned frequency of administration of the study drug, and planned route of administration of the study drug will vary from one sub-protocol to the other, but similar information as for COV-01-001 sub-protocol will be captured on the *Exposure* page of the eCRF of these other sub-protocol.

### Exposure to study drug

The exposure to study drug will be summarized by treatment arm (breaking down the Placebo + SoC arm by sub-protocol) based on the safety analysis set as follows:

- Duration of exposure:
  - o Duration of exposure (days) as a continuous variable
  - Ouration of exposure (days) as a categorical variable: 1 to 3, > 3 to 7, > 7 to 14, > 14 to 29, and > 29
  - Total number of doses received as a continuous variable, where the total number of dosed received is defined as the total number of doses received by each patient, not the total number of doses received across all patients
  - For patients randomized to COV-01-001 sub-protocol only, number and percentages of patients who
    received only one dose and number and percentages of patients who received two doses.
- Dose modifications:
  - o For patients randomized to COV-01-001 sub-protocol only, number and percentage of patients with at least one dose partially administered overall and for each dose
  - Number and percentage of patients with at least one interrupted dose
  - Number and percentage of patients with at least one dose interruption by reason for dose interruption:
    - Adverse events
    - Other.
  - o Total number of dose interruptions as a continuous variable, where the total number of dose

Version Number: Amendment 3, v1.0
Version Date: 23-Jul-2021

interruptions is defined similarly to the total number of doses received

 Among patients with a dose interruption, number and percentage of patients with dose subsequently restarted at planned dose level.

All dosing and exposure data will also be listed. A listing including patients with at least one dose modification only will also be provided.

### 14.1. DERIVATIONS

For patients randomized to a study drug planned to be administered on a daily basis, duration of exposure to study drug, in days, will be computed as follows:

• Duration of exposure (days) = (Date of last dose of study drug – Date of first dose of study drug) + 1

For all other patients (i.e. randomized to a study drug planned to be administered not on a daily basis), duration of exposure to study drug, in days, will be computed as follows:

Duration of exposure (days) = {[Earliest date of (end of planned study treatment period, hospital discharge or discontinuation from study drug)] – Date of first dose of study drug} + 1

### 15. COMPLIANCE WITH STUDY DRUG

Compliance with study drug will be summarized by treatment arm (breaking down the Placebo + SoC arm by sub-protocol) based on the safety analysis set. In addition to the descriptive summary, number and percentage of patients in each of the following compliance categories will be presented:

- < 50%
- $\geq 50 \text{ to} < 80\%$
- $\geq 80\%$  to  $\leq 100\%$
- > 100%.

Compliance data will also be listed.



### 15.1. DERIVATIONS

For each patient, the compliance will be computed as follows:

Compliance (%) = (Actual total number of doses / Expected total number of doses) x 100

#### where:

- Actual total number of doses is defined as the sum of all doses taken through the course of the study
- Expected total number of doses is defined as the sum of protocol-defined doses to be taken through the course
  of the study and is computed as follows:
  - o For patients randomized to a study drug administered on a daily basis:
    - Expected total number of doses = expected number of doses per day \* expected number of days under treatment, where the expected number of days under treatment is defined as: {[Earliest date of (end of planned study treatment period, hospital discharged or discontinuation from study drug)] Date of first dose of study drug} + 1.
  - o For patients randomized to a study drug planned to be administered not on a daily basis:
    - Expected total number of doses = Expected number of doses (injections) per day \* expected number of administration days between randomization and the earliest of (end of planned study treatment period, hospital discharged or discontinuation from study drug).
      - For example, if a study drug is planned to be administered once on Day 1 and once on Day 4, the expected total number of doses is 2; unless patient discontinued from study drug or was discharged from the hospital on or after Day 1 but before Day 4, in which case the expected total number of doses is 1. As another example, if the study drug is planned to be administered twice daily on every other day from Day 1 to Day 14, the expected total number of doses is 14; unless patient discontinued from study drug or was discharged from the hospital let say, on Day 10, in which case the expected total number of doses is 10 (i.e., 2 doses [injection] per days \* 5 administration days).



### 16. EFFICACY ENDPOINTS

Given that only 29 patients were randomized into COV-01-001 sub-protocol and that is expected ~34 patients will be included in final analysis of this sub-protocol when taking the shared placebo arm into account instead of ~700 as required by the sample size (refer to Master SAP Section 7.1), no statistical inferences will be performed for any efficacy endpoint, but two-sided 95% exact binomial Confidence Interval (CI) within each treatment arm will be provided, when possible.

In conformance with the FDA's Guidance for Submission of Abbreviated Report and Synopsis in Support of Marking and publication requirements of *ClinicalTrials.gov*, summary tables will be presented for the primary and key secondary efficacy endpoints (refer to Master SAP Sections 16.1.1, 16.2.1.1, 16.2.1.2, and 16.2.1.3). Although not required by the previously mentioned FDA's Guidance, summary tables will also be provided for the other secondary efficacy endpoints (refer to Master SAP Sections 16.2.1.4 to 16.2.1.9) in order to be compliant with the publication requirements of *ClinicalTrials.gov*.

Efficacy summaries will be performed as described in the Master COV-01 SAP, except that all endpoints will be analyzed on the primary analysis set (refer to Section 5.1) instead of the FAS.

### 16.1. PRIMARY EFFICACY

# 16.1.1. TIME TO CONFIRMED CLINICAL RECOVERY THROUGH DAY 29, WITHOUT RE-HOSPITALIZATION THROUGH DAY 29

Details are provided in the Master COV-01 SAP.

### 16.1.2. MISSING DATA IMPUTATION METHOD FOR PRIMARY EFFICACY ENDPOINT

Details are provided in the Master COV-01 SAP.

### 16.1.3. MAIN ANALYSIS OF PRIMARY EFFICACY ENDPOINT

For the time to confirmed clinical recovery through Day 29, without re-hospitalization through Day 29, as defined in the Master SAP Section 16.1.1, the number and percentage of patients with and without the event will be presented by randomized treatment arm. Two-sided 95% exact binomial CI for the percentage of patients with the event within



each treatment group will be provided. For patients who did not meet the event, the main reason for censoring will be summarized similarly.

Kaplan-Meier curves (product-limit estimate) will be provided by treatment arm for the time to confirmed clinical recovery though Day 29, without re-hospitalization through Day 29. Kaplan-Meier estimate of the time to confirmed clinical recovery through Day 29, without re-hospitalization through Day 29, in days, will be provided at the 25<sup>th</sup>, 50<sup>th</sup> (median), and 75<sup>th</sup> percentiles time along with their corresponding two-sided 95% CIs. The estimates of the SEs will be computed using the Greenwood's formula, the CI for the median will be calculated according to Brookmeyer and Crowley (1982), and the CIs for the survival function estimates at above mentioned time points will be derived from the Kaplan-Meier estimates using the log-log transformation. Kaplan-Meier estimates of the probability of having the event will also be provided at Day 29 along with the number of patients with the event and the number of patients at risk at that time.

#### 16.1.4. SENSITIVITY ANALYSES FOR PRIMARY EFFICACY ENDPOINT

No sensitivity analyses will be performed for this sub-protocol.

### 16.1.5. SUPPLEMENTARY ANALYSES FOR PRIMARY EFFICACY ENDPOINT

No supplementary analyses will be performed for this sub-protocol.

### 16.2. SECONDARY EFFICACY

### 16.2.1. SECONDARY EFFICACY ENDPOINTS

### 16.2.1.1. Incidence of Patients with Oxygen-Free Recovery at Day 29

Details are provided in the Master COV-01 SAP.

# 16.2.1.2. Incidence of Patients with ≥ 2-point Improvement from Baseline or Fit for Discharge on the Ordinal Scale at Day 29

Details are provided in the Master COV-01 SAP.



### 16.2.1.3. Incidence of All-Cause Mortality through Day 29

Details are provided in the Master COV-01 SAP.

## 16.2.1.4. Distribution of Patients across the Categories of the 8-point Ordinal Scale for Clinical Severity at Days 8, 15, and 29

Details are provided in the Master COV-01 SAP.

### 16.2.1.5. Worst Post-Baseline Score on 8-point Ordinal Scale from Baseline to Day 29

Details are provided in the Master COV-01 SAP.

### 16.2.1.6. Number of ICU Days from Day 1 through Day 29

Details are provided in the Master COV-01 SAP.

### 16.2.1.7. Number of Invasive Mechanical Ventilator Days from Day 1 through Day 29

Details are provided in the Master COV-01 SAP.

### 16.2.1.8. Incidence of Patients with Clinical Recovery by Days 8, 15, and 29

Details are provided in the Master COV-01 SAP.

# 16.2.1.9. Incidence of Patients with Sustained Clinical Recovery as Confirmed by Day 60 Follow-up

Details are provided in the Master COV-01 SAP.

### 16.2.2. MISSING DATA IMPUTATION METHOD FOR SECONDARY EFFICACY ENDPOINTS

### 16.2.2.1. Binary Endpoints

Details are provided in the Master COV-01 SAP.


### 16.2.2.2. Ordinal Endpoints

Details are provided in the Master COV-01 SAP.

### 16.2.3. MAIN ANALYSIS OF SECONDARY EFFICACY ENDPOINTS

### 16.2.3.1. Binary Endpoints

For the incidence of patients with oxygen-free recovery at Day 29 (refer to Section 16.2.1.1), incidence of patients with  $\geq$  2-point improvement from baseline or fit for discharge on the ordinal scale at Day 29 (refer to Section 16.2.1.2), incidence of all-cause mortality through Day 29 (refer to Section 16.2.1.3), incidence of patients with clinical recovery at Days 8, 15 and 29 (refer to Section 16.2.1.8), and incidence of patients with sustained clinical recovery as confirmed by Day 60 follow-up (refer to Section 16.2.1.9), the number and percentage of patients with and without the event will be provided by treatment arm. Two-sided 95% exact binomial CI for the percentage of patients with the event within each treatment group will be provided.

For the incidence of all-cause mortality, primary reason of death will also be summarized by treatment arm.

### 16.2.3.2. Ordinal Endpoints

For the incidence of patients in each category of the 8-point ordinal scale for clinical severity at Days 8, 15, and 29 endpoints (refer to Section 16.2.1.4), the number and percentage of patients in each ordinal scale category will be provided at each specified Day for each treatment arm. The worst post-baseline score on the 8-point ordinal scale for clinical severity from randomization to Day 29 (refer to Section 16.2.1.5) and each "number of days" endpoint (refer to Sections 16.2.1.6 and 16.2.1.7) will be summarized similarly.

Shift tables from baseline to each post-baseline day up to Day 29 as well as to the worst post-baseline score will also be provided for the 8-point ordinal scale for clinical severity.

#### 16.2.4. Sensitivity Analyses for Secondary Efficacy Endpoints

No sensitivity analyses will be performed for this sub-protocol.



### 16.2.5. SUPPLEMENTARY ANALYSES FOR SECONDARY EFFICACY ENDPOINTS

The only supplementary analyses that will be performed for this sub-protocol is that Kaplan-Meier product-limit estimates of the time to all-cause mortality through Day 29 as described in the Master SAP Section 16.2.5, but the hazard ratio of the Lanadelumab-IV + SoC vs. shared placebo + SoC, its associated two-sided 95% CI, and p-value based on the Cox proportional hazard model described in the Master SAP will not be provided.

### 16.3. EXPLORATORY EFFICACY

CC

### 16.4. ADDITIONAL EFFICACY

CCI

### 16.5. INTERIM ANALYSIS

No IAs will be performed for this sub-protocol since enrollment into this sub-protocol was early terminated by the Sponsor before the trigger for the first IA was reached (refer to Master SAP Section 16.5).

### 17. SAFETY ENDPOINTS

The safety analyses will be performed as described in the Master COV-01 SAP based on the safety analysis set.

In addition, the following analyses will also be performed for the sub-protocol COV-01-001 based on the safety analysis set.



### 17.1. ADVERSE EVENTS

#### 17.1.1. ADVERSE EVENTS OF SPECIAL INTEREST

The following are defined as adverse events of special interest (AESIs) for Lanadelumab-IV and will be identified based on investigator-reported AESIs on the AE page of the CRF:

- Hypersensitivity reactions (refer to Appendix 1);
- Events of disordered coagulation (i.e., bleeding AESIs or hypercoagulable AESIs; refer to Appendix 2)

A summary of AESIs, overall and by AESI category and PT will be prepared by treatment arm for patients randomized to COV-01-001 only. Should a patient experience multiple events within an AESI category or PT, the patient will be counted only once for that AESI category or PT. Additionally, the risk difference of the overall incidence rates of having any treatment-emergent AESI between the treatment arms will be presented along with its 95% two-sided Wald CI.

A listing of all AESIs will be provided.

### 17.2. LABORATORY EVALUATIONS

In addition to the laboratory tests listed in Appendix 5 of the Master COV-01 SAP, the fibrin degradation products (FDPs) will be included in the outputs.

The analysis for laboratory parameters is described in the Master COV-01 SAP.

### 17.3. VITAL SIGNS

Analysis of vital signs data will be performed as described in the Master COV-01 SAP.

### 17.4. ECG EVALUATION

Electrocardiogram (ECG) evaluation will be performed at screening and on the day of discharge from the hospital. The following ECG parameters will be collected:



- Heart rate (beats per minutes [bpm]);
- PR interval (milliseconds [msec]);
- RR interval (msec);
- QRS interval (msec);
- QT interval (msec);
- QTc interval (msec);
- QTcB interval (msec);
- QTcF inerval (msec);
- Overall ECG interpretation as assessed by Investigator (normal; abnormal, not clinically significant; and abnormal, clinically significant).

The observed and change from baseline values of each continuous ECG parameter will be summarized using descriptive statistics by treatment arm and visit based on the safety analysis set.

Number and percentage of patients in each category of the overall ECG interpretation as assessed by the Investigator will also be provided by treatment arm and visit based on the safety analysis set.

### 17.5. PHYSICAL EXAMINATION

Analysis of physical examination data will be performed as described in the Master COV-01 SAP.

### 18. PHARMACOKINETICS

PK concentrations of Lanadelumab-IV will be summarized by visit and timepoint (refer to Section 3.2) based on the PK analysis set (refer to Section 5.2) overall and broken down further by the ordinal scale for clinical severity score at baseline (2 or 3 to 5). Concentrations that are below the limit of quantification (BLQ) will be treated as a numeric value of zero and will be excluded from the geometric statistics. All PK concentrations will be reported and analyzed with 3 significant figures. For the reporting of descriptive statistics, the mean, standard deviation, standard error (if reported), and confidence interval (if reported) will be presented to one digit more precision than the source



data. The minimum, median, and maximum will be presented to the same precision as the source data. Coefficient of variation will always be reported to 2 decimal places.

For Day 1, PK concentrations of Lanadelumab-IV will be summarized for the pre- and post-infusion separately.

Post-dose timepoints will be presented for Days 4, 7, 15, 29, and day of discharge as PK blood samples can be collected at any time during each of these days.

PK concentrations will be listed according to nominal time points scheduled.

### 19. PHARMACODYNAMICS

CCI

### 20. PLASMA ANTI-DRUG ANTIBODY TESTING

Absence (negative) or presence (positive) of ADA will be summarized and listed by treatment arm across all visits (refer to Section 3.2) based on the ADA analysis set. Positive ADA will be broken down further by neutralizing and non-neutralizing ADA.

### 21. DATA NOT SUMMARIZED OR PRESENTED

The list of data not summarized or presented is available in the Master COV-01 SAP.


### **APPENDIX 1 HYPERSENSITIVITY REACTIONS**

### **Preferred Term**

- Administration site hypersensitivity
- Documented hypersensitivity to administered product
- Drug hypersensitivity
- Hypersensitivity
- Infusion related hypersensitivity reaction
- Infusion site hypersensitivity
- Injection site hypersensitivity
- Type I hypersensitivity
- Type II hypersensitivity
- Type IV hypersensitivity

CCI

PPD

Version Number:

Amendment 3, v1.0


### **APPENDIX 2 EVENTS OF DISORDERED COAGULATION**

### Preferred Term

- Abnormal clotting factor
- Acquired antithrombin III deficiency
- Acquired dysfibrinogenaemia
- Acquired factor IX deficiency
- Acquired factor VIII deficiency
- Acquired factor XI deficiency
- Acquired haemophilia
- Acquired protein S deficiency
- Acquired Von Willebrand's disease
- Activated protein C resistance
- Acute haemorrhagic oedema of infancy
- Anaphylactoid syndrome of pregnancy
- Antiphospholipid syndrome
- Antithrombin III deficiency
- Chronic pigmented purpura
- Coagulation disorder neonatal
- Coagulation factor deficiency
- Coagulation factor mutation
- Coagulopathy




- Congenital coagulopathy
- Congenital dysfibrinogenaemia
- Congenital hypercoagulation
- Dilutional coagulopathy
- Disseminated intravascular coagulation
- Disseminated intravascular coagulation in newborn
- Ecchymosis
- Endothelial protein C receptor polymorphism
- Factor I deficiency
- Factor II deficiency
- Factor II inhibition
- Factor II mutation
- Factor III deficiency
- Factor IX deficiency
- Factor IX inhibition
- Factor V deficiency
- Factor V inhibition
- Factor V Leiden mutation
- Factor VII deficiency
- Factor VII inhibition



- Factor VIII deficiency
- Factor VIII inhibition
- Factor X deficiency
- Factor X inhibition
- Factor XI deficiency
- Factor XII deficiency
- Factor XIII deficiency
- Factor XIII Inhibition
- Haemophilia
- Haemophilia A with anti factor VIII
- Haemophilia A without inhibitors
- Haemophilia B with anti factor IX
- Haemophilia B without inhibitors
- Haemophilic pseudotumour
- Haemorrhage
- Haemorrhagic diathesis
- Haemorrhagic disease of newborn
- Haemorrhagic disorder
- Haemorrhagic vasculitis
- Henoch-Schonlein purpura

| CCI | | |
|-----|----------------------------------|----------------------------------|
| PPD | Version Number:<br>Version Date: | Amendment 3, v1.0<br>23-Jul-2021 |
| CCI | | |

- Henoch-Schonlein purpura nephritis
- Heparin resistance
- Heparin-induced thrombocytopenia
- Hermansky-Pudlak syndrome
- Hypercoagulation
- Hyperfibrinogenaemia
- Hyperfibrinolysis
- Hyperhomocysteinaemia
- Hyperprothrombinaemia
- Hypersensitivity vasculitis
- Hyperthrombinaemia
- Hypocoagulable state
- Hypofibrinogenaemia
- Hypoprothrombinaemia
- Hypothrombinaemia
- Hypothromboplastinaemia
- Increased tendency to bruise
- Infantile scurvy
- Methylenetetrahydrofolate reductase deficiency
- Methylenetetrahydrofolate reductase polymorphism


- Mouth haemorrhage
- Oral purpura
- Petechiae
- Plasminogen activator inhibitor polymorphism
- Protein C deficiency
- Protein S deficiency
- Pulmonary embolism
- Purpura
- Purpura fulminans
- Purpura neonatal
- Purpura non-thrombocytopenic
- Purpura senile
- Secondary thrombocytosis
- Septic coagulopathy
- Spontaneous haematoma
- Spontaneous haemorrhage
- Thrombocytosis
- Thrombotic microangiopathy
- Vascular purpura
- Vitamin C deficiency

| CCI | | |
|-----|----------------------------------|----------------------------------|
| PPD | Version Number:<br>Version Date: | Amendment 3, v1.0<br>23-Jul-2021 |
| CCI | | |

COV-01-001 Statistical Analysis Plan

Page 33 of 33

### **Preferred Term**

- Von Willebrand's disease
- Von Willebrand's factor inhibition


# DocuSign<sup>a</sup>

| Certificate Of Completion | | |
|-------------------------------------------|-------------|--------------------|
| PPD | | Status: Completed |
| PPD | | |
| Record Tracking | | |
| Status: Original<br>7/26/2021 10:50:49 AM | Holder: PPD | Location: DocuSign |
| Signer Events | Signature | Timestamp |

| Signer Events | Signature | Timestamp |
|-------------------------|-----------|-----------|
| PPD | | |
| In Person Signer Events | Signature | Timestamp |

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Favolana Cummanu Fuanta | | |
| Envelope Summary Events | Status | Timestamps |
| Envelope Summary Events Envelope Sent | Status Hashed/Encrypted | <b>Timestamps</b><br>7/26/2021 10:52:45 AM |
| • | | • |
| Envelope Sent | Hashed/Encrypted | 7/26/2021 10:52:45 AM |
| Envelope Sent<br>Certified Delivered | Hashed/Encrypted<br>Security Checked | 7/26/2021 10:52:45 AM<br>7/26/2021 10:58:59 AM |
| Envelope Sent Certified Delivered Signing Complete | Hashed/Encrypted Security Checked Security Checked | 7/26/2021 10:52:45 AM<br>7/26/2021 10:58:59 AM<br>7/26/2021 11:00:43 AM |

### CONSENT TO ELECTRONIC DELIVERY AND EXECUTION OF DOCUMENTS

From time to time, [C] ("we" or "us") may provide you certain written contracts, notices, disclosures, authorizations, acknowledgements or other documents (collectively, the "Documents") electronically. Please read this consent form carefully. It explains the terms and conditions under which such Documents are provided by us and executed by you electronically through your DocuSign, Inc. ("DocuSign") user account. If you consent to the delivery and execution of such Documents electronically, please click the "I Agree" button.

### **Documents** will be sent to you electronically

If you consent to electronic delivery, Documents will be sent to your DocuSign user account. You may request a paper copy of documents previously made available through your DocuSign user account, but an additional charge may be incurred. Alternatively, you can download and print documents sent to your DocuSign user account. Unless otherwise noted, you can access a Document up to 30 days from the date we first sent the Document to you.

### Withhold Consent or Withdrawing Consent to Electronic Delivery

If you withhold consent to electronic delivery or execution, or withdraw your consent at a later date, all Documents will be sent to your mailing address following our receipt of notice of such action. The following sections explain the consequences of withholding or withdrawing your consent to electronic delivery and execution of Documents, and also the procedures you must follow in order to effectuate delivery to your mailing address.

### **Consequences of Withdrawing Consent**

By electing to only receive and execute Documents sent to your mailing address, we will not be able to carry out transactions or services as efficiently. For instance, some transactions or services require your express consent. We can perform these transaction or services only if we first receive an acknowledgement that indicates you received and consent to the Document related to the proposed transaction or service.

To withhold consent now or withdraw consent at a later date, please sign DocuSign's "Withdraw Consent" form on the signing page of your DocuSign user account. This will indicate that you have withdrawn your consent to receive Documents electronically. Once you sign the "Withdraw Consent" form, you will no longer be able to use your DocuSign user account to execute Documents electronically and we will send Documents to your mailing address. Withdrawal of consent does not affect the validity of any Documents previously executed electronically prior to such withdrawal of Consent. In addition, should you execute any Documents electronically, your execution of such Documents shall indicate your continued consent to execute such Documents electronically.

### How to contact **CC**:

If you would like us to send the Documents to a different e-mail address, request paper copies of Documents you have previously received electronically, or withdraw your consent to receive electronic documents, please follow the instructions below. If you have any other questions, please contact: CCI

## 1. To advise ccl of your new e-mail address

If you would like your Documents sent to a different e-mail address, you must send an e-mail message to column and the body of the e-mail please state the following: (i) your previous e-mail address, and (ii) your new e-mail address. No other information is required.

In addition, you must notify DocuSign of your new e-mail address. Please log into your DocuSign user account, and follow the instructions to update your e-mail address.

# 2. To request paper copies from CCI

To request paper copies of Documents you have received previously through your DocuSign user account, send an e-mail to CCI

In the body of the e-mail please state the following: (i) your e-mail address, (ii) full name, (iii) U.S. Postal address, and (iv) telephone number. Additional charges may apply for such paper copies.

### 3. To withdraw your consent with CC

To withdraw your consent to receiving and executing Documents in an electronic format, you may do one of the following:

i. decline to sign a document from within your DocuSign user account, and on the subsequent page, select the check-box indicating you wish to withdraw your consent; or ii. send us an e-mail to CCI and and in the body of such request you must state your e-mail, full name, US Postal Address, telephone number, and account number. No additional information is necessary.

### Required hardware and software

| Operating Systems: | Windows® 2000, Windows® XP, Windows Vista®; Mac OS® X |
|---|---|
| Browsers: | <ul> <li>Internet Explorer (Windows Only) 8.0 or above – compatibility mode is supported only for 9.0 and above.</li> <li>Windows Edge Current Version</li> <li>Mozilla Firefox Current Version</li> <li>Safari (Mac OS only) 6.2 or above</li> <li>Google Chrome Current Version</li> </ul> |
| PDF Reader: | Acrobat® or similar software may be required to view and print PDF files |
| Screen Resolution: | 1024 x 768 Recommended |
| Enabled Security Settings: | Allow per session cookies |
| Mobile Signing: | <ul><li>Apple iOS 7.0 or above</li><li>Android 4.0 or above</li></ul> |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, we will provide you with an e-mail message at the e-mail address we have on file for you at the time the hardware and software requirements are revised.

Pre-release (e.g. beta) versions of operating systems and browsers are not supported.

### Acknowledging your access and consent to receive materials electronically

To confirm you can access this information electronically and that you consent to receiving and executing Documents electronically on the terms and conditions described above, please let us know by clicking the "I Agree" button.

By clicking the "I Agree" button, you confirm that

- You can access and read this Consent To Electronic Delivery and Execution of Documents; and
- You can print on paper the disclosure or save or send the disclosure to a place where you can print it, for future reference and access; and
- Until or unless you notify occur as described above, you consent to the delivery and execution of Documents electronically.

# COV-01-004 STATISTICAL ANALYSIS PLAN

INDUSTRY ALLIANCE PLATFORM TRIAL TO ASSESS THE EFFICACY AND SAFETY OF MULTIPLE CANDIDATE AGENTS FOR THE TREATMENT OF COVID-19 IN HOSPITALIZED PATIENTS

**SUB-PROTOCOL NUMBER: COV-01-004** 

SUB-PROTOCOL FOR CANDIDATE AGENT: APREMILAST

**AUTHOR: PPD** 

VERSION NUMBER AND DATE: AMENDMENT 1 v1.0, 23Apr2021



# SUB-PROTOCOL STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

Sub-protocol Statistical Analysis Plan (SAP) Amendment 1 v1.0 (dated 23Apr2021) for sub-protocol COV-01-004.

| | Name | Signature | Date (DDMmmYYYY) |
|-----------|------|-----------|------------------|
| Author: | PPD | PPD | |
| Position: | PPD | | |
| Company: | CCI | | |

Upon review of this document, the undersigned approves this version of the sub-protocol COV-01-004 SAP, authorizing that the content is acceptable for the reporting specific to this sub-protocol.

| | Name | Signature | Date (DDMmmYYYY) |
|---------------|-------------|-----------|------------------|
| Approved by: | PPD | PPD | |
| Position: | PPD | | |
| Company: | CCI | | |
| On behalf of: | PPD | | |
| Position: | PPD | | |
| Company: | CCI | | |
| Approved by: | PPD | PPD | |
| Position: | PPD | | |
| Company: | Amgen, Inc. | | |



# **MODIFICATION HISTORY**

| Unique<br>Identifier for<br>this Version | Date of the<br>Document<br>Version | Author | Significant Changes from Previous Version |
|---|---|---|---|
| Final, v1.0 | 24Nov2020 | PPD | Not Applicable – First Version |
| Amendment 1, v1.0 | 23Apr2021 | PPD | Updated COV-01-004 sub-protocol version on which this subprotocol SAP is based from version 3.1, dated 26Oct2020, to version 4.0. dated 14Apr2021 Removed Section 11 (COVID-19 Co-Morbidities) since this section is now combined with Section 12 (Medical History) in Master SAP Updated title of former Sections 12 (now Section 11) and 14 (now 13) to be in line with Master SAP. Added pharmacodynamic (PD) analysis set |



# TABLE OF CONTENTS

| 1. | INTRODUCTION | ······ |
|---|---|---|
| 2. | STUDY OBJECTIVES | |
| 3. | STUDY DESIGN | |
| 3.1. | General Description | |
| 3.2. | 2. Schedule of Activities | |
| 3.3. | 3. Changes to Planned Analyses from Master Protocol COV-01 and Sub-Proto | col COV-01-0047 |
| 4. | PLANNED ANALYSES | 8 |
| 5. | ANALYSIS SETS | 8 |
| 5.1. | Pharmacokinetic Analysis Set | 8 |
| 5.2. | 2. Pharmacodynamic Analysis Set | 8 |
| 5.3. | 3. Process for Analysis Set Assignment | 8 |
| 6. | GENERAL CONSIDERATIONS | 9 |
| 7. | STATISTICAL CONSIDERATIONS | 9 |
| 7.1. | Sample Size Calculation | 9 |
| 7.2. | 2. Missing Data | 9 |
| 7.3. | 3. Statistical Tests | 9 |
| 7.4. | 4. Multiple Comparisons/Multiplicity | |
| 7.5. | 5. Multicenter Study | 9 |
| CCI | | |
| PPD | Version Number: Version Date: | Amendment 1, v1.0<br>23Apr2021 |

| 7.6. | Adjustments for Covariates and Factors to be Included in Analyses | 9 |
|---|---|---|
| 7.7. | Examination of Subgroups | 10 |
| 7.8. | Software Version | 10 |
| 8. | OUTPUT PRESENTATIONS | 10 |
| 9. | DISPOSITION AND WITHDRAWALS | 10 |
| 10. | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 10 |
| 11. | DISEASE HISTORY | 11 |
| 12. | MEDICAL HISTORY | 11 |
| 13. | PRIOR AND CONCOMITANT MEDICATIONS | 11 |
| 14. | EXPOSURE TO STUDY DRUG | 11 |
| 14.1. | Derivations | 13 |
| 15. | COMPLIANCE WITH STUDY DRUG | 14 |
| 15.1. | Derivations | 14 |
| 16. | EFFICACY ENDPOINTS | 15 |
| 17. | SAFETY ENDPOINTS | 15 |
| 17.1. | Adverse Events | 15 |
| 17.2. | Laboratory Evaluations | 10 |
| 17.3. | Vital Signs | 16 |
| CCI | | |
| PPD | Version Number: Amendr<br>Version Date: | nent 1, v1.0<br>23Apr2021 |

| COV-01-004 | Statistical | Analy | sis F | Plan |
|------------|-------------|-------|-------|------|

Page 6 of 18

| 17.4. | ECG Evaluations | 16 |
|-------|----------------------------------|----|
| 17.5. | Physical Examination | 16 |
| 18. | PHARMACOKINETICS | 16 |
| 18.1. | Derivations | 17 |
| 19. | PHARMACODYNAMICS | 18 |
| 20 | DATA NOT SUMMARIZED OR PRESENTED | 18 |

### 1. Introduction

This statistical analysis plan (SAP) describes the rules and conventions to be used in the presentation and analysis of data specific to sub-protocol COV-01-004 of master protocol COV-01. It describes the specific data to be summarized and analyzed, including specifics of the statistical analyses to be performed.

This sub-protocol SAP is based on version 4.0 of the sub-protocol COV-01-004, dated 14Apr2021.

For the rules and conventions to be used in the presentation and analysis of data common across all sub-protocols, refer to the Master COV-01 SAP.

### 2. STUDY OBJECTIVES

The study objectives are described in the Master COV-01 SAP.

### 3. STUDY DESIGN

### 3.1. GENERAL DESCRIPTION

The general description is available in the Master COV-01 SAP.

### 3.2. SCHEDULE OF ACTIVITIES

The schedule of activities can be found in Section 1.2 of the sub-protocol COV-01-004.

# 3.3. CHANGES TO PLANNED ANALYSES FROM MASTER PROTOCOL COV-01 AND SUB-PROTOCOL COV-01-004

There are no changes to the analyses planned for master protocol COV-01 and sub-protocol COV-01-004.



### 4. PLANNED ANALYSES

The planned analyses are listed and described in the Master COV-01 SAP.

All outputs described in this sub-protocol SAP will be produced at the time of sub-protocol COV-01-004 primary analysis (refer to COV-01 Master SAP).

In addition to the outputs planned to be produced at the time of COV-01-004 sub-protocol final analysis (refer to COV-01 Master SAP), safety outputs described in this sub-protocol SAP will also be produced at the time of COV-01-004 sub-protocol final analysis (refer to Section 17.1).

### 5. ANALYSIS SETS

Analysis sets are described in the Master COV-01 SAP.

An additional analysis set that is specific to sub-protocol COV-01-004 is described below:

### 5.1. PHARMACOKINETIC ANALYSIS SET

The pharmacokinetic (PK) analysis set will include all patients included in the safety analysis set (refer to Master COV-01 SAP Section 5.2) who were randomized to the apremilast plus Standard of Care (SoC) treatment group and have at least one measured PK concentration.

### 5.2. PHARMACODYNAMIC ANALYSIS SET

The pharmacodynamic (PD) analysis set will include all patients included in the safety analysis set (refer to Master COV-01 SAP Section 5.2) who were randomized to the COV-01-004 sub-protocol (i.e., apremilast plus SoC or placebo to apremilast + SoC treatment groups) and have at least one measured post-baseline biomarker level.

### 5.3. PROCESS FOR ANALYSIS SET ASSIGNMENT

As the PK analysis set is defined based on objective criteria only, the authorization of this sub-protocol SAP will stand for the agreement and authorization of the inclusion/exclusion of each patient in this PK analysis set.



### 6. GENERAL CONSIDERATIONS

Details are provided in the Master COV-01 SAP.

### 7. STATISTICAL CONSIDERATIONS

### 7.1. SAMPLE SIZE CALCULATION

Details are defined in the Master COV-01 SAP.

### 7.2. MISSING DATA

Details are defined in the Master COV-01 SAP.

### 7.3. STATISTICAL TESTS

Details are defined in the Master COV-01 SAP.

### 7.4. MULTIPLE COMPARISONS/MULTIPLICITY

Details are defined in the Master COV-01 SAP.

### 7.5. MULTICENTER STUDY

Details are defined in the Master COV-01 SAP.

# 7.6. ADJUSTMENTS FOR COVARIATES AND FACTORS TO BE INCLUDED IN ANALYSES

Details are defined in the Master COV-01 SAP.



### 7.7. EXAMINATION OF SUBGROUPS

For sub-protocol COV-01-004, additional subgroup analyses will be performed for selected safety data (refer to Section 17.1). The additional subgroup is:

• Patients randomized to sub-protocol COV-01-004 (apremilast plus SoC and placebo plus SoC treatment groups) plus patients included in COV-01-004 control arm (refer to Master COV-01 SAP Section 4.5) that have been randomized to the placebo plus SoC treatment group of a sub-protocol other than COV-01-004 and who did not receive any concomitant dose of apremilast during the course of the study (refer to Master COV-01 SAP Section 14 for concomitant use definition). That is, placebo plus SoC patients included in the control arm of COV-01-004 who were randomized to a sub-protocol other than COV-01-004 and who concomitantly took apremilast during the course of the study will be excluded from this subgroup.

It is to be noted that these subgroup analyses will be performed only if more than 10% of patients included in COV-01-004 control arm, that have been randomized to a sub-protocol other than COV-01-004, concomitantly took apremilast during the course of the study.

### 7.8. SOFTWARE VERSION

Details are defined in the Master COV-01 SAP.

### 8. OUTPUT PRESENTATIONS

Output presentations are described in the Master COV-01 SAP.

### 9. DISPOSITION AND WITHDRAWALS

Analysis of disposition and withdrawals is described in the Master COV-01 SAP.

### 10. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Analysis of demographic and other baseline characteristics is described in the Master COV-01 SAP.



### 11. DISEASE HISTORY

Analysis of disease history at screening is described in the Master COV-01 SAP.

### 12. MEDICAL HISTORY

Analysis of medical history is described in the Master COV-01 SAP.

### 13. PRIOR AND CONCOMITANT MEDICATIONS

Analysis of prior and concomitant medications is described in the Master COV-01 SAP.

### 14. EXPOSURE TO STUDY DRUG

### Patients randomized to sub-protocol COV-01-004

Patients randomized to the apremilast plus SoC or placebo plus SoC treatment groups of COV-01-004 sub-protocol will receive either an apremilast 30 mg or matching placebo tablet, as applicable, twice daily (BID) in a double-blind manner for 14 days or until hospital discharge, death, or discontinuation of study drug, whichever occurs first, in addition to SoC.

Reason for dose modification of study drug (i.e., dose increased, dose reduced, drug interrupted, drug withdrawal, and unknown) will be captured on the *Exposure* page of the electronic Case Report Form (eCRF).

# Patients included in the control arm of COV-01-004 sub-protocol who were randomized to the placebo plus SoC group of a sub-protocol other than COV-01-004

It is to be noted that the planned duration of exposure to a study drug, planned frequency of administration of the study drug, and planned route of administration of the study drug will vary from one sub-protocol to the other, but similar information as for COV-01-004 sub-protocol will be captured on the *Exposure* page of the eCRF of these other sub-protocols.



### Exposure to study drug

The exposure to study drug will be summarized by treatment arm (breaking down the placebo plus SoC arm by sub-protocol) based on the safety analysis set as follows:

- Duration of exposure:
  - O Duration of exposure (days) as a continuous variable;
  - Duration of exposure (days) as a categorical variable: 1 to 3, > 3 to 7, > 7 to 14, and > 14;
  - Total number of doses received as a continuous variable, where the total number of doses received is
    defined as the total number of doses received by each patient, not the total number of doses received
    across all patients.
- Average dose (mg/day) only for patients randomized to sub-protocol COV-01-004;
- Dose modifications:
  - o Number and percentage of patients with at least one dose reduction;
  - o Number and percentage of patients with a dose reduction by reason for dose reductions:
    - Adverse events;
    - Due to creatinine clearance < 30 mL/min\*;
    - Due to renal replacement therapy\*;
    - Other.
  - Total number of dose reductions as a continuous variable, where the total number of dose reductions defined similarly to the total number of doses received;
  - Among patients with a dose reduction, number and percentage of patients with dose subsequently increased back to the planned dose level;
  - o Number and percentage of patients with at least one interrupted dose;



- Number and percentage of patients with at least one dose interruption by reason for dose interruption:
  - Adverse events:
  - Due to creatinine clearance < 30 mL/min\*;</li>
  - Due to renal replacement therapy\*;
  - Other.
- Total number of dose interruptions as a continuous variable, where the total number of dose interruptions is defined similarly to the total number of doses received;
- Among patients with a dose interruption, number and percentage of patients with dose subsequently restarted at planned dose level;
- o Number and percentage of patients with at least one overdose.
- \* Applicable only for patients randomized to sub-protocol COV-01-004.

All dosing and exposure data will also be listed.

### 14.1. DERIVATIONS

For patients randomized to a study drug planned to be administered on a daily basis, duration of exposure to study drug, in days, will be computed as follows:

• Duration of exposure (days) = (Date of last dose of study drug – Date of first dose of study drug) + 1

For all other patients (i.e. randomized to a study drug planned to be administered not on a daily basis), duration of exposure to study drug, in days, will be computed as follows:

• Duration of exposure (days) = {[Earliest date of (end of planned study treatment period, hospital discharge or discontinuation from study drug)] – Date of first dose of study drug} + 1

For patients randomized to sub-protocol COV-01-004 only, the average dose per day will be computed as follows:

• Average dose (mg/day) = Total cumulative dose (mg) / duration of exposure (days)



where the total cumulative dose is the computed total cumulative dose (mg) taken by a patient during the course of the study.

### 15. COMPLIANCE WITH STUDY DRUG

Compliance with study drug will be summarized by treatment arm (breaking down the placebo plus SoC arm by sub-protocol) based on the safety analysis set. In addition to the descriptive summary, the following compliance categories will be presented:

- < 80%;
- $\geq 80\%$  to < 100%
- 100%;
- > 100%.

Compliance data will also be listed.

### 15.1. DERIVATIONS

For each patient, the compliance will be computed as follows:

• Compliance (%) = (Actual total number of doses / Expected total number of doses) x 100

### where:

- Actual total number of doses is defined as the sum of all doses taken through the course of the study
- Expected total number of doses is defined as the sum of protocol-defined doses to be taken through the course
  of the study and is computed as follows:
  - o For patients randomized to a study drug administered on a daily basis:
    - Expected total number of doses = expected number of doses (injections) per day \* expected number of days under treatment, where the expected number of days under treatment is defined as:
       {[Earliest date of (end of planned study treatment period, hospital discharged or discontinuation



from study drug)] – Date of first dose of study drug} + 1

- o For patients randomized to a study drug planned to be administered not on a daily basis:
  - Expected total number of doses = Expected number of doses (injections) per day \* number of expected administration days between randomization and the earliest of (end of planned study treatment period, hospital discharged or discontinuation from study drug).

For example, if a study drug is planned to be administered once on Day 1 and once on Day 4, the expected total number of doses is 2; unless patient discontinued from study drug or was discharged from the hospital on or after Day 1 but before Day 4, in which case the expected total number of doses is 1. As another example, if the study drug is planned to be administered twice daily on every other day from Day 1 to Day 14, the expected total number of doses is 14; unless patient discontinued from study drug or was discharged from the hospital let say, on Day 10, in which case the expected total number of doses is 10 (i.e., 2 doses [injection] per days \* 5 administration days).

### 16. EFFICACY ENDPOINTS

Efficacy analyses are described in the Master COV-01 SAP.

### 17. SAFETY ENDPOINTS

### 17.1. ADVERSE EVENTS

In addition to the safety analyses described in the Master COV-01 SAP, the following analyses will be repeated for the subgroup of patients defined in Section 7.7 based on the safety analysis set:

- Overview of treatment-emergent adverse events (TEAEs);
- TEAEs by maximum Common Terminology Criteria for Adverse Events (CTCAE) grade, System Organ Class and Preferred Term (PT);



- TEAEs with a CTCAE grade  $\geq$  3 by System Organ Class and PT:
- Fatal TEAEs by System Organ Class and PT;
- Serious TEAEs by System Organ Class and PT;
- Most common serious TEAEs by PT, where a most common is defined as at least 1% in at least one treatment arm:
- TEAEs leading to dose modification by System Organ Class and PT;
- TEAEs leading to discontinuation of study drug by System Organ Class and PT;

Patients excluded from the subgroup defined in Section 7.7 will be flagged in the listings of all fatal AEs, all SAEs, and all AEs leading to permanent discontinuation of study drug.

Refer the Master COV-01 SAP Section 18.1 for additional details about these summaries and listings.

### 17.2. LABORATORY EVALUATIONS

Analysis of laboratory evaluations is described in the Master COV-01 SAP.

### 17.3. VITAL SIGNS

Analysis of vital signs is described in the Master COV-01 SAP.

### 17.4. ECG EVALUATIONS

Analysis of electrocardiogram (ECG) evaluations is described in the Master COV-01 SAP.

### 17.5. PHYSICAL EXAMINATION

Analysis of physical examination is described in the Master COV-01 SAP.



### 18. PHARMACOKINETICS

PK concentrations of apremilast will be summarized and listed by visit and timepoints based on the PK analysis set. In addition to the descriptive statistics mentioned in Master COV-01 SAP Appendix 2, the coefficient of variation (CV%), geometric mean, geometric standard deviation (SD), and geometric CV% will also be provided for the PK concentrations. Concentrations that are below the limit of quantification (BLQ) will be treated as a numeric value of zero.

PK concentrations of apremilast will be summarized for the following time categories:

- 0 < 3 hours post morning administration of study drug;
- 3 <6 hours post morning administration of study drug;
- 6 < 9 hours post morning administration of study drug;
- 9 <12 hours post morning administration of study drug
- 0 < 3 hours post evening administration of study drug;
- 3 <6 hours post evening administration of study drug;
- 6 < 9 hours post evening administration of study drug;
- 9 <12 hours post evening administration of study drug.

Scatter plots of plasma concentrations against the time since last dose, in hours, will be provided for each day and each dose of study drug (i.e., Day 8 post morning administration of study drug, Day 8 post evening administration of study drug, Day 15 post morning administration of study drug, and Day 15 post evening administration of study drug).

## 18.1. DERIVATIONS

For each day where a blood sample for PK concentration is planned to collected, the time of the two administrations of study drug taken on a day will be compared with the time of the blood sample for PK concentration collected on that day as follows in order to derive the timepoint categories specified in Section 18:



- Time post morning administration of study drug (hours) = {[Time (hours & minutes) of collection of the blood sample for PK concentration Time (hours & minutes) of the morning administration of the study drug] + 1} / 60 minute if time of collection of the blood sample for PK concentration is before the time of the evening administration of the study drug;
- Time post evening administration of study drug (hours) = {[Time (hours & minutes) of collection of the blood sample for PK concentration Time (hours & minutes) of the evening the administration of study drug] + 1} / 60 minute if time of collection of the blood sample for PK concentration is on or after the time of the evening administration of the study drug but before the time of the morning administration of study drug of the next day.

### 19. PHARMACODYNAMICS



### 20. DATA NOT SUMMARIZED OR PRESENTED

The list of data not summarized or presented is available in the Master COV-01 SAP.





| Certificate Of Completion | | | |
|---------------------------------------|-------------|--------------------|--|
| PPD | | Status: Completed | |
| PPD | | | |
| Record Tracking | | | |
| Status: Original 4/23/2021 4:17:13 PM | Holder: PPD | Location: DocuSign | |
| Signer Events PPD | Signature | Timestamp | |
| Signer Events | Signature | Timestamp |
|-------------------------|-----------|-----------|
| PPD | | |
| In Person Signer Events | Signature | Timestamp |
| Editor Delivery Events | Status | Timestamp |
| • | | • |

| in Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent Certified Delivered Signing Complete Completed | Hashed/Encrypted Security Checked Security Checked Security Checked | 4/23/2021 4:19:03 PM<br>4/23/2021 4:20:35 PM<br>4/23/2021 4:21:02 PM<br>4/23/2021 6:03:23 PM |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disclosure | | |

#### CONSENT TO ELECTRONIC DELIVERY AND EXECUTION OF DOCUMENTS

From time to time, ("we" or "us") may provide you certain written contracts, notices, disclosures, authorizations, acknowledgements or other documents (collectively, the "Documents") electronically. Please read this consent form carefully. It explains the terms and conditions under which such Documents are provided by us and executed by you electronically through your DocuSign, Inc. ("DocuSign") user account. If you consent to the delivery and execution of such Documents electronically, please click the "I Agree" button.

#### **Documents** will be sent to you electronically

If you consent to electronic delivery, Documents will be sent to your DocuSign user account. You may request a paper copy of documents previously made available through your DocuSign user account, but an additional charge may be incurred. Alternatively, you can download and print documents sent to your DocuSign user account. Unless otherwise noted, you can access a Document up to 30 days from the date we first sent the Document to you.

#### Withhold Consent or Withdrawing Consent to Electronic Delivery

If you withhold consent to electronic delivery or execution, or withdraw your consent at a later date, all Documents will be sent to your mailing address following our receipt of notice of such action. The following sections explain the consequences of withholding or withdrawing your consent to electronic delivery and execution of Documents, and also the procedures you must follow in order to effectuate delivery to your mailing address.

#### **Consequences of Withdrawing Consent**

By electing to only receive and execute Documents sent to your mailing address, we will not be able to carry out transactions or services as efficiently. For instance, some transactions or services require your express consent. We can perform these transaction or services only if we first receive an acknowledgement that indicates you received and consent to the Document related to the proposed transaction or service.

To withhold consent now or withdraw consent at a later date, please sign DocuSign's "Withdraw Consent" form on the signing page of your DocuSign user account. This will indicate that you have withdrawn your consent to receive Documents electronically. Once you sign the "Withdraw Consent" form, you will no longer be able to use your DocuSign user account to execute Documents electronically and we will send Documents to your mailing address. Withdrawal of consent does not affect the validity of any Documents previously executed electronically prior to such withdrawal of Consent. In addition, should you execute any Documents electronically, your execution of such Documents shall indicate your continued consent to execute such Documents electronically.

#### How to contact **CC**:

If you would like us to send the Documents to a different e-mail address, request paper copies of Documents you have previously received electronically, or withdraw your consent to receive electronic documents, please follow the instructions below. If you have any other questions, please contact: CCI

## 1. To advise color of your new e-mail address

If you would like your Documents sent to a different e-mail address, you must send an e-mail message to column and the body of the e-mail please state the following: (i) your previous e-mail address, and (ii) your new e-mail address. No other information is required.

In addition, you must notify DocuSign of your new e-mail address. Please log into your DocuSign user account, and follow the instructions to update your e-mail address.

## 2. To request paper copies from CCI

To request paper copies of Documents you have received previously through your DocuSign user account, send an e-mail to CCI

In the body of the e-mail please state the following: (i) your e-mail address, (ii) full name, (iii) U.S. Postal address, and (iv) telephone number. Additional charges may apply for such paper copies.

### 3. To withdraw your consent with CC

To withdraw your consent to receiving and executing Documents in an electronic format, you may do one of the following:

i. decline to sign a document from within your DocuSign user account, and on the subsequent page, select the check-box indicating you wish to withdraw your consent; or ii. send us an e-mail to CCI and in the body of such request you must state your e-mail, full name, US Postal Address, telephone number, and account number. No additional information is necessary.

#### Required hardware and software

| Operating Systems: | Windows® 2000, Windows® XP, Windows Vista®; Mac OS® X |
|---|---|
| Browsers: | <ul> <li>Internet Explorer (Windows Only) 8.0 or above – compatibility mode is supported only for 9.0 and above.</li> <li>Windows Edge Current Version</li> <li>Mozilla Firefox Current Version</li> <li>Safari (Mac OS only) 6.2 or above</li> <li>Google Chrome Current Version</li> </ul> |
| PDF Reader: | Acrobat® or similar software may be required to view and print PDF files |
| Screen Resolution: | 1024 x 768 Recommended |
| Enabled Security Settings: | Allow per session cookies |
| Mobile Signing: | <ul><li>Apple iOS 7.0 or above</li><li>Android 4.0 or above</li></ul> |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, we will provide you with an e-mail message at the e-mail address we have on file for you at the time the hardware and software requirements are revised.

Pre-release (e.g. beta) versions of operating systems and browsers are not supported.

#### Acknowledging your access and consent to receive materials electronically

To confirm you can access this information electronically and that you consent to receiving and executing Documents electronically on the terms and conditions described above, please let us know by clicking the "I Agree" button.

By clicking the "I Agree" button, you confirm that

- You can access and read this Consent To Electronic Delivery and Execution of Documents; and
- You can print on paper the disclosure or save or send the disclosure to a place where you can print it, for future reference and access; and
- Until or unless you notify occur as described above, you consent to the delivery and execution of Documents electronically.

COV-01-005 Statistical Analysis Plan

UCB Biopharma SRL Sub-Protocol COV-01-005


## COV-01-005 STATISTICAL ANALYSIS PLAN

INDUSTRY ALLIANCE PLATFORM TRIAL TO ASSESS THE EFFICACY AND SAFETY OF MULTIPLE CANDIDATE AGENTS FOR THE TREATMENT OF COVID-19 IN HOSPITALIZED PATIENTS

**SUB-PROTOCOL NUMBER: COV-01-005** 

SUB-PROTOCOL FOR CANDIDATE AGENT: ZILUCOPLAN

AUTHOR: PPD

VERSION NUMBER AND DATE: Amendment 2 v1.0, 28-Jul-2021

# SUB-PROTOCOL COV-01-005 STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

Sub-protocol COV-01-005 Statistical Analysis Plan (SAP) Amendment 2 v1.0 (dated 28-Jul-2021).

| | Name | Signature | Date (DD-Mmm-YYYY) |
|-----------|------|-----------|--------------------|
| Author: | PPD | PPD | |
| Position: | PPD | | |
| Company: | CCI | | |

Upon review of this document, the undersigned approves this version of the sub-protocol COV-01-005 SAP, authorizing that the content is acceptable for the reporting specific to this sub-protocol.

| | Name | Signature | Date (DD-Mmm-YYYY) |
|---------------|-------------------|-----------|--------------------|
| On behalf of: | PPD | PPD | |
| Position: | PPD | | |
| Company: | CCI | | |
| | ' | | |
| Approved By: | PPD | PPD | |
| Position: | PPD | | |
| Company: | UCB Biopharma SRL | | |

## **MODIFICATION HISTORY**

| Unique<br>Identifier for<br>this Version | Date of the<br>Document<br>Version | Author | Significant Changes from Previous Authorized Version |
|---|---|---|---|
| Final, v1.0 | 11-Jan-2021 | PPD | Not Applicable – First Version |
| Amendment 1, v1.0 | 27-Apr-2021 | PPD | Update title of Sections 11 and 13 to be in line with Master SAP; Removed the Ukrainian and Non-Ukrainian subgroups and related supplementary analyses; Removed supplementary analyses adjusted for Ukrainians vs. Non-Ukrainians patients' status; Added subgroup of patients randomized to this subprotocol and related supplementary analyses; Added that the risk difference of the overall incidence rates of having any treatmentemergent AESI between the treatment groups will be presented along with its 95% two-sided |
| | | | Wald CI. |

| Unique<br>Identifier for<br>this Version | Date of the<br>Document<br>Version | Author | Significant Changes from Previous Authorized Version |
|---|---|---|---|
| Amendment 2, v1.0 | 28-Jul-2021 | PPD | Specified that the two Interim Analyses (IAs) and Primary Analysis at Day 29 will not be performed for this sub-protocol since enrollment into this sub-protocol was terminated early by the Sponsor on 07-Jun-2021 before the trigger of each of these analyses was met. Exception of summary statistics for the primary efficacy endpoint, secondary efficacy endpoints (key and other), and the additional efficacy endpoint of all-cause mortality through Day 60, removed all planned efficacy analyses given that 1) enrollment into this sub-protocol was terminated early by the Sponsor on 07-Jun-2021, 2) number of patients to be included in COV-01-005 sub-protocol final analysis, and 3) an abbreviated Clinical Study Report will be created for this sub-protocol. Added two-sided 95% exact binomial Confidence Interval within each treatment arm, when applicable. Removed additional subgroup analyses that were to be performed for sub-protocol primary and key secondary efficacy endpoints. |

| CCI | | |
|-----|------------------------|---------------------------------|
| PPD | Version N<br>Version D | mendment 2, v1.0<br>28-Jul-2021 |
| CCI | | ı |

## **TABLE OF CONTENTS**

| 1. | Intro | duction | 8 |
|---|---|---|---|
| 2. | Study | y Objectives | 8 |
| 3. | Cad. | y Design | |
| э. | • | • | |
| | 3.1. | General Description | |
| | 3.2. | Schedule of Activities | 8 |
| | 3.3. | Changes to Analysis from Master Protocol COV-01 and Sub-Protocol COV-01-005 | 8 |
| 4. | Planr | ned Analyses | 9 |
| | 4.1. | IDMC Safety Analyses | 9 |
| | 4.2. | Interim Analyses | 9 |
| | 4.3. | Primary Analysis | 9 |
| | 4.4. | Final Analysis | 9 |
| | 4.5.<br>4.5.1<br>4.5.2 | | 10 |
| 5. | Analy | ysis Sets | 11 |
| | 5.1. | Pharmacokinetic Analysis Set | 1 |
| | 5.2. | Pharmacodynamic Analysis Set | 11 |
| | 5.3. | Anti-Drug Antibody Analysis Set | 1 |
| | 5.4. | Process for Analysis Set Assignment | 1 |
| 6. | | eral Considerations | |
| 7. | Statis | stical Considerations | |
| | 7.1. | Sample Size Calculation | 12 |
| | 7.2. | Missing Data | 12 |
| | 7.3. | Statistical Tests | 12 |
| | 7.4. | Multiple Comparisons/Multiplicity | 12 |
| | 7.5. | Multicenter Study | 12 |
| | 7.6. | Adjustments for Covariates and Factors to be Included in Analyses | 13 |





Version Number: Version Date: Amendment 2, v1.0 28-Jul-2021



| 7 | .7. | Examination of Subgroups | 13 |
|---|---|---|---|
| 7 | .8. | Software Version | 13 |
| 8. | Outp | out Presentations | 13 |
| 9. | Dispo | osition and Withdrawals | 13 |
| 10. | Dem | nographic and Other Baseline Characteristics | 13 |
| 11. | Disea | ase Historyase | 13 |
| 12. | Med | lical History | 14 |
| 13. | Prior | r and Concomitant Medications | 14 |
| 1 | 3.1. | Derivation | 14 |
| 14. | Ехро | osure to Study Drug | 15 |
| 1 | 4.1. | Derivations | 16 |
| 15. | Com | pliance with Study Drug | 16 |
| 1 | 5.1. | Derivations | 17 |
| 16. | Effica | acy Endpoints | 18 |
| 1 | 6.1. | Primary Efficacy | 19 |
| | 16.1. | <ol> <li>Time to Confirmed Clinical Recovery through Day 29, without Re-Hospitalization Throu</li> <li>19</li> </ol> | gh Day 29 |
| | 16.1. | .2. Missing Data Imputation Method for Primary Efficacy Endpoint | 19 |
| | 16.1. | | |
| | 16.1. | | |
| | 16.1. | .5. Supplementary Analyses for Primary Efficacy Endpoint | 20 |
| 1 | 6.2. | Secondary Efficacy | 20 |
| | 16.2. | .1. Secondary Efficacy Endpoints | 20 |
| | 16.2. | .2. Missing Data Imputation Method for Secondary Efficacy Endpoints | 20 |
| | 16.2. | , , , , | |
| | | 6.2.3.1. Binary Endpoints | |
| | | 6.2.3.2. Ordinal Endpoints | |
| | 16.2. | | |
| _ | 16.2. | | |
| 1 | 6.3. | Exploratory Efficacy | |
| 1 | 6.4. | Additional Efficacy | 22 |

CCI

PPD

Version Number: Version Date: Amendment 2, v1.0 28-Jul-2021



| | 16.4. | 1. | Additional Efficacy Endpoint | 22 |
|---|---|---|---|---|
| | 16 | .4.1.1 | • | |
| | 16.4. | 2. | Missing Data Imputation Method for Additional Efficacy Endpoint | 22 |
| | 16.4. | 3. | Analysis of Additional Efficacy Endpoint | 22 |
| | 16.4. | 4. | Sensitivity Analyses for Additional Efficacy Endpoint | 22 |
| | 16.4. | 5. | Supplementary Analyses for Additional Efficacy Endpoint | 23 |
| 16 | 5.5. | Inter | rim Analysis | 23 |
| 17. | Safet | y End | lpoints | 23 |
| 17 | .1. | Adve | erse Events | 24 |
| | 17.1. | 1. | Adverse Events of Special Interest | 24 |
| 17 | .2. | Labo | pratory Evaluations | 25 |
| | 17.2. | 1. | Potential Hy's Law Events | 25 |
| 17 | <i>'.3.</i> | Vital | Signs | 25 |
| 17 | '.4. | Elect | rocardiogram Evaluations | 25 |
| 17 | <i>7.5.</i> | Phys | ical Examination | 25 |
| 18. | Phari | macol | kinetic Assessments | 25 |
| 18 | 3.1. | Deriv | vation | 26 |
| 19. | Phari | maco | dynamic and Other Biomarker Assessments | 26 |
| 20. | Anti- | Drug . | Antibody Testing | 27 |
| 21. | Data | Not S | Summarized or Presented | 28 |


#### 1. Introduction

This sub-protocol statistical analysis plan (SAP) describes the rules and conventions to be used in the presentation and analysis of data specific to COV-01-005 sub-protocol of Master Protocol COV-01. It describes the specific data to be summarized and analyzed, including specifics of the statistical analyses to be performed.

This sub-protocol SAP is based on sub-protocol version 1.2, dated 03-Nov-2020.

For the rules and conventions to be used in the presentation and analysis of data common across all sub-protocols, refer to the Master COV-01 SAP.

CCI

#### 2. STUDY OBJECTIVES

The study objectives are described in the Master COV-01 SAP.

## 3. STUDY DESIGN

#### 3.1. GENERAL DESCRIPTION

The general description is available in the Master COV-01 SAP.

#### 3.2. SCHEDULE OF ACTIVITIES

Schedule of activities can be found in Section 1.2 of COV-01-005 sub-protocol.

# 3.3. CHANGES TO ANALYSIS FROM MASTER PROTOCOL COV-01 AND SUB-PROTOCOL COV-01-005

Enrollment into sub-protocol COV-01-005 was prematurely terminated by the Sponsor on 07-Jun-2021. In conformance with the Food and Drug Administration (FDA) Guidance for Submission of Abbreviated Report and Synopsis in Support of Marking Application, an abbreviated Clinical Study Report (CSR) will be written for this

Version Number: Amendment 2, v1.0
Version Date: 28-Jul-2021

sub-protocol. As such, not all analyses initially planned in the Master Protocol COV-01 and Sub-protocol COV-01-005 will be performed for this sub-protocol (refer to Section COV-01-005 will be performed for this sub-protocol).

## 4. PLANNED ANALYSES

The analyses initially planned to be performed are listed and described in the Master COV-01 SAP. It is to be noted that enrollment into sub-protocol COV-01-005 was terminated early by the Sponsor on 07-Jun-2021 before the trigger for the two Interim Analyses (IAs) for futility and Primary Analysis have been reached (refer to Master SAP Sections 4.2 and 4.3, respectively). Hence, these analyses will not be performed for this sub-protocol and the only analysis that will be performed, in addition to the monthly IDMC Safety analyses, is the final analysis (refer to Section 4.4).

## 4.1. IDMC SAFETY ANALYSES

Details are provided in the Master COV-01 SAP.

### 4.2. INTERIM ANALYSES

No IAs will be performed for this sub-protocol (refer to Section 4).

## 4.3. PRIMARY ANALYSIS

No primary analysis will be performed for this sub-protocol (refer to Section 4).

#### 4.4. FINAL ANALYSIS

The final analysis for this sub-protocol will take place after:

All patients to be included in this sub-protocol final analysis who were ongoing at the time Sponsor terminated
early this sub-protocol completed the study (Day 60 visit) or discontinued early from the study, whichever
occurs first.

PPD Version Number: Amendment 2, v1.0 Version Date: 28-Jul-2021

- Sponsor Authorization of this SAP.
- Final database lock of the database including data from screen failed patients.
- Final database lock of the database of each sub-protocol contributing to the control arm of this sub-protocol (refer to Section 4.5).
- Final database lock of the database of this sub-protocol.

All planned analyses identified in this sub-protocol SAP will be performed by Biostatistics at the time of the final analysis of this sub-protocol.

## 4.5. SELECTION OF THE CONTROL ARM FOR AN ANALYSIS

#### 4.5.1. IDMC SAFETY ANALYSES

Details are provided in Master SAP Section 4.5.

#### 4.5.2. FINAL ANALYSIS

For final analysis of this sub-protocol, the control arm (also referred to as shared placebo plus standard of care (SoC) arm) will include all patients randomized to the placebo arm of any sub-protocol at a site at which:

- This sub-protocol was opened for enrollment.
- At least one patient was randomized to either this sub-protocol active (zilucoplan plus SoC) or placebo (placebo to zilucoplan plus SoC) arms.

That is, patients that satisfy these criteria will be included in the control arm of this sub-protocol regardless of 1) the timing of patient's randomization into a sub-protocol (i.e., regardless of if patient was randomized before or after this sub-protocol was opened for enrollment at the site) and 2) patient's eligibility to this sub-protocol specific inclusion/ exclusion criteria.

The purpose of this change from the Master SAP control arm definition (Master SAP Section 4.5) is to minimize the randomization imbalance issue noted by the CCI Unblinded Biostatistician and IDMC members at the time of At the time this sub-protocol SAP was finalized, the randomization imbalance was estimated to be approximately 7:1

PPD Version Number: Amendment 2, v1.0

between this sub-protocol active and control arms, should the original control arm definition would have been retained for the final analysis of this sub-protocol.

### 5. ANALYSIS SETS

Analysis sets are described in the Master COV-01 SAP.

Additional analysis sets that are specific to sub-protocol COV-01-005 are described below.

#### 5.1. PHARMACOKINETIC ANALYSIS SET

The pharmacokinetic (PK) analysis set will include patients from the safety analysis set (refer to Master COV-01 SAP Section 5.2) who were randomized to the zilucoplan plus SoC treatment arm and had at least one measured post-baseline concentration (refer to Master COV-01 SAP Section 6.2 for baseline definition).

## 5.2. PHARMACODYNAMIC ANALYSIS SET

The pharmacodynamic (PD) analysis set will include patients from the safety analysis set (refer to Master COV-01 SAP Section 5.2) who were randomized to COV-01-005 sub-protocol and had at least one measured biomarker (e.g., C5, etc.).

#### 5.3. ANTI-DRUG ANTIBODY ANALYSIS SET

The anti-drug antibody (ADA) analysis set will include patients from the safety analysis set (refer to Master COV-01 SAP Section 5.2) who were randomized to COV-01-005 sub-protocol and had at least one evaluated ADA sample (negative or positive).

#### 5.4. PROCESS FOR ANALYSIS SET ASSIGNMENT

As the PK, PD, and ADA analysis sets are defined based on objective criteria only, the authorization of this subprotocol SAP will stand for the agreement and authorization of the inclusion/exclusion of each patient in these PK, PD, and ADA analysis sets.

Version Number: Amendment 2, v1.0 Version Date: 28-Jul-2021

## 6. GENERAL CONSIDERATIONS

Details are provided in the Master COV-01 SAP.

## 7. STATISTICAL CONSIDERATIONS

## 7.1. SAMPLE SIZE CALCULATION

Details are defined in the Master COV-01 SAP.

## 7.2. MISSING DATA

Details are defined in the Master COV-01 SAP.

## 7.3. STATISTICAL TESTS

Not applicable since no statistical inferences will be performed for the final analysis of this sub-protocol (refer to Section 16).

## 7.4. MULTIPLE COMPARISONS/MULTIPLICITY

Not applicable since no statistical inferences will be performed for the final analysis of this sub-protocol (refer to Section 16).

## 7.5. MULTICENTER STUDY

Details are defined in the Master COV-01 SAP.

## 7.6. ADJUSTMENTS FOR COVARIATES AND FACTORS TO BE INCLUDED IN ANALYSES

Not applicable since no statistical inferences will be performed for the final analysis of this sub-protocol (refer to Section 16).

## 7.7. EXAMINATION OF SUBGROUPS

No subgroup analyses will be performed for the final analysis of this sub-protocol (refer to Section 16).

#### 7.8. SOFTWARE VERSION

Details are defined in the Master COV-01 SAP.

#### 8. OUTPUT PRESENTATIONS

Output presentations are described in the Master COV-01 SAP.

#### 9. DISPOSITION AND WITHDRAWALS

Analysis of disposition and withdrawals will be presented as described in the Master COV-01 SAP.

#### 10. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Demographic characteristics and other baseline characteristics data will be presented as described in the Master COV-01 SAP.

#### 11. DISEASE HISTORY

Analysis of disease history at screening will be performed as described in the Master COV-01 SAP.



### 12. MEDICAL HISTORY

Analysis of medical history will be performed as described in the Master COV-01 SAP.

## 13. PRIOR AND CONCOMITANT MEDICATIONS

In addition to the analysis of prior and concomitant medications described in the Master COV-01 SAP, antibiotic prophylaxis, collected on the *Antibiotic Prophylaxis* page of the electronic Case Report Form (eCRF), will also be coded to the World Health Organization (WHO) Drug Global dictionary, version B3 March 2020 (or later).

Concomitant use (refer to Master COV-01 SAP Section 13 for definition of concomitant use) of antibiotic for any indication as well as of antibiotic prophylaxis for Neisseria infection will be summarized separately by Anatomical Therapeutic Class (ATC) level 2, preferred drug name, and treatment arm based on the FAS (refer to Master COV-01 SAP Section 5.1). Separate summary of patients randomized to COV-01-005 placebo plus SoC treatment group will be provided. A patient having more than one medication within the same ATC level 2 or preferred drug name will be counted only once for that ATC level 2 or preferred drug name.

Furthermore, duration of concomitant use of antibiotic for any indication (days) and number and percentage of patients who received antibiotic prophylaxis for Neisseria infections concurrently while receiving the study drug and up to 14 days after the last dose of the study drug will be presented by treatment arm based on the FAS. Separate summary of patients randomized to COV-01-005 placebo plus SoC treatment group will be provided.

All antibiotic prophylaxis will be listed.

#### 13.1. DERIVATION

Duration of concomitant use of antibiotic for any indication, in days, will be derived as follows:

• Duration of concomitant use of antibiotic for any indication (days) = {[Date of latest stop date of any antibiotic received on or after the first dose of study drug – Latest of (date of earliest start date of antibiotic received on or after the first dose of study drug, date of first dose of study drug)] + 1} – [sum of any gap (days) in concomitant use of antibiotics for any indication on or after the first dose of study drug]

#### 14. EXPOSURE TO STUDY DRUG

#### Patients randomized to sub-protocol COV-01-005

Patients randomized to zilucoplan plus standard of care (SoC) and placebo plus SoC treatment arms of COV-01-005 sub-protocol will receive a single daily dose of 32.4 mg of the study drug (prefilled syringes containing 0.81 mL of zilucoplan or placebo, as appropriate) administered by subcutaneous (SC) injection in the abdomen (preferred site), thigh or upper arm.

The daily administration of study treatment will start on Day 1 (baseline) and continue to Day 14 or until hospital discharge, whichever occurs first. If the patient is discharged before 14 days of treatment, zilucoplan or placebo should be stopped at time of discharge or 24 hours before discharge.

Reason for dose modification of study drug (i.e. dose interrupted or drug withdrawal) will be captured in the *Exposure* page of the eCRF.

## Patients included in the control arm of COV-01-005 sub-protocol who were randomized to the placebo plus SoC group of a sub-protocol other than COV-01-005

It is to be noted that the planned duration of exposure to a study drug, planned frequency of administration of the study drug, and planned route of administration of the study drug will vary from one sub-protocol to the other, but similar information as for COV-01-005 sub-protocol will be captured on the *Exposure* page of the eCRF of these other sub-protocols.

#### Exposure to study drug

The exposure to study drug will be summarized by treatment arm (breaking down the placebo plus SoC arm by sub-protocol) based on the safety analysis set as follows:

- Duration of exposure:
  - Duration of exposure (days) as a continuous variable;
  - Ouration of exposure (days) as a categorical variable: 1 to 3, > 3 to 7, > 7 to 14, and > 14;
  - Total number of doses received as a continuous variable, where the total number of doses received is
    defined as the total number of doses received by each patient, not the total number of doses received
    across all patients.

PPD Version Number: Amendment 2, v1.0 Version Date: 28-Jul-2021

- Dose modifications:
  - o Number and percentage of patients with at least one interrupted dose;
  - Number and percentage of patients with at least one dose interruption by reason for dose interruptions:
    - Adverse events:
    - Other.
  - Total number of dose interruptions as a continuous variable, where the total number of dose interruptions is defined similarly to the total number of doses received;
- Number and percentage of patients with at least one overdose.

All dosing and exposure data will also be listed.

#### 14.1. DERIVATIONS

For patients randomized to a study drug planned to be administered on a daily basis, duration of exposure to study drug, in days, will be computed as follows:

• Duration of exposure (days) = (Date of last dose of study drug – Date of first dose of study drug) + 1

For all other patients (i.e. randomized to a study drug planned to be administered not on a daily basis), duration of exposure to study drug, in days, will be computed as follows:

Duration of exposure (days) = {[Earliest date of (end of planned study treatment period, hospital discharge or discontinuation from study drug)] – Date of first dose of study drug} + 1

#### 15. COMPLIANCE WITH STUDY DRUG

Compliance with study medication will be summarized by treatment arm (breaking down the placebo plus SoC control arm by sub-protocol) based on the safety analysis set. In addition to the descriptive summary, the following compliance categories will be presented:



- < 80%;
- $\geq 80\%$  to < 100%;
- 100%;
- > 100%.

Compliance data will also be listed.

## 15.1. DERIVATIONS

For each patient, the compliance will be computed as follows:

Compliance (%) = (Actual total number of doses / Expected total number of doses) x 100

#### where:

- Actual total number of doses is defined as the total number of doses (injections) taken (received) through the course of the study;
- Expected total number of doses is defined as the total number of protocol-defined doses (injections) to be taken (received) through the course of the study and is computed as follows:
  - o For patients randomized to a study drug administered on a daily basis:
    - Expected total number of doses = Expected number of doses (injections) per day \*
       expected number of days under treatment, where the expected number of days under treatment is defined as: {[Earliest date of (end of planned study treatment period, hospital discharged or discontinuation from study drug)] Date of first dose of study drug} + 1

- o For patients randomized to a study drug planned to be administered not on a daily basis:
  - Expected total number of doses = Expected number of doses (injections) per day \*
    expected number of administration days between randomization and the earliest of (end
    of planned study treatment period, hospital discharged or discontinuation from study
    drug)
- o For example, if a study drug is planned to be administered once on Day 1 and once on Day 4, the expected total number of doses is 2; unless patient discontinued from study drug or was discharged from the hospital on or after Day 1 but before Day 4, in which case the expected total number of doses is 1. As another example, if the study drug is planned to be administered twice daily on every other day from Day 1 to Day 14, the expected total number of doses is 14; unless patient discontinued from study drug or was discharged from the hospital let say, on Day 10, in which case the expected total number of doses is 10 (i.e., 2 doses [injection] per day \* 5 administration days).

## 16. EFFICACY ENDPOINTS

Given that only 108 patients were randomized into COV-01-005 sub-protocol by the time enrollment into this sub-protocol was terminated early by the Sponsor and that is expected that less than the third of the total number of patients required by the sample size (i.e., ~700; refer to Master SAP Section 7.1) will be included in the final analysis of this sub-protocol, no statistical inferences will be performed for any efficacy endpoint, but two-sided 95% confidence interval (CI) within each treatment arm will be provided, when possible.

In conformance with the FDA's Guidance for Submission of Abbreviated Report and Synopsis in Support of Marking, summary tables will be presented for the primary and key secondary efficacy endpoints (refer to Master SAP Sections 16.1.1, 16.2.1.1, 16.2.1.2, and 16.2.1.3). Although not required by the previously mentioned FDA's Guidance, summary tables will also be provided for the other secondary efficacy endpoints (refer to Master SAP Sections 16.2.1.4 to 16.2.1.9) in order to be compliant with the publication requirements of *ClinicalTrials.gov*. In addition, summary tables will also be provided for the additional efficacy endpoint of incidence of all-cause mortality through Day 60 (refer to Master SAP Section 16.4.1.1).

Efficacy summaries will be performed as described in the Master COV-01 SAP.


## 16.1. PRIMARY EFFICACY

## 16.1.1. TIME TO CONFIRMED CLINICAL RECOVERY THROUGH DAY 29, WITHOUT RE-HOSPITALIZATION THROUGH DAY 29

Details are provided in the Master COV-01 SAP.

#### 16.1.2. MISSING DATA IMPUTATION METHOD FOR PRIMARY EFFICACY ENDPOINT

Details are provided in the Master COV-01 SAP.

#### 16.1.3. MAIN ANALYSIS OF PRIMARY EFFICACY ENDPOINT

For the time to confirmed clinical recovery through Day 29, without re-hospitalization through Day 29, as defined in the Master SAP Section 16.1.1, the number and percentage of patients with and without the event will be presented by randomized treatment arm. Two-sided 95% exact binomial Confidence Interval (CI) will also be provided by treatment arm for the percentage of patients with the event. For patients who did not meet the event, the main reason for censoring will be summarized similarly.

Kaplan-Meier curves (product-limit estimate) will be provided by treatment arm for the time to confirmed clinical recovery though Day 29, without re-hospitalization through Day 29. Kaplan-Meier estimate of the time to confirmed clinical recovery through Day 29, without re-hospitalization through Day 29, in days, will be provided at the 25<sup>th</sup>, 50<sup>th</sup> (median), and 75<sup>th</sup> percentiles time along with their corresponding two-sided 95% CIs. The estimates of the SEs will be computed using the Greenwood's formula, the CI for the median will be calculated according to Brookmeyer and Crowley (1982), and the CIs for the survival function estimates at above mentioned time points will be derived from the Kaplan-Meier estimates using the log-log transformation. Kaplan-Meier estimates of the probability of having the event will also be provided at Day 29 along with the number of patients with the event and the number of patients at risk at that time.

#### 16.1.4. SENSITIVITY ANALYSES FOR PRIMARY EFFICACY ENDPOINT

No sensitivity analyses will be performed for this sub-protocol.


#### 16.1.5. SUPPLEMENTARY ANALYSES FOR PRIMARY EFFICACY ENDPOINT

No supplementary analyses will be performed for this sub-protocol.

## 16.2. SECONDARY EFFICACY

#### 16.2.1. SECONDARY EFFICACY ENDPOINTS

Details are provided in the Master COV-01 SAP.

#### 16.2.2. MISSING DATA IMPUTATION METHOD FOR SECONDARY EFFICACY ENDPOINTS

Details are provided in the Master COV-01 SAP.

#### 16.2.3. MAIN ANALYSIS OF SECONDARY EFFICACY ENDPOINTS

Details are provided in the Master COV-01 SAP.

#### 16.2.3.1. Binary Endpoints

For the incidence of patients with oxygen-free recovery at Day 29 (refer to Master SAP Section 16.2.1.1), incidence of patients with  $\geq$  2-point improvement from baseline or fit for discharge on the ordinal scale at Day 29 (refer to Master SAP Section 16.2.1.2), incidence of all-cause mortality through Day 29 (refer to Master SAP Section 16.2.1.3), incidence of patients with clinical recovery at Days 8, 15 and 29 (refer to Master SAP Section 16.2.1.8), and incidence of patients with sustained clinical recovery as confirmed by Day 60 follow-up (refer to Master SAP Section 16.2.1.9), the number and percentage of patients with and without the event will be provided by treatment arm. Two-sided 95% exact binomial CI will also be provided by treatment arm for the percentage of patients with the event.

For the incidence of all-cause mortality, primary reason of death will also be summarized by treatment arm.

#### 16.2.3.2. Ordinal Endpoints

For the incidence of patients in each category of the 8-point ordinal scale for clinical severity at Days 8, 15, and 29 endpoints (refer to Master SAP Section 16.2.1.4), the number and percentage of patients in each ordinal scale

PPD Version Number: Amendment 2, v1.0 Version Date: 28-Jul-2021

category will be provided at each specified Day for each treatment arm. The worst post-baseline score on the 8-point ordinal scale for clinical severity from randomization to Day 29 (refer to Master SAP Section 16.2.1.5) and each "number of days" endpoint (refer to Master SAP Sections 16.2.1.6 and 16.2.1.7) will be summarized similarly.

Shift tables from baseline to each post-baseline day up to Day 29 as well as to the worst post-baseline score will also be provided for the 8-point ordinal scale for clinical severity.

#### 16.2.4. SENSITIVITY ANALYSES FOR SECONDARY EFFICACY ENDPOINTS

No sensitivity analyses will be performed for this sub-protocol.

#### 16.2.5. SUPPLEMENTARY ANALYSES FOR SECONDARY EFFICACY ENDPOINTS

For the incidence of all-cause mortality through Day 29 key secondary efficacy endpoint, the time to all-cause mortality through Day 29, in days, associated will be derived as follows:

• Time to all-cause mortality through Day 29 (days) =

(Date of death / Date of censoring - Date of Study Day 1 [refer to Maser SAP Section 6.1]) + 1.

The date of death will be taken from data captured on the Death Details page of the eCRF.

For patients who were alive on Day 29, time to all cause-mortality will be censored at Day 29. For patients with an unknown alive status at the time of the analysis due to missing data, time to all-cause mortality will be censored at the latest date on which the patient was known to be alive before or on the data cut-off date of the analysis. The last date the patient was known to be alive will be the latest date collected on any page of the eCRF. For patients who discontinued from the study before the time of the analysis, time to all-cause mortality will be censored at the date of study discontinuation, as captured on the *Disposition* page of the eCRF.

Number and percentage of patients with and without the event will be presented by randomized treatment arm. For patients who did not meet the event, the main reason for censoring will be summarized similarly.

Kaplan-Meier survival curves by treatment arm will be provided. The 25<sup>th</sup> percentile, 50<sup>th</sup> percentile (median), and 75<sup>th</sup> percentile of time to all-cause mortality through Day 29 (days) with the corresponding two-sided 95% CIs based on the Kaplan-Meier survival curves (refer to Master SAP Section 16.2.4) for each treatment arm will also be presented. The estimate of the SEs will be computed using Greenwood's formula, the CI for the median will be calculated according to Brookmeyer and Crowley (1982) and the other CIs will be derived from the Kaplan-Meier


estimates using the log-log transformation. Kaplan-Meier estimates of the probability of having the event will also be provided at Day 29 along with the number of patients with the event and the number of patients at risk at that time.

No supplementary analyses will be performed for the any other secondary efficacy endpoints.

## 16.3. EXPLORATORY EFFICACY



## 16.4. ADDITIONAL EFFICACY

#### 16.4.1. ADDITIONAL EFFICACY ENDPOINT

#### 16.4.1.1. Incidence of All-Cause Mortality through Day 60

Details are provided in the Master COV-01 SAP.

#### 16.4.2. MISSING DATA IMPUTATION METHOD FOR ADDITIONAL EFFICACY ENDPOINT

Details are provided in the Master COV-01 SAP.

#### 16.4.3. ANALYSIS OF ADDITIONAL EFFICACY ENDPOINT

The number and percentage of patients alive and dead through Day 60 (refer to Section 16.4.1.1) will be provided by treatment arm along with the two-sided 95% exact binomial CI for the percentage of patients dead through Day 60. Primary reason of death will also be summarized by treatment arm.

#### 16.4.4. SENSITIVITY ANALYSES FOR ADDITIONAL EFFICACY ENDPOINT

No sensitivity analyses will be performed for the additional efficacy endpoint.



#### 16.4.5. Supplementary Analyses for Additional Efficacy Endpoint

The time to all-cause death through Day 60, in days, will be derived as follows:

• Time to all-cause mortality through Day 60 (days) =

(Date of death / Date of censoring - Date of Study Day 1 [refer to Maser SAP Section 6.1]) + 1.

The date of death will be taken from data captured on the *Death Details* page of the eCRF.

For patients who were alive or patients with an unknown alive status at the time of the analysis due to missing data, time to all-cause mortality will be censored at the latest date on which the patient was known to be alive before or on Day 60. The last date the patient was known to be alive will be the latest date collected on any page of the eCRF. For patients who discontinued from the study before Day 60, time to all-cause mortality will be censored at the date of study discontinuation, as captured on the *Disposition* page of the eCRF.

Number and percentage of patients with and without the event will be presented by treatment arm. For patients who did not meet the event, the main reason for censoring will be summarized similarly.

Kaplan-Meier survival curves by treatment arm will be provided. The 25<sup>th</sup> percentile, 50<sup>th</sup> percentile (median), and 75<sup>th</sup> percentile of time to all-cause mortality (days) through Day 60 with the corresponding two-sided 95% CIs based on the Kaplan-Meier survival curves for each treatment arm will be presented. The estimate of the SEs will be computed using Greenwood's formula, the CI for the median will be calculated according to Brookmeyer and Crowley (1982) and the CIs for the survival function estimates at above mentioned time points will be derived from the Kaplan-Meier estimates using the log-log transformation. Kaplan-Meier estimates of the probability of having the event will also be provided at Day 60 along with the number of patients with the event and the number of patients at risk at that time.

#### 16.5. INTERIM ANALYSIS

No IAs will be performed for this sub-protocol since the trigger for the first IA was not reached by the time enrollment into this sub-protocol was terminated early by Sponsor (refer to Master SAP Section 16.5).

#### 17. SAFETY ENDPOINTS

In addition to the safety analyses are described in Master COV-01 SAP, the following safety analysis will also be provided based on the safety analysis set (refer to Master SAP Section 5.2).



## 17.1. ADVERSE EVENTS

#### 17.1.1. ADVERSE EVENTS OF SPECIAL INTEREST

The following are defined as adverse events of special interest (AESIs) for this sub-protocol and will be identified based on pre-defined coded preferred terms (PTs), high-level terms (HLTs, and/or system organ class:

- Anaphylactic reactions (Medical Dictionary for Regulatory Activities [MedDRA] algorithmic approached; refer to Appendix 1);
- Serious anaphylactic reactions (MedDRA algorithmic approached; refer to Appendix 1);
- Hypersensitivity reactions (standardized MedDRA query [SMQ] narrow scope; refer to Appendix 2);
- Serious hypersensitivity reactions (SMQ narrow scope: refer to Appendix 2);
- Infections (MedDRA system organ class of 'Infections and infestations');
- Serious infections (MedDRA system organ class of 'Infections and infestations');
- Neisseria infections (MedDRA high level term [HLT] of 'Neisseria infections');
- Serious Neisseria infections (HLT of 'Neisseria infections');
- Drug related hepatic disorders (SMQ comprehensive search; refer to Appendix 3), excluding the 'Liver neoplasms, benign (incl. cysts and polyps)' and 'Liver neoplasms, malignant and unspecified' sub-SMQs.

A summary of treatment-emergent (refer to Master COV-01 SAP Section 17.1) AESIs overall and by AESI category and preferred term (PT) will be prepared by treatment arm for patients randomized to COV-01-005 only. Should a patient experience multiple events within an AESI category or PT, the patient will be counted only once for that AESI category or PT. The risk difference of the overall incidence rates of having any treatment-emergent AESI between the treatment arms will be presented along with its two-sided 95% Wald CI. A listing of all AESIs will be provided for patients randomized to COV-01-005 only.

#### 17.2. LABORATORY EVALUATIONS

#### 17.2.1. POTENTIAL HY'S LAW EVENTS

In addition to the laboratory analyses described in the Master COV-01 SAP for the identification of the potential Hy' law events, the following summary will also be provided:

Number and percentages of patients with (ALT > 3 x ULN or AST > 3 x ULN) AND (total bilirubin > 2 x ULN) AND (alkaline phosphatase [ALP] < 2 x ULN) at any time after the first dose of study drug and by visit for each treatment arm as well as for the subset of patients randomized to the placebo to zilucoplan + SoC treatment arm.</li>

#### 17.3. VITAL SIGNS

Analysis of vital signs is described in the Master COV-01 SAP.

#### 17.4. ELECTROCARDIOGRAM EVALUATIONS

Analysis of electrocardiogram (ECG) evaluations is described in the Master COV-01 SAP.

#### 17.5. PHYSICAL EXAMINATION

Analysis of physical examination is described in the Master COV-01 SAP.

#### 18. PHARMACOKINETIC ASSESSMENTS

Concentrations of zilucoplan will be summarized descriptively at each scheduled assessment based on the PK analysis set (refer to Section 5.1). Geometric mean (geoMean), geometric coefficient of variation (geoCV) and 95% CI for the geoMean will also be presented in the summaries of zilucoplan concentration data. Geometric coefficient of variation will be reported as a percentage to 1 decimal place and the 95% CI for the geoMean will use the same number of decimal places as the geoMean. It will be left blank if the geoCV is 0.

When reporting individual zilucoplan concentration data in listings and presenting summary statistics in tables, the following rules will apply:



- Missing data should be reported as 'NV' (no value) in the listings;
- Concentrations below the lower limit of quantification (LLOQ) should be reported as BLQ (below the limit of quantification) in the listings;
- To calculate summary statistics, BLQ values should be set to half the LLOQ value and missing values should be excluded;
- When the total number of BLQ and missing values exceeds one third of the total then only minimum and maximum should be reported for this scheduled assessment. Other summary statistics should be reported as missing ("-"). The minimum should be reported as BLQ;
- When the mean value includes one or more replaced BLQ values then a footnote should be included to say "contains one or more BLQ values replaced by half the LLOQ value";
- A minimum of 3 values are required to calculate summary statistics. If only 2 values are available, then these should be presented as the minimum and maximum with other summary statistics reported as missing ("-").

Zilucoplan concentrations will be listed.

## 18.1. DERIVATION

The geoCV, in percentage, will be calculated using the following formula where SD is the standard deviation from the log-transformed data:

• GeoCV (%) =  $sqrt[exp(SD^2) - 1] \times 100$ 

## 19. PHARMACODYNAMIC AND OTHER BIOMARKER ASSESSMENTS





#### 20. ANTI-DRUG ANTIBODY TESTING

Number and percentage of patients with a negative ADA response (i.e., either [negative screen] or [positive screen and negative immunodepletion]) and a positive ADA response (i.e., positive screen and positive immunodepletion) will be summarized by scheduled visit and treatment arm based on the ADA analysis set (refer to Section 5.3).

Number and percentage of patients in each of the following categories will also be summarized by treatment arm:

- 1. Treatment-induced ADA negative, defined as patients who were ADA negative at baseline as well as at all post-baseline scheduled visit;
- 2. Treatment-induced ADA positive, defined as patients who were ADA negative at baseline and ADA positive at at least one post-baseline scheduled visit. This category also includes patients with a missing ADA response status at baseline who had at least one ADA positive response at any post-baseline scheduled visit;
- 3. Treatment-reduced ADA, defined as patients who were ADA positive at baseline and ADA negative at all post-baseline scheduled visit:
- 4. Treatment-unaffected ADA, defined as patients who were ADA positive at baseline and ADA positive at at least one post-baseline scheduled visit with titer values of the same magnitude as baseline (i.e., equal or less than a pre-defined fold difference increase from the baseline value, where the pre-defined fold difference increase from the baseline value is defined as the minimum significant ratio [MSR] determined during assay validation);
- 5. Treatment-boosted ADA positive, defined as patients who were ADA positive at baseline and ADA positive at at least one post-baseline scheduled visit with increased in titer values as compare to baseline (i.e., greater than the pre-defined fold difference increase from baseline value);
- 6. Inconclusive, defined as patients who were ADA negative or positive at baseline for whom some post-baseline ADA response assessments are missing, while all other post-baseline ADA response assessments are ADA negative;
- 7. Total prevalence of pre-Ab i.e., patients in categories 3, 4, and 5 combined;
- 8. Total incidence of treatment-emergent ADA positive i.e., patients in categories 2 and 5 combined.


The fold difference increase from baseline (i.e., the MSR determined during the assay validation) needed to consider a titer value reported post-baseline to be above the assay validation will be noted in the relevant tables and listings.

All ADA data will be listed.

## 21. DATA NOT SUMMARIZED OR PRESENTED

The list of data not summarized or presented is available in the Master COV-01 SAP.

## APPENDIX 1 MEDDRA ALGORITHMIC APPROACH TO ANAPHYLAXIS

The SMQ anaphylactic reactions consists of three parts:

A narrow search containing PTs that represent core anaphylactic reaction terms:

#### Category A

- Anaphylactic reaction
- Anaphylactic shock
- Anaphylactic transfusion reaction
- Anaphylactoid reaction
- Anaphylactoid shock
- Circulatory collapse
- Dialysis membrane reaction
- Kronis syndrome
- Shock
- Shock symptom
- Type I hypersensitivity

A broad search that contains additional terms that are added to those included in the narrow search. These additional terms are signs and symptoms possibly indicative of anaphylactic reaction and categorized in B, C or D.

| Category B (Upper Airway/ Respiratory) | | | | | |
|---|---|---|---|---|---|
| 0 | Acute respiratory failure | 0 | Irregular breathing | 0 | Respiratory failure |
| 0 | Asthma | 0 | Laryngeal dyspnea | 0 | Reversible airways obstruction |
| 0 | Bronchial oedema | 0 | Laryngeal oedema | 0 | Sensation of foreign body |
| 0 | Brochospasm | 0 | Laryngospasm | 0 | Sneezing |
| 0 | Cardio-respiratory distress | 0 | Laryngotracheal oedema | 0 | Stridor |
| 0 | Chest discomfort | 0 | Mouth swelling | 0 | Swollen tongue |
| 0 | Chocking | 0 | Nasal obstruction | 0 | Tachypnoea |
| 0 | Chocking sensation | 0 | Oedema mouth | 0 | Throat tightness |
| 0 | Circumoral oedema | 0 | Oropharyngeal spasm | 0 | Tongue oedema |
| 0 | Cough | 0 | Oropharyngeal swelling | 0 | Tracheal obstruction |
| 0 | Cyanosis | 0 | Respiratory arrest | 0 | Tracheal oedema |
| 0 | Dyspnoea | 0 | Respiratory distress | 0 | Upper airway obstruction |
| 0 | Hyperventilation | 0 | Respiratory dyskinesia | 0 | Wheezing |
| Cate | egory C (Angioedema/ Urticaria | / Prı | uritus/ Flush) | | |
| 0 | Allergic oedema | 0 | Injection site urticaria | 0 | Rash |
| 0 | Angioedema | 0 | Lip oedema | 0 | Rash erythematous |
| 0 | Erythema | 0 | Lip swelling | 0 | Rash generalized |




Amendment 2, v1.0 28-Jul-2021






| e | gory C (Angioedema/ Urticar | ia/ Pru | ritus/ Flush) | | |
|---|---|---|---|---|---|
| | Eye oedema | 0 | Nodular rash | 0 | Rash pruritic |
| | Eye pruritus | 0 | Ocular hyperaemia | 0 | Skin swelling |
| | Eye swelling | 0 | Oedema | 0 | Swelling |
| , | Eyelid oedema | 0 | Periorbital oedema | 0 | Swelling face |
| ) | Face oedema | 0 | Pruritus | 0 | Urticaria |
| , | Flushing | 0 | Pruritus allergic | 0 | Urticaria papular |
| ) | Generalised erythema | 0 | Pruritus generalised | | |
| te | gory D (Cardiovascular / Hyp | otensi | on) | | |
| ) | Blood pressure decreased | 0 | Cardiac arrest | 0 | Diastolic hypotension |
| ) | Blood pressure diastolic decreased | 0 | Cardio-respiratory arrest | 0 | Hypotension |
| ) | Blood pressure systolic decreased | 0 | Cardiovascular insufficiency | | |


Amendment 2, v1.0 28-Jul-2021


- An algorithm approach which combines a number of anaphylactic reaction symptoms in order to increase
  specificity will be used for this sub-protocol. A potential anaphylactic reaction is defined meeting at least one
  of the following criteria where the different terms occur on either the same day as when an injection was
  administered or one day after:
  - o A narrow PT from Category A;
  - o A PT from Category B AND a PT from Category C;
  - o A PT from Category D AND (a PT from Category B OR a term from Category C).

Version Number: Amendment 2, v1.0 Version Date: 28-Jul-2021
# APPENDIX 2 SMQ OF HYPERSENSITIVITY REACTIONS (NARROW SCOPE)

#### **Preferred Term**

- Administration site hypersensitivity
- Documented hypersensitivity to administered product
- Drug hypersensitivity
- Hypersensitivity
- Infusion related hypersensitivity reaction
- Infusion site hypersensitivity
- Injection site hypersensitivity
- Type I hypersensitivity
- Type II hypersensitivity
- Type IV hypersensitivity

PPD


# APPENDIX 3 SMQ OF DRUG RELATED HEPATIC DISORDERS (COMPREHENSIVE SEARCH)

| Preferred Term | Preferred Term | | |
|---|---|---|---|
| • 5'nucleotidase incr | eased | • | Acute graft versus host disease in liver |
| • Abnormal LFTs | | • | Acute hepatic congestion |
| Abnormal liver fur | nction tests | • | Acute hepatic failure |
| • Acholia | | • | Acute liver damage |
| Acquired afibrinog | genaemia | • | Acute liver failure |
| Acquired afibrinog | enemia | • | Acute liver injury |
| Acquired antithron | nbin III deficiency | • | Acute on chronic hepatic failure |
| Acquired factor IX | deficiency | • | Acute on chronic liver failure |
| Acquired factor VI | II deficiency | • | Acute yellow liver atrophy |
| Acquired factor XI | deficiency | • | Advanced chronic liver disease |
| Acquired fibrinoge | en deficiency | • | Aggravated bilirubinemia |
| Acquired hepatoce | rebral degeneration | • | Alanine aminotransferase abnormal |
| Acquired protein S | deficiency | • | Alanine aminotransferase abnormal NOS |
| Acute cholestatic h | nepatitis | • | Alanine aminotransferase increase |
| Acute cytolytic hep | patitis | • | Alanine aminotransferase increased |
| Acute derangemen | t of liver function | • | Alkaline phosphatase raised |
| Acute fatty liver | | • | Alkaline phosphatase increased |



PPD

Acute fulminant hepatitis


Alkaline phosphatase NOS increased



| Pr | efe | rred | Teri | n |
|----|-----|------|------|---|

- Alkaline phosphatase serum increased
- Allergic hepatitis
- Alloimmune hepatitis
- ALP increased
- Al-P increased
- ALPPS
- ALT flare up
- ALT high
- ALT increased
- Ammonia abnormal
- Ammonia abnormal NOS
- Ammonia increased
- Angioma spider
- Anicteric cholestasis
- Anorectal varices
- Anorectal varices bleeding
- Anorectal varices hemorrhage
- Anti factor X activity abnormal
- Anti factor X activity decreased

- Antithrombin III decreased
- Artificial extracorporeal liver support
- Ascites
- Ascites chylous
- Aspartate aminotransferase abnormal
- Aspartate aminotransferase abnormal NOS
- Aspartate aminotransferase increase
- Aspartate aminotransferase increased
- Associating liver partition and portal vein ligation for staged hepatectomy
- AST flare up
- AST high
- AST increased
- AST/ALT ratio abnormal
- Asterixis
- AT-3 decreased
- Atrophy liver
- Atrophy of hepatocytes
- Autoimmune hepatitis
- Anti factor X activity increased

PPD




| Pr | efe | rred | Teri | n |
|----|-----|------|------|---|

- Bacterascites
- Bile output abnormal
- Bile output decreased
- Biliary ascites
- Biliary cirrhosis
- Biliary cirrhosis NOS
- Biliary cirrhosis primary
- Biliary cirrhosis secondary
- Biliary enzyme increased
- Biliary fibrosis
- Biliary stasis
- Bilirubin abnormal
- Bilirubin conjugated abnormal
- Bilirubin conjugated increased
- Bilirubin elevated
- Bilirubin excretion disorder
- Bilirubin excretion disorder NOS
- Bilirubin increased
- Bilirubin indirect increased
- Bilirubin non-glucuronides high

- Bilirubin total abnormal
- Bilirubin total high
- Bilirubin total increased
- Bilirubin unconjugated increased
- Bilirubin urine present
- Bilirubin value increased
- Bilirubinaemia
- Bilirubinaemia aggravated
- Bilirubinemia
- Bilirubinemia aggravated
- Biliverdin increased
- Biopsy liver abnormal
- Bleeding esophageal varices
- Bleeding oesophageal varices
- Blood alkaline phosphatase abnormal
- Blood alkaline phosphatase bone increased
- Blood alkaline phosphatase high
- Blood alkaline phosphatase increased
- Blood alkaline phosphatase intestine increased
- Blood alkaline phosphatase liver increased

PPD




- Blood alkaline phosphatase NOS increased
- Blood alkaline phosphatase placental increased
- Blood alkaline phosphatase renal abnormal
- Blood alkaline phosphatase renal increased
- Blood antithrombin III low
- Blood bilirubin abnormal
- Blood bilirubin increased
- Blood bilirubin indirect increased
- Blood bilirubin unconjugated increased
- Blood cholinesterase abnormal
- Blood cholinesterase decreased
- Blood fibrinogen abnormal
- Blood fibrinogen abnormal NOS
- Blood fibrinogen decreased
- Blood galactose tolerance abnormal
- Blood thrombin abnormal
- Blood thrombin abnormal NOS
- Blood thrombin decreased
- Blood thromboplastin abnormal
- Blood thromboplastin abnormal NOS

- Blood alkaline phosphatase NOS abnormal
- Blood thromboplastin decreased
- Bone alkaline phosphatase increased
- Bromosulphthalein retention
- Bromosulphthalein test abnormal
- Bromsulphalein retention
- Bromsulphthalein retention
- Bruised liver
- BSP abnormal
- BSP excretion delayed
- Caput medusae
- Cardia variceal ligation
- Cardiohepatic syndrome
- Charcot's cirrhosis
- Child-Pugh-Turcotte score abnormal
- Child-Pugh-Turcotte score increased
- Child-Turcotte-Pugh class A
- Child-Turcotte-Pugh class B
- Child-Turcotte-Pugh class C
- Cholemia

<u>CCI</u>

PPD




| Pr | eferi | red | Term |
|----|-------|-----|------|

- Cholestasis extrahepatic
- Cholestasis intrahepatic
- Cholestatic hepatic disorder
- Cholestatic hepatitis
- Cholestatic icterus
- Cholestatic jaundice
- Cholestatic liver disease
- Cholestatic liver injury
- Cholestatic pruritus
- Cholinesterase blood decreased
- Cholinesterase decreased
- Cholinesterase low
- Chronic active hepatitis
- Chronic graft versus host disease in liver
- Chronic hepatic failure
- Chronic hepatitis
- Chronic hepatitis, unspecified
- Chronic hepatopathy due to metabolic defect
- Chronic liver disease
- Chronic liver injury

- Cholestasis
- Chronic non-suppurative destructive cholangitis
- Chronic passive congestion of liver
- Chronic persistent hepatitis
- Chylous ascites
- Cirrhosis biliary
- Cirrhosis liver
- Cirrhosis liver post necrotic
- Cirrhosis liver postnecrotic
- Cirrhosis of liver
- Cirrhosis of liver without mention of alcohol
- Coagulation factor decreased
- Coagulation factor II level abnormal NOS
- Coagulation factor II level decreased
- Coagulation factor IX level abnormal
- Coagulation factor IX level abnormal NOS
- Coagulation factor IX level decreased
- Coagulation factor IX level low
- Coagulation factor V level abnormal
- Coagulation factor V level abnormal NOS

PPD




- Coagulation factor V level low
- Coagulation factor VII level abnormal
- Coagulation factor VII level abnormal NOS
- Coagulation factor VII level decreased
- Coagulation factor VII level low
- Coagulation factor X level abnormal
- Coagulation factor X level abnormal NOS
- Coagulation factor X level decreased
- Coagulation factors decreased
- Coloring yellow
- Colouring yellow
- Coma hepatic
- Compensated cirrhosis
- Complications of transplanted liver
- Computerized tomogram liver
- Computerized tomogram liver abnormal
- Congestive gastropathy
- Conjugated bilirubin level increased
- Conjugated bilirubin level raised
- Conjugated bilirubinaemia

- Coagulation factor V level decreased
- Conjugated bilirubinemia
- Conjunctiva bulbi coloring yellow
- Conjunctiva bulbi colouring yellow
- Conjunctiva coloring yellow
- Conjunctiva colouring yellow
- Cruveilhier-Baumgarten syndrome
- Cryptogenic cirrhosis
- CT scan liver
- Cytolytic hepatitis
- Damage liver
- De Ritis ratio abnormal
- Decompensated cirrhosis
- Decreased INR
- Decreased plasma fibrinogen
- Deficiency of bile secretion
- Degeneration fatty liver
- Deranged liver function tests
- Derangement of liver function tests
- Diabetic hepatopathy

CCL

PPD




| Pref | erred | Term |
|------|-------|------|

- DILI
- Direct bilirubin abnormal
- Direct bilirubin increased
- Direct hyperbilirubinaemia
- Direct hyperbilirubinemia
- Disease hepatocellular
- Disorder hepatic
- Disorder liver
- Disturbance of liver function tests
- Drug-induced hepatitis
- Drug-induced hepatotoxicity
- Drug-induced liver disease
- Drug-induced liver injury
- Duodenal varices
- Dyscholia
- Dyscholia
- Dysfunction hepatic non-icteric
- Edema due to hepatic disease
- Elevated liver enzyme levels
- Elevated liver enzymes

- Encephalopathy hepatic
- End stage liver disease
- Esophageal varices
- Esophageal varices hemorrhage
- Esophageal varices in cirrhosis of liver
- Esophageal varices ruptured
- Esophageal varices with bleeding
- Esophageal varices without mention of bleeding
- Esophagogastric devascularization
- Exaggerated hypoprothrombinemia
- Failure hepatorenal
- Failure liver
- Fatty liver
- Fatty liver infiltration
- Fatty liver metamorphosis
- Fetor hepaticus
- Fibrinogen decreased
- Fibrinogen plasma decreased
- Fibrinogenopenia
- Fibrinopenia



PPD




| Pr | efe | rred | Teri | n |
|----|-----|------|------|---|

- Fibrosis biliary
- Fibrosis liver
- Flapping tremor
- Focal hepatic steatosis
- Foetor hepaticus
- Fulminant hepatic failure
- Function liver abnormal
- Function liver decreased
- Function tests multiple liver abnormal
- Galactose elimination capacity test abnormal
- Galactose elimination capacity test decreased
- Gallbladder ejection fraction decreased
- Gallbladder varices
- Gamma glutamyl transpeptidase increased
- Gamma GT abnormal
- Gamma GT increased
- Gamma GT raised
- Gamma-glutamyltransferase abnormal
- Gamma-glutamyltransferase abnormal NOS

- Gamma-glutamyltransferase high
- Gamma-glutamyltransferase increased
- Gammaglutamyltranspeptidase abnormal
- Gamma-GT increased
- Gastric variceal injection
- Gastric variceal ligation
- Gastric varices
- Gastric varices bleeding
- Gastric varices hemorrhage
- Gastric varices ruptured
- Gastroesophageal variceal hemorrhage prophylaxis
- Gastroesophageal varices
- Gastroesophageal varices hemorrhage
- Gastrooesophageal variceal hemorrhage prophylaxis
- Gastrooesophageal varices
- Gastrooesophageal varices haemorrhage
- GGT increased
- GGTP abnormal
- GGTP increase

PPD




- Glutamate dehydrogenase increased
- Glutamic-oxaloacetic transaminase increased
- Glutamic-pyruvate transaminase increased
- Glutamic-pyruvic transaminase increased
- Glycocholic acid increased
- Glycogenic hepatopathy
- GOT abnormal
- GOT increased
- GOT increased transient
- GPT abnormal
- GPT increased
- GPT increased transient
- Graft versus host disease in liver
- Granulomatous liver disease
- Guanase increased
- Hanot's cirrhosis
- Hemihepatectomy
- Hemorrhagic ascites
- Hepaplastin abnormal
- Hepaplastin decreased

- Hepaplastin value decreased
- Hepaplastin low
- Hepatectomy
- Hepatectomy NOS
- Hepatic artery flow decreased
- Hepatic atrophy
- Hepatic calcification
- Hepatic cirrhosis
- Hepatic cirrhosis NOS
- Hepatic cirrhosis post necrotic
- Hepatic coma
- Hepatic congestion
- Hepatic cyst excision
- Hepatic cytolysis
- Hepatic damage
- Hepatic damage (NOS)
- Hepatic decompensation
- Hepatic disease
- Hepatic disease NOS
- Hepatic disorder aggravated

CCI

PPD




| Pr | eferi | red | Term |
|----|-------|-----|------|

- Hepatic disorder NOS
- Hepatic dysfunction allergic
- Hepatic dysfunction non-icteric
- Hepatic dysfunction NOS
- Hepatic dysfunction transient
- Hepatic encephalopathy
- Hepatic encephalopathy prophylaxis
- Hepatic enzyme abnormal
- Hepatic enzyme decreased
- Hepatic enzyme increased
- Hepatic enzymes increased
- Hepatic failure
- Hepatic fibrosis
- Hepatic fibrosis marker abnormal
- Hepatic fibrosis marker increased
- Hepatic function abnormal
- Hepatic function abnormal NOS
- Hepatic function decreased
- Hepatic function disorder
- Hepatic granuloma

- Hepatic hydrothorax
- Hepatic hypertrophy
- Hepatic impairment
- Hepatic induced edema
- Hepatic induced oedema
- Hepatic infiltration eosinophilic
- Hepatic insufficiency
- Hepatic intracellular deposit of bilirubin
- Hepatic intracellular pigmentation
- Hepatic lesion
- Hepatic lesion NOS
- Hepatic lipogranuloma
- Hepatic lobule necrosis
- Hepatic lymphocytic infiltration
- Hepatic macrosteatosis
- Hepatic mass
- Hepatic microsteatosis
- Hepatic necrosis
- Hepatic necrosis extensive
- Hepatic pain

CCL

PPD




| Pr | eferi | red | Term |
|----|-------|-----|------|

- Hepatic sequestration
- Hepatic shock
- Hepatic size reduced
- Hepatic steato-fibrosis
- Hepatic steatosis
- Hepatic trauma
- Hepatic vascular resistance increased
- Hepatic venous pressure gradient abnormal
- Hepatic venous pressure gradient increased
- Hepatitis
- Hepatitis acute
- Hepatitis acute toxic
- Hepatitis aggravated
- Hepatitis allergic drug-induced
- Hepatitis autoimmune
- Hepatitis cholestatic
- Hepatitis chronic active
- Hepatitis chronic active (immune)
- Hepatitis chronic active aggravated
- Hepatitis chronic NOS

- Hepatitis chronic persistent
- Hepatitis drug-induced
- Hepatitis flare
- Hepatitis fulminant
- Hepatitis granulomatous
- Hepatitis granulomatous NOS
- Hepatitis necrotising
- Hepatitis necrotizing
- Hepatitis non-icteric
- Hepatitis nonspecific
- Hepatitis NOS
- Hepatitis reactive non-specific
- Hepatitis symptom
- Hepatitis toxic
- Hepatitis toxic drug-induced
- Hepatitis toxic obstructive
- Hepatitis, unspecified
- Hepatobiliary disease
- Hepatobiliary disease NOS
- Hepatobiliary insufficiency

CCL

PPD




| Pr | eferi | red | Term |
|----|-------|-----|------|

- Hepatobiliary pain
- Hepatobiliary scan abnormal
- Hepatocellular abnormality
- Hepatocellular damage
- Hepatocellular damage aggravated
- Hepatocellular damage NOS
- Hepatocellular disturbances
- Hepatocellular foamy cell syndrome
- Hepatocellular injury
- Hepatomegaly
- Hepatopathy
- Hepatopulmonary syndrome
- Hepatorenal failure
- Hepatorenal syndrome
- Hepatosis
- Hepatosis aggravated
- Hepatosplenomegaly
- Hepatosplenomegaly NOS
- Hepatotoxic effect
- Hepatotoxicity

- Hepatotoxicity aggravated
- Hepatotoxicity NOS
- Hyperammonemia
- Hyperbilirubinaemia aggravated
- Hyperbilirubinemia
- Hyperbilirubinemia aggravated
- Hypercholia
- Hyperfibrinolysis
- Hypertension portal
- Hypertransaminasaemia
- Hypertransaminasemia
- Hypertrophic cirrhosis
- Hypoalbuminemia
- Hypocholia
- Hypocoagulable state
- Hypofibrinogenemia
- Hypohepatia
- Hypoprothrombinemia
- Hypothrombinemia
- Hypothromboplastinaemia

PPD




| Pr | efe | rred | Term |
|----|-----|------|------|

- Hypothromboplastinemia
- Hy's law case
- Icteric conjunctivae
- Icteric sclera
- Icterus
- Icterus index increased
- Idiopathic portal hypertension
- Immune-mediated hepatitis
- Impaired liver function
- Increased liver stiffness
- Indirect bilirubin increased
- Indirect hyperbilirubinaemia
- Indirect hyperbilirubinemia
- Infiltration fatty liver
- Injury to liver
- Injury to liver with open wound into cavity
- Injury to liver with open wound into cavity, unspecified laceration
- Injury to liver without mention of open wound into cavity

- INR abnormal
- INR decreased
- INR increased
- International normalised ratio abnormal NOS
- International normalized ratio abnormal
- International normalized ratio decreased
- International normalized ratio increased
- Intestinal varices
- Intestinal varices bleeding
- Intestinal varices hemorrhage
- Intra-abdominal venous shunt
- Intrahepatic portal hepatic venous fistula
- Ischemic hepatitis
- Jaundice
- Jaundice (excl neonatal)
- Jaundice cholestatic
- Jaundice hepatocellular
- Jaundice NOS

PPD




| Pr | eferi | red | Term |
|----|-------|-----|------|

| Pr | eferred Term | | |
|---|---|---|---|
| • | Jaundice, unspecified, not of newborn | • | Liver cirrhosis |
| • | Kayser-Fleischer ring | • | Liver cholestasis |
| • | Kupffer cell decrease | • | Liver contusion |
| • | Kupffer cell increase | • | Liver damage |
| • | Laceration of liver, major, with open wound into cavity | • | Liver damage aggravated |
| • | Laceration of liver, major, without mention of open wound into cavity | • | Liver dialysis |
| • | Laceration of liver, minor, with open wound into cavity | • | Liver disorder |
| • | Laceration of liver, minor, without mention of open wound into cavity | • | Liver enlargement |
| • | Laceration of liver, moderate, with open wound into cavity | • | Liver enzyme abnormal |
| • | Laceration of liver, moderate, without mention of open wound into cavity | • | Liver failure |
| • | Leucine aminopeptidase increased | • | Liver fatty |
| • | LFTs raised | • | Liver fatty change |
| • | Liver and pancreas transplant rejection | • | Liver fatty degeneration |
| • | Liver and small intestine transplant | • | Liver fatty deposit |
| • | Liver biopsy abnormal | • | Liver fatty deposition |
| • | Liver cell damage | • | Liver fatty infiltration |






| Pr | efer | red | Term |
|----|------|-----|------|

- Liver fatty metamorphosis
- Liver fatty phanerosis
- Liver function test abnormal
- Liver function test decreased
- Liver function test increased
- Liver function tests abnormal
- Liver function tests abnormal NOS
- Liver function tests NOS abnormal
- Liver function tests raised
- Liver graft dysfunction
- Liver graft function delayed
- Liver graft loss
- Liver induration
- Liver inflammation
- Liver injury
- Liver iron concentration abnormal
- Liver iron concentration increased
- Liver lobectomy
- Liver necrosis

- Liver nodule
- Liver operation
- Liver operation NOS
- Liver pain
- Liver palpable
- Liver palpable subcostal
- Liver repair
- Liver resection
- Liver retransplantation
- Liver sarcoidosis
- Liver scan abnormal
- Liver scan NOS abnormal
- Liver tender
- Liver tenderness
- Liver tenderness of
- Liver transplant
- Liver transplant failure
- Liver transplant rejection
- Liver transplantation

PPD




| P | ref | er | red | I T | 'erm |
|---|-----|----|-----|-----|------|

- Living donor liver transplant
- Lupoid hepatic cirrhosis
- Lupus hepatitis
- Magnetic resonance imaging liver abnormal
- Magnetic resonance proton density fat fraction measurement
- MELD score abnormal
- MELD score increased
- Mesenteric varices
- Mesocaval shunt
- Metabolic liver injury
- Metamorphosis fatty liver
- Micronodular cirrhosis
- Microvesicular fat disease of liver
- Minimal hepatic encephalopathy
- Mitochondrial aspartate aminotransferase increased
- Mixed hepatocellular-cholestatic injury
- Mixed liver injury
- Model for end stage liver disease score abnormal
- Model for end stage liver disease score increased

- Molar ratio of total branched-chain amino acid to tyrosine
- Monomicrobial non-neutrocytic bacterascites
- MRI-PDFF
- Multivisceral transplantation
- Naevus spider acquired
- Necrosis hepatocellular
- Necrosis liver
- Necrosis liver focal
- Nevus spider acquired
- Nodular regenerative hyperplasia
- Non-alcoholic fatty liver
- Nonalcoholic fatty liver disease
- Non-alcoholic steatohepatitis
- Non-cirrhotic portal fibrosis
- Non-cirrhotic portal hypertension
- Nonspecific abnormal results of function study of liver
- Nonspecific hepatitis
- Nuclear magnetic resonance imaging liver abnormal
- Obstructive jaundice

PPD




- Ocular icterus
- Oesophageal varices in cirrhosis of liver
- Oesophageal varices NOS
- Oesophageal varices ruptured
- Oesophageal varices with bleeding
- Oesophageal varices without mention of bleeding
- Oesophagogastric devascularisation
- Oligocholia
- Orthotopic liver transplant
- Parenteral nutrition associated cholestasis
- Parenteral nutrition associated liver disease
- Partial hepatectomy
- Partial splenic embolization
- Pericardial devascularization
- Perihepatic discomfort
- Perihepatic fluid collection
- Perinatal jaundice due to hepatocellular damage
- Peripancreatic varices
- Periportal edema
- Peritoneal effusion

- Peritoneal effusion (chronic)
- Peritoneal effusion bloody
- Peritoneal fluid protein abnormal
- Peritoneal fluid protein decreased
- Peritoneal fluid protein increased
- Peritoneovenous shunt
- Phanerosis fatty liver
- Phosphatase alkaline increased
- Plasma cholinesterase decreased
- Plasma fibrinogen abnormal
- Plasma thrombin abnormal
- Plasma thrombin decreased
- Plasma thromboplastin abnormal
- Plasma thromboplastin decreased
- Pneumobilia
- Polymicrobial bacterascites
- Portacaval shunt
- Portal anastomosis
- Portal fibrosis
- Portal hypertension

CCL

PPD




| D. | 4 | · | | Terr | |
|----|-----|----|-----|------|---|
| rı | rei | er | rea | ren | п |

- Portal hypertensive colopathy
- Portal hypertensive enteropathy
- Portal hypertensive gastropathy
- Portal shunt
- Portal shunt procedure
- Portal systemic shunt
- Portal systemic shunt procedure
- Portal tract inflammation
- Portal triaditis
- Portal vein cavernous transformation
- Portal vein dilatation
- Portal vein enlarged
- Portal vein flow decreased
- Portal vein pressure increased
- Portopulmonary hypertension
- Prehepatic portal hypertension
- Primary biliary cholangitis
- Primary biliary cirrhosis
- Primary liver transplant nonfunction
- Prophylaxis of gastroesophageal variceal bleeding

- Prophylaxis of gastrooesophageal variceal bleeding
- Protein C antigen decreased
- Protein C decreased
- Protein S abnormal
- Protein S antigen abnormal
- Protein S antigen decreased
- Protein S decreased
- Protein S free decreased
- Protein S total abnormal
- Protein S total decreased
- Prothrombin abnormal
- Prothrombin activity decreased
- Prothrombin consumption increased
- Prothrombin decreased
- Prothrombin level abnormal
- Prothrombin level abnormal NOS
- Prothrombin level decreased
- Prothrombin ratio decreased
- Prothrombin time abnormal
- Prothrombin time abnormal NOS

PPD




- Prothrombin time ratio abnormal NOS
- Prothrombin time ratio decreased
- Prothrombin time increased
- Prothrombin time prolonged
- Prothrombin time ratio abnormal
- Prothrombin time ratio high
- Prothrombin time ratio increased
- Prothrombin time ratio low
- Prothrombinopenia
- PT increased
- PT prolonged
- Pure intrahepatic cholestasis
- Quick's value decreased
- Radiation hepatitis
- Radiation-induced liver disease
- Raised bilirubin
- Raised INR
- Raised LFTs
- Raised liver enzymes

- Raised liver function tests
- Regenerative siderotic hepatic nodule
- Rejection acute hepatic
- Rejection chronic hepatic
- Renal and liver transplant
- Retention sulfobromophthalein
- Retinol binding protein decreased
- Retrograde portal vein flow
- Reye's syndrome
- Reynold's syndrome
- Scan liver NOS abnormal
- Scleral icterus
- Serum alkaline phosphatase elevated
- Serum bilirubin increased
- Serum cholinesterase decreased
- Serum glutamic-oxaloacetic ta increased
- Serum glutamic-oxaloacetic transaminase increased
- Serum glutamic-pyruvic ta increased
- Serum glutamic-pyruvic transaminase increased

CCI

PPD




| P <sub>1</sub> | refer | red | Term |
|----------------|-------|-----|------|

- Serum transaminase increased
- SGOT increased
- SGPT increased
- Single pass albumin dialysis
- Skin coloring yellow
- Skin colouring yellow
- Small-for-size liver syndrome
- Spider angioma
- Spider naevi
- Spider nevi
- Spider nevus
- Splenic varices
- Splenic varices bleeding
- Splenic varices hemorrhage
- Splenorenal shunt
- Splenorenal shunt procedure
- Splenorenal varices
- Spontaneous intrahepatic portosystemic venous shunt
- Steatohepatitis

- Steatosis hepatic
- Stomal varices
- Subacute fulminant hepatitis
- Subacute hepatic failure
- Subacute hepatic necrosis
- Subacute liver disease
- Subicteric
- Sugiura procedure
- Sulfobromophthalein retention
- Sulphobromophthalein retention
- Supratherapeutic INR
- Syncytial giant cell hepatitis
- Syndrome hepatorenal
- Telangiectases acquired
- Tenderness liver
- Thrombin clotting time abnormal
- Thrombin clotting time prolonged
- Thrombin decreased
- Thrombin time abnormal

PPD




| D. | 4 | · | | Terr | |
|----|-----|----|-----|------|---|
| rı | rei | er | rea | ren | п |

- Thrombin time prolonged
- Thromboplastin decreased
- Todd's cirrhosis
- Total bile acids increased
- Total hepatectomy
- Toxaemia of liver
- Toxemia of liver
- Toxic acute liver disease
- Transaminase glutamic-oxalacetic increased
- Transaminase glutamic-pyruvic increased
- Transaminase NOS increased
- Transaminase value increased
- Transaminases abnormal
- Transaminases increased
- Transaminitis
- Transjugular intrahepatic portosystemic shunt
- Ultrasound liver abnormal
- Unconjugated bilirubinaemia

- Unconjugated bilirubinemia
- Unspecified chronic liver disease without mention of alcohol
- Unspecified disorder of liver
- Unspecified injury to liver with open wound into cavity
- Unspecified injury to liver without mention of open wound into cavity
- Urine ammonia increased
- Urine bilirubin increased
- Urobilin urine absent
- Urobilin urine present
- Urobilinogen appeared
- Urobilinogen negative
- Urobilinogen urine decreased
- Urobilinogen urine increased
- Urobilinogen urine positive
- Varices esophageal
- Varicose veins of abdominal wall
- Vascular spider
- White nipple sign

CCL

PPD






UCB Biopharma SRL Sub-Protocol COV-01-005

COV-01-005 Statistical Analysis Plan


#### **Preferred Term**

- X-ray biliary abnormal
- X-ray hepatobiliary abnormal
- Yellow ocular coloring

| | T 7 11 | | | |
|---|--------|--------|-----|--------|
| • | Yellow | ocular | col | ouring |

Yellow skin

PPD






| Certificate Of Completion | | |
|---------------------------------------|-------------|--------------------|
| Certificate Of Completion PPD | | Status: Completed |
| PPD | | |
| Record Tracking | | |
| Status: Original 7/28/2021 5:21:34 PM | Holder: PPD | Location: DocuSign |
| Signer Events | Signature | Timestamp |

| Signer Events<br>PPD | Signature | Timestamp |
|----------------------|-----------|-----------|

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent Certified Delivered Signing Complete Completed | Hashed/Encrypted Security Checked Security Checked Security Checked | 7/28/2021 5:26:08 PM<br>7/28/2021 8:04:05 PM<br>7/28/2021 8:07:28 PM<br>7/29/2021 5:46:00 AM |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disc | | |

#### CONSENT TO ELECTRONIC DELIVERY AND EXECUTION OF DOCUMENTS

From time to time, [C] ("we" or "us") may provide you certain written contracts, notices, disclosures, authorizations, acknowledgements or other documents (collectively, the "Documents") electronically. Please read this consent form carefully. It explains the terms and conditions under which such Documents are provided by us and executed by you electronically through your DocuSign, Inc. ("DocuSign") user account. If you consent to the delivery and execution of such Documents electronically, please click the "I Agree" button.

#### **Documents** will be sent to you electronically

If you consent to electronic delivery, Documents will be sent to your DocuSign user account. You may request a paper copy of documents previously made available through your DocuSign user account, but an additional charge may be incurred. Alternatively, you can download and print documents sent to your DocuSign user account. Unless otherwise noted, you can access a Document up to 30 days from the date we first sent the Document to you.

#### Withhold Consent or Withdrawing Consent to Electronic Delivery

If you withhold consent to electronic delivery or execution, or withdraw your consent at a later date, all Documents will be sent to your mailing address following our receipt of notice of such action. The following sections explain the consequences of withholding or withdrawing your consent to electronic delivery and execution of Documents, and also the procedures you must follow in order to effectuate delivery to your mailing address.

#### **Consequences of Withdrawing Consent**

By electing to only receive and execute Documents sent to your mailing address, we will not be able to carry out transactions or services as efficiently. For instance, some transactions or services require your express consent. We can perform these transaction or services only if we first receive an acknowledgement that indicates you received and consent to the Document related to the proposed transaction or service.

To withhold consent now or withdraw consent at a later date, please sign DocuSign's "Withdraw Consent" form on the signing page of your DocuSign user account. This will indicate that you have withdrawn your consent to receive Documents electronically. Once you sign the "Withdraw Consent" form, you will no longer be able to use your DocuSign user account to execute Documents electronically and we will send Documents to your mailing address. Withdrawal of consent does not affect the validity of any Documents previously executed electronically prior to such withdrawal of Consent. In addition, should you execute any Documents electronically, your execution of such Documents shall indicate your continued consent to execute such Documents electronically.

### How to contact **CC**

If you would like us to send the Documents to a different e-mail address, request paper copies of Documents you have previously received electronically, or withdraw your consent to receive electronic documents, please follow the instructions below. If you have any other questions, please contact: CCI

## 1. To advise CC of your new e-mail address

If you would like your Documents sent to a different e-mail address, you must send an e-mail message to column and the body of the e-mail please state the following: (i) your previous e-mail address, and (ii) your new e-mail address. No other information is required.

In addition, you must notify DocuSign of your new e-mail address. Please log into your DocuSign user account, and follow the instructions to update your e-mail address.

# 2. To request paper copies from CCI

To request paper copies of Documents you have received previously through your DocuSign user account, send an e-mail to CCI

In the body of the e-mail please state the following: (i) your e-mail address, (ii) full name, (iii) U.S. Postal address, and (iv) telephone number. Additional charges may apply for such paper copies.

#### 3. To withdraw your consent with CC

To withdraw your consent to receiving and executing Documents in an electronic format, you may do one of the following:

i. decline to sign a document from within your DocuSign user account, and on the subsequent page, select the check-box indicating you wish to withdraw your consent; or ii. send us an e-mail to CCI and and in the body of such request you must state your e-mail, full name, US Postal Address, telephone number, and account number. No additional information is necessary.

#### Required hardware and software

| Operating Systems: | Windows® 2000, Windows® XP, Windows Vista®; Mac OS® X |
|---|---|
| Browsers: | <ul> <li>Internet Explorer (Windows Only) 8.0 or above – compatibility mode is supported only for 9.0 and above.</li> <li>Windows Edge Current Version</li> <li>Mozilla Firefox Current Version</li> <li>Safari (Mac OS only) 6.2 or above</li> <li>Google Chrome Current Version</li> </ul> |
| PDF Reader: | Acrobat® or similar software may be required to view and print PDF files |
| Screen Resolution: | 1024 x 768 Recommended |
| Enabled Security Settings: | Allow per session cookies |
| Mobile Signing: | <ul><li>Apple iOS 7.0 or above</li><li>Android 4.0 or above</li></ul> |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, we will provide you with an e-mail message at the e-mail address we have on file for you at the time the hardware and software requirements are revised.

Pre-release (e.g. beta) versions of operating systems and browsers are not supported.

#### Acknowledging your access and consent to receive materials electronically

To confirm you can access this information electronically and that you consent to receiving and executing Documents electronically on the terms and conditions described above, please let us know by clicking the "I Agree" button.

By clicking the "I Agree" button, you confirm that

- You can access and read this Consent To Electronic Delivery and Execution of Documents; and
- You can print on paper the disclosure or save or send the disclosure to a place where you can print it, for future reference and access; and
- Until or unless you notify occur as described above, you consent to the delivery and execution of Documents electronically.